CLINICAL TRIAL: NCT00310388
Title: A Multicenter, Open-Label, Long-Term, Safety, Tolerability and Efficacy Study of Retigabine in Adult Epilepsy Patients With Partial-Onset Seizures (Extension of Study VRX-RET-E22-302)
Brief Title: Open-Label Extension Study of the Phase 3 VRX-RET-E22-302 Double-Blind Trial. 115097
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: No longer any benefit in collecting data since retigabine has been withdrawn from market.
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VRX-RET-E22-304; EUDRACT No. 2006-000956-42; RTG115097 (Other: GlaxoSmithKline)
Record Dates: First submitted 2006-03-30; First posted 2006-04-03 (Estimated); Results first posted 2018-06-06 (Actual); Last update posted 2018-11-15 (Actual); Status verified 2018-10

CONDITIONS: Epilepsy
Keywords: Partial Seizures; Epilepsy; RTG115097; Complex Partial Seizures; Anticonvulsant; Potassium Channels; Epilepsies, Partial
MeSH Terms: conditions — Epilepsy; Seizures; Epilepsies, Partial | interventions — ezogabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Retigabine (INN), Ezogabine (USAN) (Experimental): Retigabine (Ezogabine): all subjects
  Interventions: Drug: Retigabine (INN), Ezogabine (USAN)

INTERVENTIONS:
Drug: Retigabine (INN), Ezogabine (USAN) — Film-coated tablets containing 50 mg, 100 mg, or 300 mg of retigabine per tablet. Dosage and frequency will be specific to each patient so long as the patients receives between 600 and 1200 mg of retigabine per day. The duration will be until the completion of the trial, or until the patient withdraws from the trial.
  Other Names: GW582892X; D-23129; GKE-841

SUMMARY:
This Phase 3 trial is an open-label extension study of the placebo-controlled, double-blind VRX-RET-E22-302 trial. Patients who have completed the VRX-RET-E22-302 trial and who meet inclusion and exclusion criteria will be treated with 600-1200 mg/day of retigabine as an adjunct therapy to their current antiepileptic drugs (AEDs) or vagal nerve stimulation. Treatment will be continued until the subject withdraws from the study or until the program is discontinued. Patients will be recruited from 55-60 sites in Europe, Israel, Australia, and South Africa. The primary objective of the study is to evaluate the safety and tolerability of long-term therapy with retigabine administered as adjunctive therapy in adult epilepsy patients with partial-onset seizures, who completed the double-blind Study VRX-RET-E22-302. Secondary objectives are: to evaluate efficacy of long-term treatment with retigabine and patient quality of life and to evaluate whether retinal pigmentation, unexplained vision loss, pigmentation of non-retinal ocular tissue, and discoloration of nails, lips, skin or mucosa change over time after discontinuation of retigabine.

DETAILED DESCRIPTION:
This Phase 3 trial is an open-label extension study of the placebo-controlled, double-blind VRX-RET-E22-302 trial. Patients who have completed the VRX-RET-E22-302 trial and who meet inclusion and exclusion criteria will be treated with 600-1200 mg/day of retigabine as an adjunct therapy to their current antiepileptic drugs (AEDs) or vagal nerve stimulation. Treatment will be continued until retigabine is commercially available, or until the program is discontinued. Patients will be recruited from 55-60 sites in Europe, Israel, Australia, and South Africa. The safety and tolerability of long-term therapy with retigabine administered as adjunctive therapy in adult epilepsy patients with partial-onset seizures will be evaluated. In addition, the efficacy of long-term treatment with retigabine and patient quality of life will be assessed.

ELIGIBILITY:
Inclusion Criteria:

* Patient has successfully completed the Maintenance and Transition phases of Study VRX-RET-E22-302 for the treatment of partial-onset seizures
* Patient is expected to benefit from participation in the study in the opinion of the Investigator.

Exclusion Criteria:

* Patient meets any of the withdrawal criteria in the previous VRX-RET-E22-302 study or is experiencing an ongoing serious adverse event.
* Patient is receiving any investigational drug or using any experimental device in addition to Retigabine for treatment of epilepsy or any other medical condition.
* Patient has any other condition that would prevent compliance with the study procedures or proper reporting of adverse events.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 376 (Actual)
Dates: Start 2006-07-05 (Actual); Primary Completion 2017-04-18 (Actual); Study Completion 2018-05-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (67):
- Australia (5):
  - Institute of Clniical Neurosciences, Camperdown, New South Wales
  - North Coast Neurology Centre, Maroochydore, Queensland
  - Flinders Medical Centre, Bedford Park, South Australia
  - Royal Melbourne Hospital, Parkville, Victoria
  - Austin & Repatriation Medical Centre, West Heidelberg, Victoria
- Belgium (4):
  - General Hospital Middelheim -- Department of Neurology, Antwerp
  - AZ Sint-Jan, Bruges
  - Universitaire Ziekenhuizen Gasthuisberg -- Department Neurology, Leuven
  - Centre Neurologique William Lennox, Ottignies
- France (4):
  - Hopital Civil de Steasbourg Clinique Neurologie, Levallois-Perret
  - Hopital Neurologique Pierre Wertheimer, Lyon
  - CHU Pontchaillou, Rennes
  - Centre Medical de La Teppe, Tain-l'Hermitage
- Germany (6):
  - Zentrum Epilepsie Erlangen (ZEE) der Universitaet Erlangen, Erlangen, Bavaria
  - Universitaet Giessen / Marburg Neurologie, Marburg, Hesse
  - Universitaetsklinik Mainz Neurologische Klinik, Mainz, Rhineland-Palatinate
  - University of Bonn -- Department for Epileptplogy, Bonn
  - Private Neurologische Paraxis, Muenchen, by
  - Universitaetslinkum Ulm Poliklinik fuer Neurologie, Ulm, BW
- Hungary (3):
  - Pecs University of Science, Clinic of Neurology, Pécs, Ret
  - Orszagos Pszichiatriai es Neurologiai Intezet, Budapest
  - Orszagos Idegsebeszeti Tudomanyos Intezet, Budapest
- Israel (7):
  - Assaf Harofeh Medical Center, Beer Yaakov
  - Rambam Medical Center, Haifa
  - Wolfson Medical Center, Holon
  - Western Galilee Hospital, Nahariya
  - Chaim Sheba Medical Center, Ramat Gan
  - Kaplan Medical Center, Rehovot
  - Tel-Aviv Sourasky Medical Center, Tel Aviv
- Poland (7):
  - Specjalistyczna Przychodnia Lekarska Medikard, Padlewskiego 4, Plock
  - Prywatna Wielospecjalistyczna Lecznica Medyczna "Zycie", Plac Hallera 5, Warszawa
  - Oddzial Neurologii -- Klinika Neurologii ICZMP, U1. Parzeczewska 35, Zgierz
  - NZOZ Przychodnia Internistyczno - Stomatologiczna "Kendron", Bialystok
  - Wojewodzki Szpital Specjalistyczny im.Mikolaja Kopernika, Gdansk
  - WSS im.Kardynala S. Wyszynskiego, Lublin
  - Instytut Psychiatrii i Neurologii II Oddzial Neurologii, Warsaw
- Russia (6):
  - Kazan State Medical University, Kazan'
  - City Hospital # 1, Moscow
  - City Hospital # 33, Moscow
  - District Antiepileptic Centre City Clinical Hospital # 71, Moscow
  - Russian Military Medical Academy, Saint Petersburg
  - Pavlov State Medical University Clinic and Department of Neurology, Saint Petersburg
- South Africa (9):
  - Sunninghill & Kopano Clinical Trials, Johannesburg, Gauteng
  - Wilgers MR & Medical Centre, Pretoria, Gauteng
  - Panorama Medi-Clinic, Parow, W Cape
  - Groote Schuur Hospital, Cape Town, WC
  - Carl Bremer Hospital, Belville, W Cape
  - Farmovs Parexel, BleomFontein, Free State
  - Inkosi Albert Luthuli Central Hospital, Durban, KZ-Natal
  - Johannesburg Hospital, Johannesburg, Gauteng
  - Triple M Research, Port Elisabeth, E Cape
- Spain (7):
  - Hospital Sta. Creu i S. Pau, Barcelona
  - Hospital de Cruces Neurology Department, Bilbao
  - Hosp. de Donostia Neurology Department, Donostia / San Sebastian
  - Hosp. Virgen de las Nieves, Granada
  - Hospital Ruber Internacional de Madrid, Madrid
  - Fundacion Jimenez Diaz, Madrid
  - Hospital Universitario Lozano Blesa Neurology Service, Zaragoza
- Ukraine (5):
  - Psychosomatic Center of Dnepropetr. Regional Clinic, Dnipro
  - Kharkov State Medical University, Kharkiv
  - Institute of Neurology, Psychiatry and Narcology of AMS, Ukr, Kharkiv
  - Epilepsy Center of Municipal Clinical Psychoneurological Hospital, Kiev
  - Odessa Regional Clinical Hospital Center for Neurology and Neurosurgery, Odesa
- United Kingdom (4):
  - The James Cook University Hospital, Middlesbrough, Mersyd
  - Fylde Coast Hospital, Blackpool
  - Western Infirmary (Epilepsy), Glasgow
  - Royal London Hospital, London

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Study Protocol: VRX-RET-E22-304 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: VRX-RET-E22-304 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: VRX-RET-E22-304 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: VRX-RET-E22-304 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: VRX-RET-E22-304 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: VRX-RET-E22-304 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: VRX-RET-E22-304 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was a multi-center, open-label, long-term, safety, tolerability and efficacy study involving 57 study sites in 13 countries (Australia, Belgium, France, Germany, Hungary, Israel, Poland, Russia, South Africa, Spain, Ukraine, the United Kingdom and the United States).
Pre-assignment Details: A total of 376 adult epilepsy participants with partial-onset seizures who completed the parent study (VRX-RET-E22-302 [NCT00235755]) entered this open label extension (OLE) study.
Groups:
- Retigabine: Eligible participants entered a 4-week transition phase of the double-blind parent study (study VRX-RET-E22-302), in which their dose of retigabine was titrated to or maintained at 300 milligrams (mg) three times daily (900 mg per day). Upon completion of the Transition phase of the parent study, participants enrolled into the extension study (RTG115097). Once enrolled in the OLE, doses were adjusted within the range of 600 mg to 1200 mg per day as an adjunct therapy to their ongoing antiepileptic drugs (AEDs) with or without vagal nerve stimulation (VNS) up to 121 months.
- Safety Follow-up Continuation Phase (SFUCP): Participants who withdraw from retigabine and who had retinal pigmentation or unexplained vision loss, pigmentation of non-retinal ocular tissue or discoloration of nails, lips, skin or mucosa entered the SFUCP. During the SFUCP, participants underwent 6-monthly comprehensive eye examinations and/or skin assessments by the investigator, ophthalmologist, retinal specialist or dermatologist as appropriate. Participants were followed up in the SFUCP until the dermatology/ophthalmology finding(s) either resolved or stabilized. Stabilization was defined in the protocol as no changes on two consecutive 6-monthly assessments over at least over 12 months after discontinuation of retigabine.
Period: Primary Reporting Phase
Arm/Group | Retigabine | Safety Follow-up Continuation Phase (SFUCP)
Started | 376 | 0
Completed (Discontinued from Study and Switched to commercial product.) | 30 | 0
Not Completed | 346 | 0
Not completed — Adverse Event | 101 | 0
Not completed — Lack of Efficacy | 56 | 0
Not completed — Withdrawal by Subject | 97 | 0
Not completed — Protocol Violation | 10 | 0
Not completed — Pregnancy | 3 | 0
Not completed — Change in participant medical condition | 3 | 0
Not completed — Persistent ALT/AST above 3 times the ULN | 3 | 0
Not completed — ALT/AST levels above 5 times the ULN | 3 | 0
Not completed — Physician Decision | 2 | 0
Not completed — Request of the sponsor | 19 | 0
Not completed — Failed to return | 8 | 0
Not completed — Participant request unrelated to study | 2 | 0
Not completed — Participant request | 2 | 0
Not completed — Ministry of Health decision | 25 | 0
Not completed — Discontinuation of study | 1 | 0
Not completed — Participant Immigrated to New Zealand | 1 | 0
Not completed — Termination of study at sponsor request | 3 | 0
Not completed — Ongoing SAE from parent study | 1 | 0
Not completed — Due to pigmentation risk concerns | 2 | 0
Not completed — Participant passed away | 1 | 0
Not completed — Participant retired the informed consent | 1 | 0
Not completed — Missing | 1 | 0
Not completed — Other | 1 | 0
Period: Safety Follow-up Continuation Phase
Arm/Group | Retigabine | Safety Follow-up Continuation Phase (SFUCP)
Started | 0 | 26
Completed | 0 | 13
Not Completed | 0 | 13
Not completed — Missing SFUCP disposition information | 0 | 5
Not completed — Adverse Event | 0 | 1
Not completed — Withdrawal by Subject | 0 | 5
Not completed — Study Closed/Terminated | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Retigabine: Eligible participants entered a 4-week transition phase of the double-blind parent study (study VRX-RET-E22-302), in which their dose of retigabine was titrated to or maintained at 300 mg three times daily (900 mg per day). Upon completion of the Transition phase of the parent study, participants enrolled into the extension study (RTG115097). Once enrolled in the OLE, doses were adjusted within the range of 600 mg to 1200 mg per day as an adjunct therapy to their ongoing AEDs with or without VNS up to 121 months.
Arm/Group | Retigabine
Number analyzed (Participants) | 376
Age, Continuous [Mean (Standard Deviation); unit: years] | 37.0 (11.85)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 195
  Male | 181
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Caucasian | 360
  African-American (Black) | 3
  Asian | 3
  Unknown | 10

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment Emergent Adverse Events (TEAEs) and Serious Adverse Events (TESAEs)
Description: An AE is defined as any untoward medical occurrence in a clinical investigation participant, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. SAE is defined as any untoward medical occurrence that, at any dose, results in death, is life threatening, requires hospitalization or prolongation of existing hospitalization, results in disability/incapacity, is a congenital anomaly/birth defect, other situations and is associated with impaired liver function. TEAEs refer to an AE for which the onset was on or after Retigabine dose in this study and on or before 30 days after the last Retigabine dose date. AEs that started in the parent study that worsened in this study were also considered as TEAEs. Analysis was performed on the safety population which included participants who took at least 1 dose of study medication after being enrolled in this OLE study.
Time Frame: Up to 122 months
Population: Safety Population
Measure: Number; unit: Participants
Arm/Group | Retigabine
Number analyzed (Participants) | 376
Participants
  Any TEAE | 324
  Any TESAE | 78

2. Primary Outcome: Number of Participants With TEAEs Leading to Treatment Discontinuation (Disc.)
Description: An AE is defined as any untoward medical occurrence in a participant or clinical investigation participant, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of a medicinal product. A summary of participants with treatment emergent AEs leading to treatment disc. up to 122 months have been presented.
Time Frame: Up to 122 months
Population: Safety Population
Measure: Number; unit: Participants
Arm/Group | Retigabine
Number analyzed (Participants) | 376
Participants | 115

3. Primary Outcome: Kaplan-Meier Estimate of the Probability of Disc. From Study Drug
Description: Kaplan-Meier estimate of the probability of disc. at the specified time for all participants is presented. The time frame of premature study disc. was defined as the time from the day of first the study medication to the time of withdrawal from study drug. For those who had a taper dose start date, the time of withdrawal was the day before the start of taper dose. Participants who switched to commercial product were censored at the last dose of study drug (excluding taper). All participants who withdrew from the study/treatment prematurely but did not switch to commercial product were counted as an event. Number of participants continuing on retigabine at each time of withdrawal were analyzed (represented by n=x in the category titles).
Time Frame: Up to 122 months
Population: Safety Population
Measure: Number; unit: Percentage Probability of disc.
Arm/Group | Retigabine
Number analyzed (Participants) | 376
Percentage Probability of disc.
  Day 0, n=374: number analyzed (Participants) | 374
  Day 0, n=374 | 0.5
  Day 1, n=371: number analyzed (Participants) | 371
  Day 1, n=371 | 1.3
  Day 2, n=369: number analyzed (Participants) | 369
  Day 2, n=369 | 1.9
  Day 3, n=368: number analyzed (Participants) | 368
  Day 3, n=368 | 2.1
  Day 4, n=367: number analyzed (Participants) | 367
  Day 4, n=367 | 2.4
  Day 5, n=366: number analyzed (Participants) | 366
  Day 5, n=366 | 2.7
  Day 6, n=365: number analyzed (Participants) | 365
  Day 6, n=365 | 2.9
  Day 11, n=364: number analyzed (Participants) | 364
  Day 11, n=364 | 3.2
  Day 13, n=363: number analyzed (Participants) | 363
  Day 13, n=363 | 3.5
  Day 14, n=362: number analyzed (Participants) | 362
  Day 14, n=362 | 3.7
  Day 16, n=361: number analyzed (Participants) | 361
  Day 16, n=361 | 4.0
  Day 21, n=360: number analyzed (Participants) | 360
  Day 21, n=360 | 4.3
  Day 22, n=359: number analyzed (Participants) | 359
  Day 22, n=359 | 4.5
  Day 27, n=356: number analyzed (Participants) | 356
  Day 27, n=356 | 5.3
  Day 28, n=350: number analyzed (Participants) | 350
  Day 28, n=350 | 6.9
  Day 29, n=348: number analyzed (Participants) | 348
  Day 29, n=348 | 7.4
  Day 30, n=344: number analyzed (Participants) | 344
  Day 30, n=344 | 8.5
  Day 32, n=343: number analyzed (Participants) | 343
  Day 32, n=343 | 8.8
  Day 35, n=341: number analyzed (Participants) | 341
  Day 35, n=341 | 9.3
  Day 40, n=340: number analyzed (Participants) | 340
  Day 40, n=340 | 9.6
  Day 41, n=339: number analyzed (Participants) | 339
  Day 41, n=339 | 9.8
  Day 42, n=338: number analyzed (Participants) | 338
  Day 42, n=338 | 10.1
  Day 45, n=337: number analyzed (Participants) | 337
  Day 45, n=337 | 10.4
  Day 50, n=336: number analyzed (Participants) | 336
  Day 50, n=336 | 10.6
  Day 56, n=335: number analyzed (Participants) | 335
  Day 56, n=335 | 10.9
  Day 61, n=334: number analyzed (Participants) | 334
  Day 61, n=334 | 11.2
  Day 62, n=333: number analyzed (Participants) | 333
  Day 62, n=333 | 11.4
  Day 63, n=331: number analyzed (Participants) | 331
  Day 63, n=331 | 12.0
  Day 71, n=330: number analyzed (Participants) | 330
  Day 71, n=330 | 12.2
  Day 77, n=329: number analyzed (Participants) | 329
  Day 77, n=329 | 12.5
  Day 82, n=328: number analyzed (Participants) | 328
  Day 82, n=328 | 12.8
  Day 85, n=326: number analyzed (Participants) | 326
  Day 85, n=326 | 13.3
  Day 86, n=325: number analyzed (Participants) | 325
  Day 86, n=325 | 13.6
  Day 88, n=324: number analyzed (Participants) | 324
  Day 88, n=324 | 13.8
  Day 90, n=322: number analyzed (Participants) | 322
  Day 90, n=322 | 14.4
  Day 91, n=316: number analyzed (Participants) | 316
  Day 91, n=316 | 16.0
  Day 92, n=313: number analyzed (Participants) | 313
  Day 92, n=313 | 16.8
  Day 94, n=312: number analyzed (Participants) | 312
  Day 94, n=312 | 17.0
  Day 95, n=310: number analyzed (Participants) | 310
  Day 95, n=310 | 17.6
  Day 99, n=309: number analyzed (Participants) | 309
  Day 99, n=309 | 17.8
  Day 104, n=308: number analyzed (Participants) | 308
  Day 104, n=308 | 18.1
  Day 105, n=307: number analyzed (Participants) | 307
  Day 105, n=307 | 18.4
  Day 107, n=306: number analyzed (Participants) | 306
  Day 107, n=306 | 18.6
  Day 110, n=305: number analyzed (Participants) | 305
  Day 110, n=305 | 18.9
  Day 112, n=303: number analyzed (Participants) | 303
  Day 112, n=303 | 19.4
  Day 118, n=302: number analyzed (Participants) | 302
  Day 118, n=302 | 19.7
  Day 121, n=300: number analyzed (Participants) | 300
  Day 121, n=300 | 20.2
  Day 122, n=299: number analyzed (Participants) | 299
  Day 122, n=299 | 20.5
  Day 126, n=298: number analyzed (Participants) | 298
  Day 126, n=298 | 20.7
  Day 132, n=297: number analyzed (Participants) | 297
  Day 132, n=297 | 21.0
  Day 134, n=296: number analyzed (Participants) | 296
  Day 134, n=296 | 21.3
  Day 135, n=295: number analyzed (Participants) | 295
  Day 135, n=295 | 21.5
  Day 138, n=294: number analyzed (Participants) | 294
  Day 138, n=294 | 21.8
  Day 139, n=293: number analyzed (Participants) | 293
  Day 139, n=293 | 22.1
  Day 141, n=292: number analyzed (Participants) | 292
  Day 141, n=292 | 22.3
  Day 152, n=291: number analyzed (Participants) | 291
  Day 152, n=291 | 22.6
  Day 155, n=290: number analyzed (Participants) | 290
  Day 155, n=290 | 22.9
  Day 161, n=289: number analyzed (Participants) | 289
  Day 161, n=289 | 23.1
  Day 164, n=288: number analyzed (Participants) | 288
  Day 164, n=288 | 23.4
  Day 172, n=287: number analyzed (Participants) | 287
  Day 172, n=287 | 23.7
  Day 176, n=286: number analyzed (Participants) | 286
  Day 176, n=286 | 23.9
  Day 179, n=282: number analyzed (Participants) | 282
  Day 179, n=282 | 25.0
  Day 180, n=278: number analyzed (Participants) | 278
  Day 180, n=278 | 26.1
  Day 181, n=275: number analyzed (Participants) | 275
  Day 181, n=275 | 26.9
  Day 182, n=273: number analyzed (Participants) | 273
  Day 182, n=273 | 27.4
  Day 183, n=272: number analyzed (Participants) | 272
  Day 183, n=272 | 27.7
  Day 184, n=271: number analyzed (Participants) | 271
  Day 184, n=271 | 27.9
  Day 187, n=270: number analyzed (Participants) | 270
  Day 187, n=270 | 28.2
  Day 188, n=269: number analyzed (Participants) | 269
  Day 188, n=269 | 28.5
  Day 189, n=268: number analyzed (Participants) | 268
  Day 189, n=268 | 28.7
  Day 192, n=267: number analyzed (Participants) | 267
  Day 192, n=267 | 29.0
  Day 195, n=265: number analyzed (Participants) | 265
  Day 195, n=265 | 29.5
  Day 198, n=264: number analyzed (Participants) | 264
  Day 198, n=264 | 29.8
  Day 199, n=263: number analyzed (Participants) | 263
  Day 199, n=263 | 30.1
  Day 204, n=262: number analyzed (Participants) | 262
  Day 204, n=262 | 30.3
  Day 214, n=261: number analyzed (Participants) | 261
  Day 214, n=261 | 30.6
  Day 216, n=260: number analyzed (Participants) | 260
  Day 216, n=260 | 30.9
  Day 218, n=259: number analyzed (Participants) | 259
  Day 218, n=259 | 31.1
  Day 221, n=258: number analyzed (Participants) | 258
  Day 221, n=258 | 31.4
  Day 228, n=257: number analyzed (Participants) | 257
  Day 228, n=257 | 31.6
  Day 231, n=256: number analyzed (Participants) | 256
  Day 231, n=256 | 31.9
  Day 233, n=255: number analyzed (Participants) | 255
  Day 233, n=255 | 32.2
  Day 235, n=254: number analyzed (Participants) | 254
  Day 235, n=254 | 32.4
  Day 236, n=253: number analyzed (Participants) | 253
  Day 236, n=253 | 32.7
  Day 237, n=251: number analyzed (Participants) | 251
  Day 237, n=251 | 33.2
  Day 252, n=250: number analyzed (Participants) | 250
  Day 252, n=250 | 33.5
  Day 260, n=249: number analyzed (Participants) | 249
  Day 260, n=249 | 33.8
  Day 264, n=248: number analyzed (Participants) | 248
  Day 264, n=248 | 34.0
  Day 265, n=247: number analyzed (Participants) | 247
  Day 265, n=247 | 34.3
  Day 269, n=246: number analyzed (Participants) | 246
  Day 269, n=246 | 34.6
  Day 270, n=245: number analyzed (Participants) | 245
  Day 270, n=245 | 34.8
  Day 272, n=240: number analyzed (Participants) | 240
  Day 272, n=240 | 36.2
  Day 274, n=239: number analyzed (Participants) | 239
  Day 274, n=239 | 36.4
  Day 275, n=238: number analyzed (Participants) | 238
  Day 275, n=238 | 36.7
  Day 276, n=236: number analyzed (Participants) | 236
  Day 276, n=236 | 37.2
  Day 278, n=235: number analyzed (Participants) | 235
  Day 278, n=235 | 37.5
  Day 279, n=234: number analyzed (Participants) | 234
  Day 279, n=234 | 37.8
  Day 292, n=233: number analyzed (Participants) | 233
  Day 292, n=233 | 38.0
  Day 299, n=231: number analyzed (Participants) | 231
  Day 299, n=231 | 38.6
  Day 301, n=230: number analyzed (Participants) | 230
  Day 301, n=230 | 38.8
  Day 310, n=229: number analyzed (Participants) | 229
  Day 310, n=229 | 39.1
  Day 315, n=228: number analyzed (Participants) | 228
  Day 315, n=228 | 39.4
  Day 316, n=227: number analyzed (Participants) | 227
  Day 316, n=227 | 39.6
  Day 317, n=226: number analyzed (Participants) | 226
  Day 317, n=226 | 39.9
  Day 322, n=225: number analyzed (Participants) | 225
  Day 322, n=225 | 40.2
  Day 325, n=224: number analyzed (Participants) | 224
  Day 325, n=224 | 40.4
  Day 339, n=223: number analyzed (Participants) | 223
  Day 339, n=223 | 40.7
  Day 351, n=222: number analyzed (Participants) | 222
  Day 351, n=222 | 41.0
  Day 357, n=221: number analyzed (Participants) | 221
  Day 357, n=221 | 41.2
  Day 358, n=219: number analyzed (Participants) | 219
  Day 358, n=219 | 41.8
  Day 363, n=218: number analyzed (Participants) | 218
  Day 363, n=218 | 42.0
  Day 372, n=217: number analyzed (Participants) | 217
  Day 372, n=217 | 42.3
  Day 375, n=216: number analyzed (Participants) | 216
  Day 375, n=216 | 42.6
  Day 377, n=215: number analyzed (Participants) | 215
  Day 377, n=215 | 42.8
  Day 416, n=214: number analyzed (Participants) | 214
  Day 416, n=214 | 43.1
  Day 419, n=213: number analyzed (Participants) | 213
  Day 419, n=213 | 43.4
  Day 425, n=212: number analyzed (Participants) | 212
  Day 425, n=212 | 43.6
  Day 429, n=211: number analyzed (Participants) | 211
  Day 429, n=211 | 43.9
  Day 437, n=210: number analyzed (Participants) | 210
  Day 437, n=210 | 44.1
  Day 447, n=209: number analyzed (Participants) | 209
  Day 447, n=209 | 44.4
  Day 455, n=208: number analyzed (Participants) | 208
  Day 455, n=208 | 44.7
  Day 458, n=207: number analyzed (Participants) | 207
  Day 458, n=207 | 44.9
  Day 460, n=206: number analyzed (Participants) | 206
  Day 460, n=206 | 45.2
  Day 461, n=205: number analyzed (Participants) | 205
  Day 461, n=205 | 45.5
  Day 478, n=204: number analyzed (Participants) | 204
  Day 478, n=204 | 45.7
  Day 480, n=203: number analyzed (Participants) | 203
  Day 480, n=203 | 46.0
  Day 482, n=202: number analyzed (Participants) | 202
  Day 482, n=202 | 46.3
  Day 485, n=200: number analyzed (Participants) | 200
  Day 485, n=200 | 46.8
  Day 492, n=197: number analyzed (Participants) | 197
  Day 492, n=197 | 47.6
  Day 493, n=196: number analyzed (Participants) | 196
  Day 493, n=196 | 47.9
  Day 497, n=194: number analyzed (Participants) | 194
  Day 497, n=194 | 48.4
  Day 498, n=193: number analyzed (Participants) | 193
  Day 498, n=193 | 48.7
  Day 501, n=192: number analyzed (Participants) | 192
  Day 501, n=192 | 48.9
  Day 523, n=191: number analyzed (Participants) | 191
  Day 523, n=191 | 49.2
  Day 525, n=190: number analyzed (Participants) | 190
  Day 525, n=190 | 49.5
  Day 534, n=189: number analyzed (Participants) | 189
  Day 534, n=189 | 49.7
  Day 536, n=188: number analyzed (Participants) | 188
  Day 536, n=188 | 50.0
  Day 541, n=187: number analyzed (Participants) | 187
  Day 541, n=187 | 50.3
  Day 553, n=186: number analyzed (Participants) | 186
  Day 553, n=186 | 50.5
  Day 556, n=185: number analyzed (Participants) | 185
  Day 556, n=185 | 50.8
  Day 587, n=184: number analyzed (Participants) | 184
  Day 587, n=184 | 51.1
  Day 593, n=183: number analyzed (Participants) | 183
  Day 593, n=183 | 51.3
  Day 594, n=182: number analyzed (Participants) | 182
  Day 594, n=182 | 51.6
  Day 596, n=181: number analyzed (Participants) | 181
  Day 596, n=181 | 51.9
  Day 601, n=180: number analyzed (Participants) | 180
  Day 601, n=180 | 52.1
  Day 602, n=178: number analyzed (Participants) | 178
  Day 602, n=178 | 52.7
  Day 610, n=177: number analyzed (Participants) | 177
  Day 610, n=177 | 52.9
  Day 612, n=176: number analyzed (Participants) | 176
  Day 612, n=176 | 53.2
  Day 617, n=175: number analyzed (Participants) | 175
  Day 617, n=175 | 53.5
  Day 618, n=174: number analyzed (Participants) | 174
  Day 618, n=174 | 53.7
  Day 632, n=173: number analyzed (Participants) | 173
  Day 632, n=173 | 54.0
  Day 635, n=172: number analyzed (Participants) | 172
  Day 635, n=172 | 54.3
  Day 669, n=171: number analyzed (Participants) | 171
  Day 669, n=171 | 54.5
  Day 676, n=170: number analyzed (Participants) | 170
  Day 676, n=170 | 54.8
  Day 678, n=169: number analyzed (Participants) | 169
  Day 678, n=169 | 55.1
  Day 685, n=168: number analyzed (Participants) | 168
  Day 685, n=168 | 55.3
  Day 700, n=167: number analyzed (Participants) | 167
  Day 700, n=167 | 55.6
  Day 702, n=165: number analyzed (Participants) | 165
  Day 702, n=165 | 56.1
  Day 703, n=164: number analyzed (Participants) | 164
  Day 703, n=164 | 56.4
  Day 707, n=163: number analyzed (Participants) | 163
  Day 707, n=163 | 56.6
  Day 714, n=162: number analyzed (Participants) | 162
  Day 714, n=162 | 56.9
  Day 719, n=161: number analyzed (Participants) | 161
  Day 719, n=161 | 57.2
  Day 720, n=160: number analyzed (Participants) | 160
  Day 720, n=160 | 57.4
  Day 721, n=159: number analyzed (Participants) | 159
  Day 721, n=159 | 57.7
  Day 724, n=158: number analyzed (Participants) | 158
  Day 724, n=158 | 58.0
  Day 729, n=157: number analyzed (Participants) | 157
  Day 729, n=157 | 58.2
  Day 760, n=156: number analyzed (Participants) | 156
  Day 760, n=156 | 58.5
  Day 775, n=155: number analyzed (Participants) | 155
  Day 775, n=155 | 58.8
  Day 777, n=154: number analyzed (Participants) | 154
  Day 777, n=154 | 59.0
  Day 778, n=153: number analyzed (Participants) | 153
  Day 778, n=153 | 59.3
  Day 779, n=152: number analyzed (Participants) | 152
  Day 779, n=152 | 59.6
  Day 781, n=151: number analyzed (Participants) | 151
  Day 781, n=151 | 59.8
  Day 796, n=150: number analyzed (Participants) | 150
  Day 796, n=150 | 60.1
  Day 803, n=149: number analyzed (Participants) | 149
  Day 803, n=149 | 60.4
  Day 818, n=148: number analyzed (Participants) | 148
  Day 818, n=148 | 60.6
  Day 835, n=147: number analyzed (Participants) | 147
  Day 835, n=147 | 60.9
  Day 840, n=146: number analyzed (Participants) | 146
  Day 840, n=146 | 61.2
  Day 841, n=144: number analyzed (Participants) | 144
  Day 841, n=144 | 61.7
  Day 842, n=143: number analyzed (Participants) | 143
  Day 842, n=143 | 62.0
  Day 844, n=142: number analyzed (Participants) | 142
  Day 844, n=142 | 62.2
  Day 845, n=141: number analyzed (Participants) | 141
  Day 845, n=141 | 62.5
  Day 855, n=140: number analyzed (Participants) | 140
  Day 855, n=140 | 62.8
  Day 856, n=139: number analyzed (Participants) | 139
  Day 856, n=139 | 63.0
  Day 863, n=138: number analyzed (Participants) | 138
  Day 863, n=138 | 63.3
  Day 870, n=137: number analyzed (Participants) | 137
  Day 870, n=137 | 63.6
  Day 884, n=136: number analyzed (Participants) | 136
  Day 884, n=136 | 63.8
  Day 893, n=135: number analyzed (Participants) | 135
  Day 893, n=135 | 64.1
  Day 904, n=134: number analyzed (Participants) | 134
  Day 904, n=134 | 64.4
  Day 924, n=133: number analyzed (Participants) | 133
  Day 924, n=133 | 64.6
  Day 927, n=132: number analyzed (Participants) | 132
  Day 927, n=132 | 64.9
  Day 938, n=131: number analyzed (Participants) | 131
  Day 938, n=131 | 65.2
  Day 944, n=130: number analyzed (Participants) | 130
  Day 944, n=130 | 65.4
  Day 947, n=128: number analyzed (Participants) | 128
  Day 947, n=128 | 66.0
  Day 952, n=127: number analyzed (Participants) | 127
  Day 952, n=127 | 66.2
  Day 975, n=126: number analyzed (Participants) | 126
  Day 975, n=126 | 66.5
  Day 980, n=125: number analyzed (Participants) | 125
  Day 980, n=125 | 66.8
  Day 994, n=123: number analyzed (Participants) | 123
  Day 994, n=123 | 67.3
  Day 1067, n=122: number analyzed (Participants) | 122
  Day 1067, n=122 | 67.6
  Day 1074, n=121: number analyzed (Participants) | 121
  Day 1074, n=121 | 67.8
  Day 1084, n=120: number analyzed (Participants) | 120
  Day 1084, n=120 | 68.1
  Day 1091, n=119: number analyzed (Participants) | 119
  Day 1091, n=119 | 68.4
  Day 1129, n=118: number analyzed (Participants) | 118
  Day 1129, n=118 | 68.6
  Day 1141, n=117: number analyzed (Participants) | 117
  Day 1141, n=117 | 68.9
  Day 1142, n=116: number analyzed (Participants) | 116
  Day 1142, n=116 | 69.1
  Day 1148, n=115: number analyzed (Participants) | 115
  Day 1148, n=115 | 69.4
  Day 1196, n=114: number analyzed (Participants) | 114
  Day 1196, n=114 | 69.7
  Day 1198, n=113: number analyzed (Participants) | 113
  Day 1198, n=113 | 69.9
  Day 1206, n=112: number analyzed (Participants) | 112
  Day 1206, n=112 | 70.2
  Day 1207, n=111: number analyzed (Participants) | 111
  Day 1207, n=111 | 70.5
  Day 1211, n=110: number analyzed (Participants) | 110
  Day 1211, n=110 | 70.7
  Day 1221, n=109: number analyzed (Participants) | 109
  Day 1221, n=109 | 71.0
  Day 1231, n=108: number analyzed (Participants) | 108
  Day 1231, n=108 | 71.3
  Day 1299, n=107: number analyzed (Participants) | 107
  Day 1299, n=107 | 71.5
  Day 1316, n=106: number analyzed (Participants) | 106
  Day 1316, n=106 | 71.8
  Day 1322, n=105: number analyzed (Participants) | 105
  Day 1322, n=105 | 72.1
  Day 1389, n=104: number analyzed (Participants) | 104
  Day 1389, n=104 | 72.3
  Day 1413, n=103: number analyzed (Participants) | 103
  Day 1413, n=103 | 72.6
  Day 1436, n=102: number analyzed (Participants) | 102
  Day 1436, n=102 | 72.6
  Day 1446, n=101: number analyzed (Participants) | 101
  Day 1446, n=101 | 72.9
  Day 1450, n=100: number analyzed (Participants) | 100
  Day 1450, n=100 | 73.1
  Day 1451, n=99: number analyzed (Participants) | 99
  Day 1451, n=99 | 73.1
  Day 1452, n=98: number analyzed (Participants) | 98
  Day 1452, n=98 | 73.4
  Day 1521, n=97: number analyzed (Participants) | 97
  Day 1521, n=97 | 73.7
  Day 1541, n=96: number analyzed (Participants) | 96
  Day 1541, n=96 | 73.7
  Day 1545, n=95: number analyzed (Participants) | 95
  Day 1545, n=95 | 73.7
  Day 1547, n=94: number analyzed (Participants) | 94
  Day 1547, n=94 | 74.0
  Day 1563, n=93: number analyzed (Participants) | 93
  Day 1563, n=93 | 74.0
  Day 1567, n=92: number analyzed (Participants) | 92
  Day 1567, n=92 | 74.2
  Day 1569, n=91: number analyzed (Participants) | 91
  Day 1569, n=91 | 74.5
  Day 1589, n=90: number analyzed (Participants) | 90
  Day 1589, n=90 | 74.5
  Day 1618, n=89: number analyzed (Participants) | 89
  Day 1618, n=89 | 74.5
  Day 1619, n=88: number analyzed (Participants) | 88
  Day 1619, n=88 | 74.5
  Day 1623, n=87: number analyzed (Participants) | 87
  Day 1623, n=87 | 74.5
  Day 1632, n=86: number analyzed (Participants) | 86
  Day 1632, n=86 | 74.5
  Day 1656, n=85: number analyzed (Participants) | 85
  Day 1656, n=85 | 74.5
  Day 1660, n=84: number analyzed (Participants) | 84
  Day 1660, n=84 | 74.5
  Day 1668, n=83: number analyzed (Participants) | 83
  Day 1668, n=83 | 74.8
  Day 1672, n=82: number analyzed (Participants) | 82
  Day 1672, n=82 | 75.1
  Day 1676, n=81: number analyzed (Participants) | 81
  Day 1676, n=81 | 75.4
  Day 1680, n=80: number analyzed (Participants) | 80
  Day 1680, n=80 | 75.4
  Day 1694, n=79: number analyzed (Participants) | 79
  Day 1694, n=79 | 75.4
  Day 1697, n=78: number analyzed (Participants) | 78
  Day 1697, n=78 | 75.4
  Day 1752, n=77: number analyzed (Participants) | 77
  Day 1752, n=77 | 75.4
  Day 1756, n=76: number analyzed (Participants) | 76
  Day 1756, n=76 | 75.8
  Day 1760, n=75: number analyzed (Participants) | 75
  Day 1760, n=75 | 75.8
  Day 1792, n=74: number analyzed (Participants) | 74
  Day 1792, n=74 | 76.1
  Day 1802, n=73: number analyzed (Participants) | 73
  Day 1802, n=73 | 76.1
  Day 1807, n=72: number analyzed (Participants) | 72
  Day 1807, n=72 | 76.1
  Day 1814, n=71: number analyzed (Participants) | 71
  Day 1814, n=71 | 76.4
  Day 1819, n=70: number analyzed (Participants) | 70
  Day 1819, n=70 | 76.4
  Day 1836, n=69: number analyzed (Participants) | 69
  Day 1836, n=69 | 76.4
  Day 1849, n=68: number analyzed (Participants) | 68
  Day 1849, n=68 | 76.4
  Day 1855, n=67: number analyzed (Participants) | 67
  Day 1855, n=67 | 76.4
  Day 1887, n=66: number analyzed (Participants) | 66
  Day 1887, n=66 | 76.4
  Day 1895, n=65: number analyzed (Participants) | 65
  Day 1895, n=65 | 76.8
  Day 1904, n=64: number analyzed (Participants) | 64
  Day 1904, n=64 | 76.8
  Day 1919, n=63: number analyzed (Participants) | 63
  Day 1919, n=63 | 76.8
  Day 1920, n=62: number analyzed (Participants) | 62
  Day 1920, n=62 | 77.1
  Day 1926, n=61: number analyzed (Participants) | 61
  Day 1926, n=61 | 77.5
  Day 1928, n=60: number analyzed (Participants) | 60
  Day 1928, n=60 | 77.5
  Day 1929, n=59: number analyzed (Participants) | 59
  Day 1929, n=59 | 77.9
  Day 1931, n=58: number analyzed (Participants) | 58
  Day 1931, n=58 | 78.3
  Day 1937, n=57: number analyzed (Participants) | 57
  Day 1937, n=57 | 78.3
  Day 1951, n=56: number analyzed (Participants) | 56
  Day 1951, n=56 | 78.6
  Day 2005, n=55: number analyzed (Participants) | 55
  Day 2005, n=55 | 79.0
  Day 2037, n=54: number analyzed (Participants) | 54
  Day 2037, n=54 | 79.4
  Day 2044, n=53: number analyzed (Participants) | 53
  Day 2044, n=53 | 79.4
  Day 2092, n=52: number analyzed (Participants) | 52
  Day 2092, n=52 | 79.8
  Day 2157, n=51: number analyzed (Participants) | 51
  Day 2157, n=51 | 80.2
  Day 2161, n=50: number analyzed (Participants) | 50
  Day 2161, n=50 | 80.6
  Day 2162, n=49: number analyzed (Participants) | 49
  Day 2162, n=49 | 81.0
  Day 2182, n=48: number analyzed (Participants) | 48
  Day 2182, n=48 | 81.3
  Day 2183, n=47: number analyzed (Participants) | 47
  Day 2183, n=47 | 81.7
  Day 2184, n=46: number analyzed (Participants) | 46
  Day 2184, n=46 | 82.1
  Day 2227, n=45: number analyzed (Participants) | 45
  Day 2227, n=45 | 82.5
  Day 2281, n=44: number analyzed (Participants) | 44
  Day 2281, n=44 | 82.9
  Day 2283, n=43: number analyzed (Participants) | 43
  Day 2283, n=43 | 83.3
  Day 2285, n=42: number analyzed (Participants) | 42
  Day 2285, n=42 | 83.7
  Day 2296, n=41: number analyzed (Participants) | 41
  Day 2296, n=41 | 83.7
  Day 2317, n=40: number analyzed (Participants) | 40
  Day 2317, n=40 | 84.1
  Day 2380, n=39: number analyzed (Participants) | 39
  Day 2380, n=39 | 84.5
  Day 2395, n=37: number analyzed (Participants) | 37
  Day 2395, n=37 | 85.3
  Day 2400, n=36: number analyzed (Participants) | 36
  Day 2400, n=36 | 85.7
  Day 2405, n=35: number analyzed (Participants) | 35
  Day 2405, n=35 | 86.1
  Day 2408, n=34: number analyzed (Participants) | 34
  Day 2408, n=34 | 86.5
  Day 2415, n=33: number analyzed (Participants) | 33
  Day 2415, n=33 | 86.9
  Day 2443, n=32: number analyzed (Participants) | 32
  Day 2443, n=32 | 86.9
  Day 2525, n=31: number analyzed (Participants) | 31
  Day 2525, n=31 | 87.3
  Day 2533, n=30: number analyzed (Participants) | 30
  Day 2533, n=30 | 87.7
  Day 2537, n=29: number analyzed (Participants) | 29
  Day 2537, n=29 | 88.1
  Day 2639, n=28: number analyzed (Participants) | 28
  Day 2639, n=28 | 88.5
  Day 2664, n=27: number analyzed (Participants) | 27
  Day 2664, n=27 | 88.9
  Day 2772, n=26: number analyzed (Participants) | 26
  Day 2772, n=26 | 89.3
  Day 2793, n=25: number analyzed (Participants) | 25
  Day 2793, n=25 | 89.7
  Day 2829, n=24: number analyzed (Participants) | 24
  Day 2829, n=24 | 90.1
  Day 2870, n=23: number analyzed (Participants) | 23
  Day 2870, n=23 | 90.6
  Day 2884, n=22: number analyzed (Participants) | 22
  Day 2884, n=22 | 91.0
  Day 2973, n=21: number analyzed (Participants) | 21
  Day 2973, n=21 | 91.4
  Day 2975, n=20: number analyzed (Participants) | 20
  Day 2975, n=20 | 91.8
  Day 2998, n=19: number analyzed (Participants) | 19
  Day 2998, n=19 | 92.2
  Day 3101, n=18: number analyzed (Participants) | 18
  Day 3101, n=18 | 92.6
  Day 3118, n=17: number analyzed (Participants) | 17
  Day 3118, n=17 | 93.0
  Day 3137, n=16: number analyzed (Participants) | 16
  Day 3137, n=16 | 93.4
  Day 3144, n=15: number analyzed (Participants) | 15
  Day 3144, n=15 | 93.8
  Day 3147, n=14: number analyzed (Participants) | 14
  Day 3147, n=14 | 94.3
  Day 3185, n=13: number analyzed (Participants) | 13
  Day 3185, n=13 | 94.7
  Day 3220, n=11: number analyzed (Participants) | 11
  Day 3220, n=11 | 95.5
  Day 3231, n=10: number analyzed (Participants) | 10
  Day 3231, n=10 | 95.9
  Day 3243, n=9: number analyzed (Participants) | 9
  Day 3243, n=9 | 96.3
  Day 3246, n=8: number analyzed (Participants) | 8
  Day 3246, n=8 | 96.7
  Day 3276, n=7: number analyzed (Participants) | 7
  Day 3276, n=7 | 97.1
  Day 3277, n=6: number analyzed (Participants) | 6
  Day 3277, n=6 | 97.5
  Day 3285, n=5: number analyzed (Participants) | 5
  Day 3285, n=5 | 97.9
  Day 3318, n=4: number analyzed (Participants) | 4
  Day 3318, n=4 | 98.4
  Day 3360, n=3: number analyzed (Participants) | 3
  Day 3360, n=3 | 98.8
  Day 3483, n=2: number analyzed (Participants) | 2
  Day 3483, n=2 | 99.2
  Day 3582, n=1: number analyzed (Participants) | 1
  Day 3582, n=1 | 99.6

4. Primary Outcome: Change From Baseline in Systolic Blood Pressure (SBP) and Diastolic Blood Pressure (DBP) Measurements in the Supine and Standing Position
Description: Vital sign measurements (supine and standing blood pressure ) were obtained throughout the study at all visits during the Open-Label Treatment Phase of the study. Evaluations of blood pressure were performed supine at each study visit, and again after the participant had been standing for approximately 2 minutes. Baseline assessment in this OLE study was defined as the last assessment of that endpoint in VRX-RET-E22-302 taken prior to the first active treatment with retigabine. Change from Baseline was calculated by subtracting the Baseline value from the post Baseline values. NA indicates standard deviation could not be calculated as only 1 participant was analyzed. Only those participants with data available at the specified time points were analyzed (represented by n=X in the category titles).
Time Frame: Baseline and up to 122 months
Population: Safety Population
Measure: Mean (Standard Deviation); unit: Millimeters of mercury
Arm/Group | Retigabine
Number analyzed (Participants) | 376
Millimeters of mercury
  Supine DBP, Visit 1 (Month 1), n=358: number analyzed (Participants) | 358
  Supine DBP, Visit 1 (Month 1), n=358 | 0.4 (10.05)
  Supine DBP, Visit 2 (Month 3), n=328: number analyzed (Participants) | 328
  Supine DBP, Visit 2 (Month 3), n=328 | 0.3 (9.83)
  Supine DBP, Visit 3 (Month 6), n=287: number analyzed (Participants) | 287
  Supine DBP, Visit 3 (Month 6), n=287 | -0.2 (10.19)
  Supine DBP, Visit 4 (Month 9), n=251: number analyzed (Participants) | 251
  Supine DBP, Visit 4 (Month 9), n=251 | 0.0 (11.09)
  Supine DBP, Visit 5 (Month 12), n=235: number analyzed (Participants) | 235
  Supine DBP, Visit 5 (Month 12), n=235 | 0.7 (10.79)
  Supine DBP, Visit 6 (Month 16), n=202: number analyzed (Participants) | 202
  Supine DBP, Visit 6 (Month 16), n=202 | 1.0 (10.02)
  Supine DBP, Visit 7 (Month 20), n=181: number analyzed (Participants) | 181
  Supine DBP, Visit 7 (Month 20), n=181 | 0.4 (10.03)
  Supine DBP, Visit 8 (Month 24), n=167: number analyzed (Participants) | 167
  Supine DBP, Visit 8 (Month 24), n=167 | 0.4 (10.63)
  Supine DBP, Visit 9 (Month 28), n=147: number analyzed (Participants) | 147
  Supine DBP, Visit 9 (Month 28), n=147 | 1.5 (10.62)
  Supine DBP, Visit 10 (Month 32), n=128: number analyzed (Participants) | 128
  Supine DBP, Visit 10 (Month 32), n=128 | 0.0 (10.42)
  Supine DBP, Visit 11 (Month 36), n=121: number analyzed (Participants) | 121
  Supine DBP, Visit 11 (Month 36), n=121 | 1.0 (10.65)
  Supine DBP,Visit 12 (Month 40), n=112: number analyzed (Participants) | 112
  Supine DBP,Visit 12 (Month 40), n=112 | 2.0 (10.37)
  Supine DBP, Visit 13 (Month 44), n=105: number analyzed (Participants) | 105
  Supine DBP, Visit 13 (Month 44), n=105 | 0.5 (9.54)
  Supine DBP, Visit 14 (Month 48), n=104: number analyzed (Participants) | 104
  Supine DBP, Visit 14 (Month 48), n=104 | 0.0 (10.30)
  Supine DBP, Visit 15 (Month 52), n=91: number analyzed (Participants) | 91
  Supine DBP, Visit 15 (Month 52), n=91 | 0.1 (11.10)
  Supine DBP, Visit 16 (Month 56), n=77: number analyzed (Participants) | 77
  Supine DBP, Visit 16 (Month 56), n=77 | 1.2 (9.68)
  Supine DBP, Visit 17 (Month 60), n=92: number analyzed (Participants) | 92
  Supine DBP, Visit 17 (Month 60), n=92 | -1.0 (11.08)
  Supine DBP, Visit 18 (Month 64), n=58: number analyzed (Participants) | 58
  Supine DBP, Visit 18 (Month 64), n=58 | 1.6 (8.29)
  Supine DBP, Visit 19 (Month 68), n=53: number analyzed (Participants) | 53
  Supine DBP, Visit 19 (Month 68), n=53 | 0.6 (8.66)
  Supine DBP, Visit 20 (Month 72), n=61: number analyzed (Participants) | 61
  Supine DBP, Visit 20 (Month 72), n=61 | 1.3 (8.38)
  Supine DBP, Visit 21 (Month 76), n=43: number analyzed (Participants) | 43
  Supine DBP, Visit 21 (Month 76), n=43 | 3.2 (8.88)
  Supine DBP, Visit 22 (Month 80), n=37: number analyzed (Participants) | 37
  Supine DBP, Visit 22 (Month 80), n=37 | 1.8 (7.66)
  Supine DBP, Visit 23 (Month 84), n=32: number analyzed (Participants) | 32
  Supine DBP, Visit 23 (Month 84), n=32 | -1.4 (8.64)
  Supine DBP, Visit 24 (Month 88), n=29: number analyzed (Participants) | 29
  Supine DBP, Visit 24 (Month 88), n=29 | 3.4 (8.83)
  Supine DBP, Visit 25 (Month 92), n=25: number analyzed (Participants) | 25
  Supine DBP, Visit 25 (Month 92), n=25 | 2.3 (7.29)
  Supine DBP, Visit 26 (Month 96), n=26: number analyzed (Participants) | 26
  Supine DBP, Visit 26 (Month 96), n=26 | 1.5 (10.10)
  Supine DBP, Visit 27 (Month 100), n=20: number analyzed (Participants) | 20
  Supine DBP, Visit 27 (Month 100), n=20 | 1.5 (8.42)
  Supine DBP, Visit 28 (Month 104), n=17: number analyzed (Participants) | 17
  Supine DBP, Visit 28 (Month 104), n=17 | 3.4 (10.56)
  Supine DBP, Visit 29 (Month 108), n=13: number analyzed (Participants) | 13
  Supine DBP, Visit 29 (Month 108), n=13 | 0.5 (6.74)
  Supine DBP, Visit 30 (Month 112), n=4: number analyzed (Participants) | 4
  Supine DBP, Visit 30 (Month 112), n=4 | 4.0 (7.30)
  Supine DBP, Visit 31 (Month 116), n=3: number analyzed (Participants) | 3
  Supine DBP, Visit 31 (Month 116), n=3 | 11.0 (7.55)
  Supine DBP, Visit 32 (Month 120), n=1: number analyzed (Participants) | 1
  Supine DBP, Visit 32 (Month 120), n=1 | -2.0 (NA) — Standard deviation could not be calculated as only 1 participant was analyzed.
  Supine DBP, Follow up, n=267: number analyzed (Participants) | 267
  Supine DBP, Follow up, n=267 | 1.3 (10.08)
  Standing DBP, Visit 1 (Month 1), n=357: number analyzed (Participants) | 357
  Standing DBP, Visit 1 (Month 1), n=357 | 0.6 (10.68)
  Standing DBP, Visit 2 (Month 3), n=328: number analyzed (Participants) | 328
  Standing DBP, Visit 2 (Month 3), n=328 | 0.2 (10.62)
  Standing DBP, Visit 3 (Month 6), n=287: number analyzed (Participants) | 287
  Standing DBP, Visit 3 (Month 6), n=287 | -0.1 (10.21)
  Standing DBP, Visit 4 (Month 9), n=251: number analyzed (Participants) | 251
  Standing DBP, Visit 4 (Month 9), n=251 | 0.2 (10.14)
  Standing DBP, Visit 5 (Month 12), n=235: number analyzed (Participants) | 235
  Standing DBP, Visit 5 (Month 12), n=235 | 0.8 (10.17)
  Standing DBP, Visit 6 (Month 16), n=202: number analyzed (Participants) | 202
  Standing DBP, Visit 6 (Month 16), n=202 | 0.3 (10.16)
  Standing DBP, Visit 7 (Month 20), n=181: number analyzed (Participants) | 181
  Standing DBP, Visit 7 (Month 20), n=181 | 0.4 (9.51)
  Standing DBP, Visit 8 (Month 24), n=167: number analyzed (Participants) | 167
  Standing DBP, Visit 8 (Month 24), n=167 | 0.2 (9.83)
  Standing DBP, Visit 9 (Month 28), n=147: number analyzed (Participants) | 147
  Standing DBP, Visit 9 (Month 28), n=147 | 0.3 (10.00)
  Standing DBP, Visit 10 (Month 32), n=128: number analyzed (Participants) | 128
  Standing DBP, Visit 10 (Month 32), n=128 | -0.6 (10.64)
  Standing DBP, Visit 11 (Month 36), n=121: number analyzed (Participants) | 121
  Standing DBP, Visit 11 (Month 36), n=121 | 0.9 (10.94)
  Standing DBP, Visit 12 (Month 40), n=111: number analyzed (Participants) | 111
  Standing DBP, Visit 12 (Month 40), n=111 | 1.4 (11.01)
  Standing DBP, Visit 13 (Month 44), n=105: number analyzed (Participants) | 105
  Standing DBP, Visit 13 (Month 44), n=105 | -0.2 (10.76)
  Standing DBP, Visit 14 (Month 48), n=104: number analyzed (Participants) | 104
  Standing DBP, Visit 14 (Month 48), n=104 | 0.3 (10.35)
  Standing DBP, Visit 15 (Month 52), n=91: number analyzed (Participants) | 91
  Standing DBP, Visit 15 (Month 52), n=91 | -1.5 (11.00)
  Standing DBP, Visit 16 (Month 56), n=77: number analyzed (Participants) | 77
  Standing DBP, Visit 16 (Month 56), n=77 | -0.3 (10.40)
  Standing DBP, Visit 17 (Month 60), n=92: number analyzed (Participants) | 92
  Standing DBP, Visit 17 (Month 60), n=92 | -1.5 (9.70)
  Standing DBP, Visit 18 (Month 64), n=58: number analyzed (Participants) | 58
  Standing DBP, Visit 18 (Month 64), n=58 | 0.5 (8.07)
  Standing DBP, Visit 19 (Month 68), n=53: number analyzed (Participants) | 53
  Standing DBP, Visit 19 (Month 68), n=53 | 0.0 (7.20)
  Standing DBP, Visit 20 (Month 72), n=61: number analyzed (Participants) | 61
  Standing DBP, Visit 20 (Month 72), n=61 | 0.3 (8.31)
  Standing DBP, Visit 21 (Month 76), n=43: number analyzed (Participants) | 43
  Standing DBP, Visit 21 (Month 76), n=43 | 1.4 (8.93)
  Standing DBP, Visit 22 (Month 80), n=37: number analyzed (Participants) | 37
  Standing DBP, Visit 22 (Month 80), n=37 | 0.3 (8.03)
  Standing DBP, Visit 23 (Month 84), n=32: number analyzed (Participants) | 32
  Standing DBP, Visit 23 (Month 84), n=32 | -0.4 (7.98)
  Standing DBP, Visit 24 (Month 88), n=29: number analyzed (Participants) | 29
  Standing DBP, Visit 24 (Month 88), n=29 | 1.6 (8.38)
  Standing DBP, Visit 25 (Month 92), n=25: number analyzed (Participants) | 25
  Standing DBP, Visit 25 (Month 92), n=25 | 1.0 (7.33)
  Standing DBP, Visit 26 (Month 96), n=26: number analyzed (Participants) | 26
  Standing DBP, Visit 26 (Month 96), n=26 | 1.6 (9.20)
  Standing DBP, Visit 27 (Month 100), n=20: number analyzed (Participants) | 20
  Standing DBP, Visit 27 (Month 100), n=20 | 0.2 (10.48)
  Standing DBP, Visit 28 (Month 104), n=17: number analyzed (Participants) | 17
  Standing DBP, Visit 28 (Month 104), n=17 | 2.8 (11.65)
  Standing DBP, Visit 29 (Month 108), n=13: number analyzed (Participants) | 13
  Standing DBP, Visit 29 (Month 108), n=13 | -0.5 (9.42)
  Standing DBP, Visit 30 (Month 112), n=4: number analyzed (Participants) | 4
  Standing DBP, Visit 30 (Month 112), n=4 | 1.3 (9.18)
  Standing DBP, Visit 31 (Month 116), n=3: number analyzed (Participants) | 3
  Standing DBP, Visit 31 (Month 116), n=3 | 8.0 (11.79)
  Standing DBP, Visit 32 (Month 120), n=1: number analyzed (Participants) | 1
  Standing DBP, Visit 32 (Month 120), n=1 | -1.0 (NA) — Standard deviation could not be calculated as only 1 participant was analyzed.
  Standing DBP, Follow up, n=267: number analyzed (Participants) | 267
  Standing DBP, Follow up, n=267 | 2.0 (10.57)
  Supine SBP, Visit 1 (Month 1), n=358: number analyzed (Participants) | 358
  Supine SBP, Visit 1 (Month 1), n=358 | -0.2 (12.03)
  Supine SBP, Visit 2 (Month 3), n=328: number analyzed (Participants) | 328
  Supine SBP, Visit 2 (Month 3), n=328 | -0.4 (12.09)
  Supine SBP, Visit 3 (Month 6), n=287: number analyzed (Participants) | 287
  Supine SBP, Visit 3 (Month 6), n=287 | 0.5 (13.53)
  Supine SBP, Visit 4 (Month 9), n=251: number analyzed (Participants) | 251
  Supine SBP, Visit 4 (Month 9), n=251 | 0.0 (15.32)
  Supine SBP, Visit 5 (Month 12), n=235: number analyzed (Participants) | 235
  Supine SBP, Visit 5 (Month 12), n=235 | 0.5 (12.99)
  Supine SBP, Visit 6 (Month 16), n=202: number analyzed (Participants) | 202
  Supine SBP, Visit 6 (Month 16), n=202 | 0.7 (14.39)
  Supine SBP, Visit 7 (Month 20), n=181: number analyzed (Participants) | 181
  Supine SBP, Visit 7 (Month 20), n=181 | -0.5 (14.34)
  Supine SBP, Visit 8 (Month 24), n=167: number analyzed (Participants) | 167
  Supine SBP, Visit 8 (Month 24), n=167 | -0.4 (14.11)
  Supine SBP, Visit 9 (Month 28), n=147: number analyzed (Participants) | 147
  Supine SBP, Visit 9 (Month 28), n=147 | 0.2 (13.78)
  Supine SBP, Visit 10 (Month 32), n=128: number analyzed (Participants) | 128
  Supine SBP, Visit 10 (Month 32), n=128 | 0.3 (13.60)
  Supine SBP, Visit 11 (Month 36), n=121: number analyzed (Participants) | 121
  Supine SBP, Visit 11 (Month 36), n=121 | 0.2 (14.90)
  Supine SBP, Visit 12 (Month 40), n=112: number analyzed (Participants) | 112
  Supine SBP, Visit 12 (Month 40), n=112 | 1.3 (13.90)
  Supine SBP, Visit 13 (Month 44), n=105: number analyzed (Participants) | 105
  Supine SBP, Visit 13 (Month 44), n=105 | 0.1 (11.28)
  Supine SBP, Visit 14 (Month 48), n=104: number analyzed (Participants) | 104
  Supine SBP, Visit 14 (Month 48), n=104 | -1.1 (13.03)
  Supine SBP, Visit 15 (Month 52), n=91: number analyzed (Participants) | 91
  Supine SBP, Visit 15 (Month 52), n=91 | -0.7 (14.05)
  Supine SBP, Visit 16 (Month 56), n=77: number analyzed (Participants) | 77
  Supine SBP, Visit 16 (Month 56), n=77 | 2.6 (13.41)
  Supine SBP, Visit 17 (Month 60), n=92: number analyzed (Participants) | 92
  Supine SBP, Visit 17 (Month 60), n=92 | -0.2 (14.48)
  Supine SBP, Visit 18 (Month 64), n=58: number analyzed (Participants) | 58
  Supine SBP, Visit 18 (Month 64), n=58 | 1.8 (12.11)
  Supine SBP, Visit 19 (Month 68), n=53: number analyzed (Participants) | 53
  Supine SBP, Visit 19 (Month 68), n=53 | 1.1 (13.00)
  Supine SBP, Visit 20 (Month 72), n=61: number analyzed (Participants) | 61
  Supine SBP, Visit 20 (Month 72), n=61 | 2.5 (10.26)
  Supine SBP, Visit 21 (Month 76), n=43: number analyzed (Participants) | 43
  Supine SBP, Visit 21 (Month 76), n=43 | 4.4 (15.51)
  Supine SBP, Visit 22 (Month 80), n=37: number analyzed (Participants) | 37
  Supine SBP, Visit 22 (Month 80), n=37 | 2.3 (15.13)
  Supine SBP, Visit 23 (Month 84), n=32: number analyzed (Participants) | 32
  Supine SBP, Visit 23 (Month 84), n=32 | 1.1 (13.90)
  Supine SBP, Visit 24 (Month 88), n=29: number analyzed (Participants) | 29
  Supine SBP, Visit 24 (Month 88), n=29 | 2.7 (12.51)
  Supine SBP, Visit 25 (Month 92), n=25: number analyzed (Participants) | 25
  Supine SBP, Visit 25 (Month 92), n=25 | 2.8 (10.44)
  Supine SBP, Visit 26 (Month 96), n=26: number analyzed (Participants) | 26
  Supine SBP, Visit 26 (Month 96), n=26 | 2.9 (14.66)
  Supine SBP, Visit 27 (Month 100), n=20: number analyzed (Participants) | 20
  Supine SBP, Visit 27 (Month 100), n=20 | 2.6 (10.61)
  Supine SBP, Visit 28 (Month 104), n=17: number analyzed (Participants) | 17
  Supine SBP, Visit 28 (Month 104), n=17 | 5.8 (10.91)
  Supine SBP, Visit 29 (Month 108), n=13: number analyzed (Participants) | 13
  Supine SBP, Visit 29 (Month 108), n=13 | -2.2 (8.68)
  Supine SBP, Visit 30 (Month 112), n=4: number analyzed (Participants) | 4
  Supine SBP, Visit 30 (Month 112), n=4 | 8.5 (6.95)
  Supine SBP, Visit 31 (Month 116), n=3: number analyzed (Participants) | 3
  Supine SBP, Visit 31 (Month 116), n=3 | 13.7 (4.93)
  Supine SBP, Visit 32 (Month 120), n=1: number analyzed (Participants) | 1
  Supine SBP, Visit 32 (Month 120), n=1 | 11.0 (NA) — Standard deviation could not be calculated as only 1 participant was analyzed
  Supine SBP, Follow up, n=267: number analyzed (Participants) | 267
  Supine SBP, Follow up, n=267 | 1.2 (14.15)
  Standing SBP, Visit 1 (Month 1), n=357: number analyzed (Participants) | 357
  Standing SBP, Visit 1 (Month 1), n=357 | -1.2 (12.20)
  Standing SBP, Visit 2 (Month 3), n=328: number analyzed (Participants) | 328
  Standing SBP, Visit 2 (Month 3), n=328 | -0.7 (13.30)
  Standing SBP, Visit 3 (Month 6), n=287: number analyzed (Participants) | 287
  Standing SBP, Visit 3 (Month 6), n=287 | -0.2 (13.89)
  Standing SBP, Visit 4 (Month 9), n=251: number analyzed (Participants) | 251
  Standing SBP, Visit 4 (Month 9), n=251 | -0.7 (15.10)
  Standing SBP, Visit 5 (Month 12), n=235: number analyzed (Participants) | 235
  Standing SBP, Visit 5 (Month 12), n=235 | -0.7 (14.56)
  Standing SBP, Visit 6 (Month 16), n=202: number analyzed (Participants) | 202
  Standing SBP, Visit 6 (Month 16), n=202 | -0.3 (14.09)
  Standing SBP, Visit 7 (Month 20), n=181: number analyzed (Participants) | 181
  Standing SBP, Visit 7 (Month 20), n=181 | -0.8 (15.19)
  Standing SBP, Visit 8 (Month 24), n=167: number analyzed (Participants) | 167
  Standing SBP, Visit 8 (Month 24), n=167 | -0.5 (15.35)
  Standing SBP, Visit 9 (Month 28), n=147: number analyzed (Participants) | 147
  Standing SBP, Visit 9 (Month 28), n=147 | -0.3 (16.30)
  Standing SBP, Visit 10 (Month 32), n=128: number analyzed (Participants) | 128
  Standing SBP, Visit 10 (Month 32), n=128 | -0.1 (15.06)
  Standing SBP, Visit 11 (Month 36), n=121: number analyzed (Participants) | 121
  Standing SBP, Visit 11 (Month 36), n=121 | 0.7 (15.51)
  Standing SBP, Visit 12 (Month 40), n=111: number analyzed (Participants) | 111
  Standing SBP, Visit 12 (Month 40), n=111 | 2.7 (14.21)
  Standing SBP, Visit 13 (Month 44), n=105: number analyzed (Participants) | 105
  Standing SBP, Visit 13 (Month 44), n=105 | -1.3 (12.57)
  Standing SBP, Visit 14 (Month 48), n=104: number analyzed (Participants) | 104
  Standing SBP, Visit 14 (Month 48), n=104 | -1.6 (14.67)
  Standing SBP, Visit 15 (Month 52), n=91: number analyzed (Participants) | 91
  Standing SBP, Visit 15 (Month 52), n=91 | -1.2 (14.35)
  Standing SBP, Visit 16 (Month 56), n=77: number analyzed (Participants) | 77
  Standing SBP, Visit 16 (Month 56), n=77 | 0.9 (15.04)
  Standing SBP, Visit 17 (Month 60), n=92: number analyzed (Participants) | 92
  Standing SBP, Visit 17 (Month 60), n=92 | -0.7 (14.92)
  Standing SBP, Visit 18 (Month 64), n= 58: number analyzed (Participants) | 58
  Standing SBP, Visit 18 (Month 64), n= 58 | 0.6 (12.84)
  Standing SBP, Visit 19 (Month 68), n=53: number analyzed (Participants) | 53
  Standing SBP, Visit 19 (Month 68), n=53 | 0.2 (11.85)
  Standing SBP, Visit 20 (Month 72), n=61: number analyzed (Participants) | 61
  Standing SBP, Visit 20 (Month 72), n=61 | 0.5 (12.43)
  Standing SBP, Visit 21 (Month 76), n=43: number analyzed (Participants) | 43
  Standing SBP, Visit 21 (Month 76), n=43 | 3.5 (12.47)
  Standing SBP, Visit 22 (Month 80), n=37: number analyzed (Participants) | 37
  Standing SBP, Visit 22 (Month 80), n=37 | 0.9 (14.31)
  Standing SBP, Visit 23 (Month 84), n=32: number analyzed (Participants) | 32
  Standing SBP, Visit 23 (Month 84), n=32 | -0.8 (14.85)
  Standing SBP, Visit 24 (Month 88), n=29: number analyzed (Participants) | 29
  Standing SBP, Visit 24 (Month 88), n=29 | -0.6 (13.28)
  Standing SBP, Visit 25 (Month 92), n=25: number analyzed (Participants) | 25
  Standing SBP, Visit 25 (Month 92), n=25 | -1.6 (10.49)
  Standing SBP, Visit 26 (Month 96), n=26: number analyzed (Participants) | 26
  Standing SBP, Visit 26 (Month 96), n=26 | -0.2 (14.68)
  Standing SBP, Visit 27 (Month 100), n=20: number analyzed (Participants) | 20
  Standing SBP, Visit 27 (Month 100), n=20 | 0.0 (12.62)
  Standing SBP, Visit 28 (Month 104), n=17: number analyzed (Participants) | 17
  Standing SBP, Visit 28 (Month 104), n=17 | 2.9 (11.70)
  Standing SBP, Visit 29 (Month 108), n=13: number analyzed (Participants) | 13
  Standing SBP, Visit 29 (Month 108), n=13 | -2.2 (10.58)
  Standing SBP, Visit 30 (Month 112), n=4: number analyzed (Participants) | 4
  Standing SBP, Visit 30 (Month 112), n=4 | 1.8 (9.60)
  Standing SBP, Visit 31 (Month 116), n=3: number analyzed (Participants) | 3
  Standing SBP, Visit 31 (Month 116), n=3 | 9.0 (1.00)
  Standing SBP, Visit 32 (Month 120), n=1: number analyzed (Participants) | 1
  Standing SBP, Visit 32 (Month 120), n=1 | 10.0 (NA) — Standard deviation could not be calculated as only 1 participant was analyzed.
  Standing SBP, Follow up, n=267: number analyzed (Participants) | 267
  Standing SBP, Follow up, n=267 | 1.4 (14.59)

5. Primary Outcome: Change From Baseline in Heart Rate (HR) Measurements in the Supine and Standing Position
Description: Vital sign measurement HR was obtained throughout the study at all visits during the Open-Label Treatment Phase of the study. Evaluations of HR was performed supine at each study visit, and again after the participant had been standing for approximately 2 minutes. Baseline assessment in this OLE study was defined as the last assessment of that endpoint in VRX-RET-E22-302 taken prior to the first active treatment with retigabine. Change from Baseline was calculated by subtracting the Baseline value from the post Baseline values. NA indicates standard deviation could not be calculated as only 1 participant was analyzed. Only those participants with data available at the specified time points were analyzed (represented by n=X in the category titles).
Time Frame: Baseline and up to 122 months
Population: Safety Population
Measure: Mean (Standard Deviation); unit: Beats per minute
Arm/Group | Retigabine
Number analyzed (Participants) | 376
Beats per minute
  Supine HR, Visit 1 (Month 1), n=358: number analyzed (Participants) | 358
  Supine HR, Visit 1 (Month 1), n=358 | -0.4 (9.89)
  Supine HR, Visit 2 (Month 3), n=328: number analyzed (Participants) | 328
  Supine HR, Visit 2 (Month 3), n=328 | -0.5 (9.93)
  Supine HR, Visit 3 (Month 6), n=287: number analyzed (Participants) | 287
  Supine HR, Visit 3 (Month 6), n=287 | 0.1 (9.62)
  Supine HR, Visit 4 (Month 9), n=252: number analyzed (Participants) | 252
  Supine HR, Visit 4 (Month 9), n=252 | 0.7 (9.69)
  Supine HR, Visit 5 (Month 12), n=235: number analyzed (Participants) | 235
  Supine HR, Visit 5 (Month 12), n=235 | 0.0 (9.83)
  Supine HR, Visit 6 (Month 16), n=202: number analyzed (Participants) | 202
  Supine HR, Visit 6 (Month 16), n=202 | 1.8 (10.56)
  Supine HR, Visit 7 (Month 20), n=181: number analyzed (Participants) | 181
  Supine HR, Visit 7 (Month 20), n=181 | 2.3 (11.87)
  Supine HR, Visit 8 (Month 24), n=167: number analyzed (Participants) | 167
  Supine HR, Visit 8 (Month 24), n=167 | 1.9 (10.28)
  Supine HR, Visit 9 (Month 28), n=147: number analyzed (Participants) | 147
  Supine HR, Visit 9 (Month 28), n=147 | 2.7 (10.86)
  Supine HR, Visit 10 (Month 32), n=128: number analyzed (Participants) | 128
  Supine HR, Visit 10 (Month 32), n=128 | 3.0 (10.50)
  Supine HR, Visit 11 (Month 36), n=121: number analyzed (Participants) | 121
  Supine HR, Visit 11 (Month 36), n=121 | 0.8 (10.33)
  Supine HR, Visit 12 (Month 40), n=112: number analyzed (Participants) | 112
  Supine HR, Visit 12 (Month 40), n=112 | 3.3 (11.20)
  Supine HR, Visit 13 (Month 44), n=105: number analyzed (Participants) | 105
  Supine HR, Visit 13 (Month 44), n=105 | 1.8 (10.59)
  Supine HR, Visit 14 (Month 48), n=104: number analyzed (Participants) | 104
  Supine HR, Visit 14 (Month 48), n=104 | 1.0 (10.78)
  Supine HR, Visit 15 (Month 52), n=91: number analyzed (Participants) | 91
  Supine HR, Visit 15 (Month 52), n=91 | 2.0 (12.20)
  Supine HR, Visit 16 (Month 56), n=77: number analyzed (Participants) | 77
  Supine HR, Visit 16 (Month 56), n=77 | 2.5 (10.70)
  Supine HR, Visit 17 (Month 60), n=92: number analyzed (Participants) | 92
  Supine HR, Visit 17 (Month 60), n=92 | 0.9 (12.25)
  Supine HR, Visit 18 (Month 64), n=58: number analyzed (Participants) | 58
  Supine HR, Visit 18 (Month 64), n=58 | 5.5 (10.44)
  Supine HR, Visit 19 (Month 68), n=53: number analyzed (Participants) | 53
  Supine HR, Visit 19 (Month 68), n=53 | 2.4 (10.19)
  Supine HR, Visit 20 (Month 72), n=61: number analyzed (Participants) | 61
  Supine HR, Visit 20 (Month 72), n=61 | 2.1 (12.23)
  Supine HR, Visit 21 (Month 76), n=43: number analyzed (Participants) | 43
  Supine HR, Visit 21 (Month 76), n=43 | 2.8 (9.30)
  Supine HR, Visit 22 (Month 80), n=37: number analyzed (Participants) | 37
  Supine HR, Visit 22 (Month 80), n=37 | 5.1 (10.13)
  Supine HR, Visit 23 (Month 84), n=32: number analyzed (Participants) | 32
  Supine HR, Visit 23 (Month 84), n=32 | 3.5 (11.98)
  Supine HR, Visit 24 (Month 88), n=29: number analyzed (Participants) | 29
  Supine HR, Visit 24 (Month 88), n=29 | 3.2 (13.66)
  Supine HR, Visit 25 (Month 92), n=25: number analyzed (Participants) | 25
  Supine HR, Visit 25 (Month 92), n=25 | 3.9 (9.89)
  Supine HR, Visit 26 (Month 96), n=26: number analyzed (Participants) | 26
  Supine HR, Visit 26 (Month 96), n=26 | 2.1 (10.37)
  Supine HR, Visit 27 (Month 100), n=20: number analyzed (Participants) | 20
  Supine HR, Visit 27 (Month 100), n=20 | 3.1 (9.82)
  Supine HR, Visit 28 (Month 104), n=17: number analyzed (Participants) | 17
  Supine HR, Visit 28 (Month 104), n=17 | 3.3 (8.62)
  Supine HR, Visit 29 (Month 108), n=13: number analyzed (Participants) | 13
  Supine HR, Visit 29 (Month 108), n=13 | 0.5 (8.93)
  Supine HR, Visit 30 (Month 112), n=4: number analyzed (Participants) | 4
  Supine HR, Visit 30 (Month 112), n=4 | 3.8 (12.84)
  Supine HR, Visit 31 (Month 116), n=3: number analyzed (Participants) | 3
  Supine HR, Visit 31 (Month 116), n=3 | 7.7 (13.43)
  Supine HR, Visit 32 (Month 120), n=1: number analyzed (Participants) | 1
  Supine HR, Visit 32 (Month 120), n=1 | 11.0 (NA) — Standard deviation could not be calculated as only 1 participant was analyzed
  Supine HR, Follow up, n=267: number analyzed (Participants) | 267
  Supine HR, Follow up, n=267 | 2.1 (10.44)
  Standing HR, Visit 1 (Month 1), n=357: number analyzed (Participants) | 357
  Standing HR, Visit 1 (Month 1), n=357 | -0.1 (11.10)
  Standing HR, Visit 2 (Month 3), n=328: number analyzed (Participants) | 328
  Standing HR, Visit 2 (Month 3), n=328 | -0.2 (11.01)
  Standing HR, Visit 3 (Month 6), n=287: number analyzed (Participants) | 287
  Standing HR, Visit 3 (Month 6), n=287 | 0.3 (10.39)
  Standing HR, Visit 4 (Month 9), n=252: number analyzed (Participants) | 252
  Standing HR, Visit 4 (Month 9), n=252 | 1.7 (11.53)
  Standing HR, Visit 5 (Month 12), n=235: number analyzed (Participants) | 235
  Standing HR, Visit 5 (Month 12), n=235 | 0.1 (11.06)
  Standing HR, Visit 6 (Month 16), n=202: number analyzed (Participants) | 202
  Standing HR, Visit 6 (Month 16), n=202 | 1.6 (12.35)
  Standing HR, Visit 7 (Month 20), n=181: number analyzed (Participants) | 181
  Standing HR, Visit 7 (Month 20), n=181 | 1.4 (12.71)
  Standing HR, Visit 8 (Month 24), n=167: number analyzed (Participants) | 167
  Standing HR, Visit 8 (Month 24), n=167 | 1.9 (10.93)
  Standing HR, Visit 9 (Month 28), n=147: number analyzed (Participants) | 147
  Standing HR, Visit 9 (Month 28), n=147 | 1.6 (11.25)
  Standing HR, Visit 10 (Month 32), n=128: number analyzed (Participants) | 128
  Standing HR, Visit 10 (Month 32), n=128 | 2.2 (11.92)
  Standing HR, Visit 11 (Month 36), n=121: number analyzed (Participants) | 121
  Standing HR, Visit 11 (Month 36), n=121 | -0.6 (11.23)
  Standing HR, Visit 12 (Month 40), n=111: number analyzed (Participants) | 111
  Standing HR, Visit 12 (Month 40), n=111 | 2.6 (12.94)
  Standing HR, Visit 13 (Month 44), n=105: number analyzed (Participants) | 105
  Standing HR, Visit 13 (Month 44), n=105 | 2.8 (11.22)
  Standing HR, Visit 14 (Month 48), n=104: number analyzed (Participants) | 104
  Standing HR, Visit 14 (Month 48), n=104 | 0.8 (11.81)
  Standing HR, Visit 15 (Month 52), n=91: number analyzed (Participants) | 91
  Standing HR, Visit 15 (Month 52), n=91 | 3.1 (12.09)
  Standing HR, Visit 16 (Month 56), n=77: number analyzed (Participants) | 77
  Standing HR, Visit 16 (Month 56), n=77 | 1.3 (12.12)
  Standing HR, Visit 17 (Month 60), n=92: number analyzed (Participants) | 92
  Standing HR, Visit 17 (Month 60), n=92 | 0.6 (12.26)
  Standing HR, Visit 18 (Month 64), n=58: number analyzed (Participants) | 58
  Standing HR, Visit 18 (Month 64), n=58 | 4.6 (12.09)
  Standing HR, Visit 19 (Month 68), n=52: number analyzed (Participants) | 52
  Standing HR, Visit 19 (Month 68), n=52 | 1.3 (10.78)
  Standing HR, Visit 20 (Month 72), n=61: number analyzed (Participants) | 61
  Standing HR, Visit 20 (Month 72), n=61 | 0.7 (13.45)
  Standing HR, Visit 21 (Month 76), n=43: number analyzed (Participants) | 43
  Standing HR, Visit 21 (Month 76), n=43 | 0.3 (10.83)
  Standing HR, Visit 22 (Month 80), n=37: number analyzed (Participants) | 37
  Standing HR, Visit 22 (Month 80), n=37 | 2.9 (10.96)
  Standing HR, Visit 23 (Month 84), n=32: number analyzed (Participants) | 32
  Standing HR, Visit 23 (Month 84), n=32 | 2.3 (9.76)
  Standing HR, Visit 24 (Month 88), n=29: number analyzed (Participants) | 29
  Standing HR, Visit 24 (Month 88), n=29 | 2.4 (10.64)
  Standing HR, Visit 25 (Month 92), n=25: number analyzed (Participants) | 25
  Standing HR, Visit 25 (Month 92), n=25 | 3.6 (12.61)
  Standing HR, Visit 26 (Month 96), n=26: number analyzed (Participants) | 26
  Standing HR, Visit 26 (Month 96), n=26 | 3.1 (12.01)
  Standing HR, Visit 27 (Month 100), n=20: number analyzed (Participants) | 20
  Standing HR, Visit 27 (Month 100), n=20 | 5.2 (9.88)
  Syanding HR, Visit 28 (Month 104), n=17: number analyzed (Participants) | 17
  Syanding HR, Visit 28 (Month 104), n=17 | 6.2 (11.00)
  Standing HR, Visit 29 (Month 108), n=13: number analyzed (Participants) | 13
  Standing HR, Visit 29 (Month 108), n=13 | -0.2 (8.94)
  Standing HR, Visit 30 (Month 112), n=4: number analyzed (Participants) | 4
  Standing HR, Visit 30 (Month 112), n=4 | 2.3 (12.84)
  Standing HR, Visit 31 (Month 116), n=3: number analyzed (Participants) | 3
  Standing HR, Visit 31 (Month 116), n=3 | 7.3 (12.10)
  Standing HR, Visit 32 (Month 120), n=1: number analyzed (Participants) | 1
  Standing HR, Visit 32 (Month 120), n=1 | 10.0 (NA) — Standard deviation could not be calculated as only 1 participant was analyzed
  Standing HR, Follow up, n=267: number analyzed (Participants) | 267
  Standing HR, Follow up, n=267 | 2.2 (11.39)

6. Primary Outcome: Change From Baseline in Body Temperature
Description: Vital sign measurement temperature was obtained throughout the study at all visits during the Open-Label Treatment Phase of the study. Baseline assessment in this OLE study was defined as the last assessment of that endpoint in VRX-RET-E22-302 taken prior to the first active treatment with retigabine. Change from Baseline was calculated by subtracting the Baseline value from the post Baseline values. NA indicates standard deviation could not be calculated as only 1 participant was analyzed. Only those participants with data available at the specified time points were analyzed (represented by n=X in the category titles).
Time Frame: Baseline and up to 122 months
Population: Safety Population
Measure: Mean (Standard Deviation); unit: Degree Celsius
Arm/Group | Retigabine
Number analyzed (Participants) | 376
Degree Celsius
  Body temperature, Visit 1 (Month 1), n=350: number analyzed (Participants) | 350
  Body temperature, Visit 1 (Month 1), n=350 | 0.02 (0.386)
  Body temperature, Visit 2 (Month 3), n=318: number analyzed (Participants) | 318
  Body temperature, Visit 2 (Month 3), n=318 | 0.02 (0.358)
  Body temperature, Visit 3 (Month 6), n=280: number analyzed (Participants) | 280
  Body temperature, Visit 3 (Month 6), n=280 | 0.03 (0.384)
  Body temperature, Visit 4 (Month 9), n=244: number analyzed (Participants) | 244
  Body temperature, Visit 4 (Month 9), n=244 | 0.00 (0.380)
  Body temperature, Visit 5 (Month 12), n=229: number analyzed (Participants) | 229
  Body temperature, Visit 5 (Month 12), n=229 | 0.01 (0.392)
  Body temperature, Visit 6 (Month 16), n=197: number analyzed (Participants) | 197
  Body temperature, Visit 6 (Month 16), n=197 | 0.02 (0.362)
  Body temperature, Visit 7 (Month 20), n=176: number analyzed (Participants) | 176
  Body temperature, Visit 7 (Month 20), n=176 | 0.04 (0.381)
  Body temperature, Visit 8 (Month 24), n=161: number analyzed (Participants) | 161
  Body temperature, Visit 8 (Month 24), n=161 | 0.02 (0.387)
  Body temperature, Visit 9 (Month 28), n=143: number analyzed (Participants) | 143
  Body temperature, Visit 9 (Month 28), n=143 | 0.01 (0.407)
  Body temperature, Visit 10 (Month 32), n=125: number analyzed (Participants) | 125
  Body temperature, Visit 10 (Month 32), n=125 | 0.02 (0.362)
  Body temperature, Visit 11 (Month 36), n=118: number analyzed (Participants) | 118
  Body temperature, Visit 11 (Month 36), n=118 | 0.02 (0.385)
  Body temperature, Visit 12 (Month 40), n=109: number analyzed (Participants) | 109
  Body temperature, Visit 12 (Month 40), n=109 | 0.01 (0.404)
  Body temperature, Visit 13 (Month 44), n=101: number analyzed (Participants) | 101
  Body temperature, Visit 13 (Month 44), n=101 | 0.04 (0.387)
  Body temperature, Visit 14 (Month 48), n=100: number analyzed (Participants) | 100
  Body temperature, Visit 14 (Month 48), n=100 | 0.05 (0.382)
  Body temperature, Visit 15 (Month 52), n=88: number analyzed (Participants) | 88
  Body temperature, Visit 15 (Month 52), n=88 | -0.02 (0.396)
  Body temperature, Visit 16 (Month 56), n=74: number analyzed (Participants) | 74
  Body temperature, Visit 16 (Month 56), n=74 | -0.01 (0.393)
  Body temperature, Visit 17 (Month 60), n=89: number analyzed (Participants) | 89
  Body temperature, Visit 17 (Month 60), n=89 | 0.03 (0.391)
  Body temperature, Visit 18 (Month 64), n=58: number analyzed (Participants) | 58
  Body temperature, Visit 18 (Month 64), n=58 | -0.01 (0.306)
  Body temperature, Visit 19 (Month 68), n=53: number analyzed (Participants) | 53
  Body temperature, Visit 19 (Month 68), n=53 | 0.05 (0.318)
  Body temperature, Visit 20 (Month 72), n=59: number analyzed (Participants) | 59
  Body temperature, Visit 20 (Month 72), n=59 | 0.06 (0.373)
  Body temperature, Visit 21 (Month 76), n=42: number analyzed (Participants) | 42
  Body temperature, Visit 21 (Month 76), n=42 | 0.06 (0.306)
  Body temperature, Visit 22 (Month 80), n=37: number analyzed (Participants) | 37
  Body temperature, Visit 22 (Month 80), n=37 | -0.04 (0.362)
  Body temperature, Visit 23 (Month 84), n=32: number analyzed (Participants) | 32
  Body temperature, Visit 23 (Month 84), n=32 | 0.05 (0.324)
  Body temperature, Visit 24 (Month 88), n=29: number analyzed (Participants) | 29
  Body temperature, Visit 24 (Month 88), n=29 | -0.06 (0.313)
  Body temperature, Visit 25 (Month 92), n=25: number analyzed (Participants) | 25
  Body temperature, Visit 25 (Month 92), n=25 | 0.00 (0.289)
  Body temperature, Visit 26 (Month 96), n=26: number analyzed (Participants) | 26
  Body temperature, Visit 26 (Month 96), n=26 | -0.10 (0.299)
  Body temperature, Visit 27 (Month 100), n=20: number analyzed (Participants) | 20
  Body temperature, Visit 27 (Month 100), n=20 | -0.03 (0.285)
  Body temperature, Visit 28 (Month 104), n=17: number analyzed (Participants) | 17
  Body temperature, Visit 28 (Month 104), n=17 | -0.02 (0.326)
  Body temperature, Visit 29 (Month 108), n=13: number analyzed (Participants) | 13
  Body temperature, Visit 29 (Month 108), n=13 | 0.04 (0.275)
  Body temperature, Visit 30 (Month 112), n=4: number analyzed (Participants) | 4
  Body temperature, Visit 30 (Month 112), n=4 | -0.02 (0.126)
  Body temperature, Visit 31 (Month 116), n=3: number analyzed (Participants) | 3
  Body temperature, Visit 31 (Month 116), n=3 | -0.20 (0.200)
  Body temperature, Visit 32 (Month 120), n=1: number analyzed (Participants) | 1
  Body temperature, Visit 32 (Month 120), n=1 | 0.10 (NA) — Standard deviation could not be calculated as only 1 participant was analyzed
  Body temperature, Follow up, n=261: number analyzed (Participants) | 261
  Body temperature, Follow up, n=261 | 0.03 (0.397)

7. Primary Outcome: Change From Baseline in Body Weight
Description: Weight in pounds or kilograms was measured in ordinary indoor clothing (without shoes) and was recorded at all study visits during the Open-Label Treatment Phase of the study. Baseline assessment in this OLE study was defined as the last assessment of that endpoint in VRX-RET-E22-302 taken prior to the first active treatment with retigabine. Change from Baseline was calculated by subtracting the Baseline value from the post Baseline values. NA indicates standard deviation could not be calculated as only 1 participant was analyzed. Only those participants with data available at the specified time points were analyzed (represented by n=X in the category titles).
Time Frame: Baseline and up to 122 months
Population: Safety Population
Measure: Mean (Standard Deviation); unit: Kilograms
Arm/Group | Retigabine
Number analyzed (Participants) | 376
Kilograms
  Body weight, Visit 1 (Month 1), n=356: number analyzed (Participants) | 356
  Body weight, Visit 1 (Month 1), n=356 | 1.19 (3.125)
  Body weight, Visit 2 (Month 3), n=325: number analyzed (Participants) | 325
  Body weight, Visit 2 (Month 3), n=325 | 1.37 (3.630)
  Body weight, Visit 3 (Month 6), n=287: number analyzed (Participants) | 287
  Body weight, Visit 3 (Month 6), n=287 | 1.51 (4.528)
  Body weight, Visit 4 (Month 9), n=252: number analyzed (Participants) | 252
  Body weight, Visit 4 (Month 9), n=252 | 1.08 (5.068)
  Body weight, Visit 5 (Month 12), n=235: number analyzed (Participants) | 235
  Body weight, Visit 5 (Month 12), n=235 | 1.56 (4.764)
  Body weight, Visit 6 (Month 16), n=202: number analyzed (Participants) | 202
  Body weight, Visit 6 (Month 16), n=202 | 1.98 (5.382)
  Body weight, Visit 7 (Month 20), n=181: number analyzed (Participants) | 181
  Body weight, Visit 7 (Month 20), n=181 | 1.79 (5.762)
  Body weight, Visit 8 (Month 24), n=167: number analyzed (Participants) | 167
  Body weight, Visit 8 (Month 24), n=167 | 1.20 (6.571)
  Body weight, Visit 9 (Month 28), n=147: number analyzed (Participants) | 147
  Body weight, Visit 9 (Month 28), n=147 | 1.67 (6.101)
  Body weight, Visit 10 (Month 32), n=128: number analyzed (Participants) | 128
  Body weight, Visit 10 (Month 32), n=128 | 1.75 (7.103)
  Body weight, Visit 11 (Month 36), n=121: number analyzed (Participants) | 121
  Body weight, Visit 11 (Month 36), n=121 | 2.07 (7.151)
  Body weight, Visit 12 (Month 40), 112: number analyzed (Participants) | 112
  Body weight, Visit 12 (Month 40), 112 | 2.12 (7.077)
  Body weight, Visit 13 (Month 44), n=105: number analyzed (Participants) | 105
  Body weight, Visit 13 (Month 44), n=105 | 1.09 (7.469)
  Body weight, Visit 14 (Month 48), n=104: number analyzed (Participants) | 104
  Body weight, Visit 14 (Month 48), n=104 | 1.08 (8.007)
  Body weight, Visit 15 (Month 52), n=91: number analyzed (Participants) | 91
  Body weight, Visit 15 (Month 52), n=91 | 0.66 (7.539)
  Body weight, Visit 16 (Month 56), n=77: number analyzed (Participants) | 77
  Body weight, Visit 16 (Month 56), n=77 | 0.71 (7.248)
  Body weight, Visit 17 (Month 60), n=91: number analyzed (Participants) | 91
  Body weight, Visit 17 (Month 60), n=91 | 1.31 (8.082)
  Body weight, Visit 18 (Month 64), n=58: number analyzed (Participants) | 58
  Body weight, Visit 18 (Month 64), n=58 | 1.32 (7.541)
  Body weight, Visit 19 (Month 68), n=53: number analyzed (Participants) | 53
  Body weight, Visit 19 (Month 68), n=53 | 1.49 (8.036)
  Body weight, Visit 20 (Month 72), n=61: number analyzed (Participants) | 61
  Body weight, Visit 20 (Month 72), n=61 | 1.65 (8.774)
  Body weight, Visit 21 (Month 76), n=43: number analyzed (Participants) | 43
  Body weight, Visit 21 (Month 76), n=43 | 1.71 (9.355)
  Body weight, Visit 22 (Month 80), n=37: number analyzed (Participants) | 37
  Body weight, Visit 22 (Month 80), n=37 | 2.30 (9.311)
  Body weight, Visit 23 (Month 84), n=32: number analyzed (Participants) | 32
  Body weight, Visit 23 (Month 84), n=32 | 2.00 (9.522)
  Body weight, Visit 24 (Month 88), n=29: number analyzed (Participants) | 29
  Body weight, Visit 24 (Month 88), n=29 | 1.12 (9.633)
  Body weight, Visit 25 (Month 92), n=25: number analyzed (Participants) | 25
  Body weight, Visit 25 (Month 92), n=25 | 0.83 (10.845)
  Body weight, Visit 26 (Month 96), n=26: number analyzed (Participants) | 26
  Body weight, Visit 26 (Month 96), n=26 | 0.12 (14.470)
  Body weight, Visit 27 (Month 100), n=20: number analyzed (Participants) | 20
  Body weight, Visit 27 (Month 100), n=20 | 1.57 (11.382)
  Body weight, Visit 28 (Month 104), n=17: number analyzed (Participants) | 17
  Body weight, Visit 28 (Month 104), n=17 | 1.62 (10.715)
  Body weight, Visit 29 (Month 108), n=13: number analyzed (Participants) | 13
  Body weight, Visit 29 (Month 108), n=13 | 2.32 (13.914)
  Body weight, Visit 30 (Month 112), n=4: number analyzed (Participants) | 4
  Body weight, Visit 30 (Month 112), n=4 | 4.85 (17.693)
  Body weight, Visit 31 (Month 116), n=3: number analyzed (Participants) | 3
  Body weight, Visit 31 (Month 116), n=3 | 9.73 (17.234)
  Body weight, Visit 32 (Month 120), n=1: number analyzed (Participants) | 1
  Body weight, Visit 32 (Month 120), n=1 | 0.50 (NA) — Standard deviation could not be calculated as only 1 participant was analyzed.
  Body weight, Follow up, n=267: number analyzed (Participants) | 267
  Body weight, Follow up, n=267 | 1.34 (5.870)

8. Primary Outcome: Change From Baseline in Electocardiogram (ECG) Parameters PR, QRS, QT, Corrected QT Interval (QTc) Bazett and QTc Friedericia
Description: A 12-lead ECG was performed at all study visits during the Open-Label Treatment Phase during the first year of the open-label extension study (Months 1, 3, 6, 9, 12) and at the end of each 12 month study cycle that the participant was enrolled (i.e., second year, third year, fourth year, etc.). The ECG parameters that were assessed were PR interval, QRS interval, QRS duration, QT interval, and QTc interval. QT intervals were corrected using both Bazett's and Friedericia's formulas. Baseline assessment in this OLE study was defined as the last assessment of that endpoint in VRX-RET-E22-302 taken prior to the first active treatment with retigabine. Change from Baseline was calculated by subtracting the Baseline value from the post Baseline values. NA indicates standard deviation could not be calculated as only 1 participant was analyzed. Only those participants with data available at the specified time points were analyzed (represented by n=X in the category titles).
Time Frame: Baseline and up to 122 months
Population: Safety Population
Measure: Mean (Standard Deviation); unit: Milliseconds
Arm/Group | Retigabine
Number analyzed (Participants) | 376
Milliseconds
  PR interval, Visit 1 (Month 1), n=355: number analyzed (Participants) | 355
  PR interval, Visit 1 (Month 1), n=355 | 0.1 (13.47)
  PR interval, Visit 2 (Month 3), n=324: number analyzed (Participants) | 324
  PR interval, Visit 2 (Month 3), n=324 | -0.4 (11.95)
  PR interval, Visit 3 (Month 6), n=278: number analyzed (Participants) | 278
  PR interval, Visit 3 (Month 6), n=278 | -1.0 (13.18)
  PR interval, Visit 4 (Month 9), n=245: number analyzed (Participants) | 245
  PR interval, Visit 4 (Month 9), n=245 | -1.7 (12.74)
  PR interval, Visit 5 (Month 12), n=233: number analyzed (Participants) | 233
  PR interval, Visit 5 (Month 12), n=233 | -1.7 (13.01)
  PR interval, Visit 8 (Month 24), n=158: number analyzed (Participants) | 158
  PR interval, Visit 8 (Month 24), n=158 | -2.1 (15.23)
  PR interval, Visit 11 (Month 36), n=113: number analyzed (Participants) | 113
  PR interval, Visit 11 (Month 36), n=113 | -1.6 (14.20)
  PR interval, Visit 14 (Month 48), n=98: number analyzed (Participants) | 98
  PR interval, Visit 14 (Month 48), n=98 | 0.3 (13.30)
  PR interval, Visit 17 (Month 60), n=87: number analyzed (Participants) | 87
  PR interval, Visit 17 (Month 60), n=87 | 0.7 (13.70)
  PR interval, Visit 20 (Month 72), n=52: number analyzed (Participants) | 52
  PR interval, Visit 20 (Month 72), n=52 | 0.9 (14.07)
  PR interval, Visit 23 (Month 84), n=30: number analyzed (Participants) | 30
  PR interval, Visit 23 (Month 84), n=30 | -3.5 (13.06)
  PR interval, Visit 26 (Month 96), n=22: number analyzed (Participants) | 22
  PR interval, Visit 26 (Month 96), n=22 | -4.4 (11.96)
  PR interval, Visit 29 (Month 108), n=13: number analyzed (Participants) | 13
  PR interval, Visit 29 (Month 108), n=13 | -1.9 (11.50)
  PR interval, Visit 32 (Month 120), n=1: number analyzed (Participants) | 1
  PR interval, Visit 32 (Month 120), n=1 | -23.7 (NA) — Standard deviation could not be calculated as only 1 participant was analyzed.
  PR interval, Follow up, n=252: number analyzed (Participants) | 252
  PR interval, Follow up, n=252 | -1.3 (12.83)
  QRS duration, Visit 1 (Month 1), n=357: number analyzed (Participants) | 357
  QRS duration, Visit 1 (Month 1), n=357 | -0.6 (8.03)
  QRS duration, Visit 2 (Month 3), n=327: number analyzed (Participants) | 327
  QRS duration, Visit 2 (Month 3), n=327 | -1.1 (7.53)
  QRS duration, Visit 3 (Month 6), n=282: number analyzed (Participants) | 282
  QRS duration, Visit 3 (Month 6), n=282 | -1.2 (7.34)
  QRS duration, Visit 4 (Month 9), n=249: number analyzed (Participants) | 249
  QRS duration, Visit 4 (Month 9), n=249 | -1.4 (6.59)
  QRS duration, Visit 5 (Month 12), n=235: number analyzed (Participants) | 235
  QRS duration, Visit 5 (Month 12), n=235 | -0.1 (8.09)
  QRS duration, Visit 8 (Month 24), n=160: number analyzed (Participants) | 160
  QRS duration, Visit 8 (Month 24), n=160 | -1.1 (7.74)
  QRS duration, Visit 11 (Month 36), n=116: number analyzed (Participants) | 116
  QRS duration, Visit 11 (Month 36), n=116 | 1.5 (7.66)
  QRS duration, Visit 14 (Month 48), n=99: number analyzed (Participants) | 99
  QRS duration, Visit 14 (Month 48), n=99 | 1.1 (7.92)
  QRS duration, Visit 17 (Month 60), n=89: number analyzed (Participants) | 89
  QRS duration, Visit 17 (Month 60), n=89 | 3.3 (12.89)
  QRS duration, Visit 20 (Month 72), n=56: number analyzed (Participants) | 56
  QRS duration, Visit 20 (Month 72), n=56 | 5.2 (16.42)
  QRS duration, Visit 23 (Month 84), n=32: number analyzed (Participants) | 32
  QRS duration, Visit 23 (Month 84), n=32 | 3.4 (18.65)
  QRS duration Visit 26 (Month 96), n=23: number analyzed (Participants) | 23
  QRS duration Visit 26 (Month 96), n=23 | 3.5 (24.77)
  QRS duration, Visit 29 (Month 108), n=13: number analyzed (Participants) | 13
  QRS duration, Visit 29 (Month 108), n=13 | 1.2 (7.73)
  QRS duration, Visit 32 (Month 120), n=1: number analyzed (Participants) | 1
  QRS duration, Visit 32 (Month 120), n=1 | 10.7 (NA) — Standard deviation could not be calculated as only 1 participant was analyzed.
  QRS duration, Follow up, n=254: number analyzed (Participants) | 254
  QRS duration, Follow up, n=254 | -0.1 (8.74)
  QT interval, Visit 1 (Month 1), n=357: number analyzed (Participants) | 357
  QT interval, Visit 1 (Month 1), n=357 | 5.5 (23.66)
  QT interval, Visit 2 (Month 3), n=324: number analyzed (Participants) | 324
  QT interval, Visit 2 (Month 3), n=324 | 4.8 (23.35)
  QT interval, Visit 3 (Month 6), n=278: number analyzed (Participants) | 278
  QT interval, Visit 3 (Month 6), n=278 | 5.3 (23.10)
  QT interval, Visit 4 (Month 9), n=246: number analyzed (Participants) | 246
  QT interval, Visit 4 (Month 9), n=246 | 3.9 (23.47)
  QT interval, Visit 5 (Month 12), n=232: number analyzed (Participants) | 232
  QT interval, Visit 5 (Month 12), n=232 | 5.0 (24.37)
  QT interval, Visit 8 (Month 24), n=157: number analyzed (Participants) | 157
  QT interval, Visit 8 (Month 24), n=157 | 3.4 (25.09)
  QT interval, Visit 11 (Month 36), n=112: number analyzed (Participants) | 112
  QT interval, Visit 11 (Month 36), n=112 | 8.8 (24.66)
  QT interval, Visit 14 (Month 48), n=96: number analyzed (Participants) | 96
  QT interval, Visit 14 (Month 48), n=96 | 7.0 (22.57)
  QT interval, Visit 17 (Month 60), n=89: number analyzed (Participants) | 89
  QT interval, Visit 17 (Month 60), n=89 | 7.9 (23.55)
  QT interval, Visit 20 (Month 72), n=56: number analyzed (Participants) | 56
  QT interval, Visit 20 (Month 72), n=56 | 12.4 (28.30)
  QT interval, Visit 23 (Month 84), n=32: number analyzed (Participants) | 32
  QT interval, Visit 23 (Month 84), n=32 | 8.4 (30.17)
  QT interval, Visit 26 (Month 96), n=23: number analyzed (Participants) | 23
  QT interval, Visit 26 (Month 96), n=23 | 4.0 (31.01)
  QT interval, Visit 29 (Month 108), n=13: number analyzed (Participants) | 13
  QT interval, Visit 29 (Month 108), n=13 | 0.8 (29.90)
  QT interval, Visit 32 (Month 120), n=1: number analyzed (Participants) | 1
  QT interval, Visit 32 (Month 120), n=1 | 64.0 (NA) — Standard deviation could not be calculated as only 1 participant was analyzed.
  QT interval, Follow up, n=254: number analyzed (Participants) | 254
  QT interval, Follow up, n=254 | 1.2 (24.95)
  QTc Bazett interval, Visit 1 (Month 1, n=357: number analyzed (Participants) | 357
  QTc Bazett interval, Visit 1 (Month 1, n=357 | 1.2 (18.07)
  QTc Bazett interval, Visit 2 (Month 3), n=324: number analyzed (Participants) | 324
  QTc Bazett interval, Visit 2 (Month 3), n=324 | 1.6 (18.09)
  QTc Bazett interval, Visit 3 (Month 6), n=278: number analyzed (Participants) | 278
  QTc Bazett interval, Visit 3 (Month 6), n=278 | 3.4 (16.97)
  QTc Bazett interval, Visit 4 (Month 9, n=246: number analyzed (Participants) | 246
  QTc Bazett interval, Visit 4 (Month 9, n=246 | 4.4 (17.33)
  QTc Bazett interval, Visit 5 (Month 12), n=232: number analyzed (Participants) | 232
  QTc Bazett interval, Visit 5 (Month 12), n=232 | 2.3 (16.61)
  QTc Bazett interval, Visit 8 (Month 24), n=157: number analyzed (Participants) | 157
  QTc Bazett interval, Visit 8 (Month 24), n=157 | 6.6 (18.27)
  QTc Bazett interval, Visit 11 (Month 36), n=112: number analyzed (Participants) | 112
  QTc Bazett interval, Visit 11 (Month 36), n=112 | 4.5 (18.10)
  QTc Bazett interval, Visit 14 (Month 48), n=96: number analyzed (Participants) | 96
  QTc Bazett interval, Visit 14 (Month 48), n=96 | 5.6 (18.18)
  QTc Bazett interval, Visit 17 (Month 60), n=89: number analyzed (Participants) | 89
  QTc Bazett interval, Visit 17 (Month 60), n=89 | 12.4 (25.68)
  QTc Bazett interval, Visit 20 (Month 72), n=56: number analyzed (Participants) | 56
  QTc Bazett interval, Visit 20 (Month 72), n=56 | 15.6 (24.79)
  QTc Bazett interval, Visit 23 (Month 84), n=32: number analyzed (Participants) | 32
  QTc Bazett interval, Visit 23 (Month 84), n=32 | 18.7 (23.90)
  QTc Bazett interval, Visit 26 (Month 96, n=23: number analyzed (Participants) | 23
  QTc Bazett interval, Visit 26 (Month 96, n=23 | 19.7 (28.67)
  QTc Bazett interval, Visit 29 (Month 108), n=13: number analyzed (Participants) | 13
  QTc Bazett interval, Visit 29 (Month 108), n=13 | 17.6 (21.09)
  QTc Bazett interval, Visit 32 (Month 120), n=1: number analyzed (Participants) | 1
  QTc Bazett interval, Visit 32 (Month 120), n=1 | 0.7 (NA) — Standard deviation could not be calculated as only 1 participant was analyzed.
  QTc Bazett interval, Follow up, n=254: number analyzed (Participants) | 254
  QTc Bazett interval, Follow up, n=254 | 4.9 (18.39)
  QTc Friedericia interval, Visit 1 (Month 1),n=357: number analyzed (Participants) | 357
  QTc Friedericia interval, Visit 1 (Month 1),n=357 | 2.7 (15.72)
  QTc Friedericia interval Visit 2 (Month 3),n=324: number analyzed (Participants) | 324
  QTc Friedericia interval Visit 2 (Month 3),n=324 | 2.7 (15.88)
  QTc Friedericia interval,Visit 3 (Month 6),n=278: number analyzed (Participants) | 278
  QTc Friedericia interval,Visit 3 (Month 6),n=278 | 4.0 (15.59)
  QTc Friedericia interval, Visit 4 (Month 9),n=246: number analyzed (Participants) | 246
  QTc Friedericia interval, Visit 4 (Month 9),n=246 | 4.1 (15.86)
  QTc Friedericia intervalVisit 5 (Month 12),n=232: number analyzed (Participants) | 232
  QTc Friedericia intervalVisit 5 (Month 12),n=232 | 3.2 (15.62)
  QTc Friedericia interval,Visit 8 (Month 24),n=157: number analyzed (Participants) | 157
  QTc Friedericia interval,Visit 8 (Month 24),n=157 | 5.4 (15.00)
  QTc Friedericia intervalVisit 11 (Month 36),n=112: number analyzed (Participants) | 112
  QTc Friedericia intervalVisit 11 (Month 36),n=112 | 5.9 (15.69)
  QTc Friedericia interval,Visit 14 (Month 48),n=96: number analyzed (Participants) | 96
  QTc Friedericia interval,Visit 14 (Month 48),n=96 | 6.1 (15.08)
  QTc Friedericia interval,Visit 17 (Month 60),n=89: number analyzed (Participants) | 89
  QTc Friedericia interval,Visit 17 (Month 60),n=89 | 10.8 (18.93)
  QTc Friedericia intervalVisit 20 (Month 72),n=56: number analyzed (Participants) | 56
  QTc Friedericia intervalVisit 20 (Month 72),n=56 | 14.4 (19.28)
  QTc Friedericia intervalVisit 23 (Month 84),n=32: number analyzed (Participants) | 32
  QTc Friedericia intervalVisit 23 (Month 84),n=32 | 15.0 (20.97)
  QTc Friedericia interval,Visit 26 (Month 96),n=23: number analyzed (Participants) | 23
  QTc Friedericia interval,Visit 26 (Month 96),n=23 | 14.3 (22.90)
  QTcFriedericia intervalVisit 29 (Month 108)n=13: number analyzed (Participants) | 13
  QTcFriedericia intervalVisit 29 (Month 108)n=13 | 11.6 (17.76)
  QTc Friedericia interval,Visit 32 (Month 120),n=1: number analyzed (Participants) | 1
  QTc Friedericia interval,Visit 32 (Month 120),n=1 | 23.7 (NA) — Standard deviation could not be calculated as only 1 participant was analyzed.
  QTcFriedericia interval, Follow up,n=254: number analyzed (Participants) | 254
  QTcFriedericia interval, Follow up,n=254 | 3.5 (16.58)

9. Primary Outcome: Change From Baseline in Alkaline Phosphatase (Alk. Phos.), Alanine Amino Transferase (ALT) and Aspartate Amino Transferase (AST)
Description: Clinical chemistry parameters included Alk. Phos., ALT and AST. The clinical laboratory evaluations were performed at all study visits during the Open-Label Treatment Phase. Baseline assessment in this OLE study was defined as the last assessment of that endpoint in VRX-RET-E22-302 taken prior to the first active treatment with retigabine. Change from Baseline was calculated by subtracting the Baseline value from the post Baseline values. NA indicates standard deviation could not be calculated as only 1 participant was analyzed. Only those participants with data available at the specified time points were analyzed (represented by n=X in the category titles).
Time Frame: Baseline and up to 122 months
Population: Safety Population
Measure: Mean (Standard Deviation); unit: International units per liter
Arm/Group | Retigabine
Number analyzed (Participants) | 376
International units per liter
  Alk. Phos., Visit 1 (Month 1), n=352: number analyzed (Participants) | 352
  Alk. Phos., Visit 1 (Month 1), n=352 | -0.9 (14.47)
  Alk. Phos., Visit 1a (Month 2), n=1: number analyzed (Participants) | 1
  Alk. Phos., Visit 1a (Month 2), n=1 | -18.0 (NA) — Standard deviation could not be calculated as only 1 participant was analyzed.
  Alk. Phos., Visit 2 (Month 3), n=322: number analyzed (Participants) | 322
  Alk. Phos., Visit 2 (Month 3), n=322 | -1.5 (14.56)
  Alk. Phos., Visit 2a (Month 4), n=1: number analyzed (Participants) | 1
  Alk. Phos., Visit 2a (Month 4), n=1 | 4.0 (NA) — Standard deviation could not be calculated as only 1 participant was analyzed.
  Alk. Phos., Visit 3 (Month 6), n=279: number analyzed (Participants) | 279
  Alk. Phos., Visit 3 (Month 6), n=279 | -1.2 (14.91)
  Alk. Phos., Visit 4 (Month 9), n=248: number analyzed (Participants) | 248
  Alk. Phos., Visit 4 (Month 9), n=248 | -3.0 (14.25)
  Alk. Phos., Visit 5 (Month 12), n=228: number analyzed (Participants) | 228
  Alk. Phos., Visit 5 (Month 12), n=228 | -1.9 (15.06)
  Alk. Phos., Visit 6 (Month 16), n=200: number analyzed (Participants) | 200
  Alk. Phos., Visit 6 (Month 16), n=200 | -1.8 (15.96)
  Alk. Phos., Visit 7 (Month 20), n=176: number analyzed (Participants) | 176
  Alk. Phos., Visit 7 (Month 20), n=176 | -3.6 (17.32)
  Alk. Phos., Visit 8 (Month 24), n=163: number analyzed (Participants) | 163
  Alk. Phos., Visit 8 (Month 24), n=163 | -4.0 (17.68)
  Alk. Phos., Visit 9 (Month 28), n=142: number analyzed (Participants) | 142
  Alk. Phos., Visit 9 (Month 28), n=142 | -3.1 (17.88)
  Alk. Phos., Visit 10 (Month 32), n=126: number analyzed (Participants) | 126
  Alk. Phos., Visit 10 (Month 32), n=126 | -4.6 (18.94)
  Alk. Phos., Visit 11 (Month 36), n=116: number analyzed (Participants) | 116
  Alk. Phos., Visit 11 (Month 36), n=116 | -6.2 (22.36)
  Alk. Phos., Visit 12 (Month 40), n=108: number analyzed (Participants) | 108
  Alk. Phos., Visit 12 (Month 40), n=108 | -4.8 (21.05)
  Alk. Phos., Visit 13 (Month 44), n=101: number analyzed (Participants) | 101
  Alk. Phos., Visit 13 (Month 44), n=101 | -5.8 (21.53)
  Alk. Phos., Visit 14 (Month 48), n=101: number analyzed (Participants) | 101
  Alk. Phos., Visit 14 (Month 48), n=101 | -7.2 (21.34)
  Alk. Phos., Visit 15 (Month 52), n=88: number analyzed (Participants) | 88
  Alk. Phos., Visit 15 (Month 52), n=88 | -2.5 (23.46)
  Alk. Phos., Visit 16 (Month 56), n=76: number analyzed (Participants) | 76
  Alk. Phos., Visit 16 (Month 56), n=76 | -0.1 (19.72)
  Alk. Phos., Visit 17 (Month 60), n=90: number analyzed (Participants) | 90
  Alk. Phos., Visit 17 (Month 60), n=90 | -5.1 (21.15)
  Alk. Phos., Visit 18 (Month 64), n=55: number analyzed (Participants) | 55
  Alk. Phos., Visit 18 (Month 64), n=55 | -2.0 (18.95)
  Alk. Phos., Visit 19 (Month 68), n=50: number analyzed (Participants) | 50
  Alk. Phos., Visit 19 (Month 68), n=50 | -0.6 (14.60)
  Alk. Phos., Visit 20 (Month 72), n=58: number analyzed (Participants) | 58
  Alk. Phos., Visit 20 (Month 72), n=58 | 0.3 (23.56)
  Alk. Phos., Visit 21 (Month 76), n=40: number analyzed (Participants) | 40
  Alk. Phos., Visit 21 (Month 76), n=40 | 0.8 (15.41)
  Alk. Phos., Visit 22 (Month 80), n=35: number analyzed (Participants) | 35
  Alk. Phos., Visit 22 (Month 80), n=35 | 3.2 (19.97)
  Alk. Phos., Visit 23 (Month 84), n=32: number analyzed (Participants) | 32
  Alk. Phos., Visit 23 (Month 84), n=32 | 0.2 (16.54)
  Alk. Phos., Visit 24 (Month 88), n=28: number analyzed (Participants) | 28
  Alk. Phos., Visit 24 (Month 88), n=28 | -0.1 (19.55)
  Alk. Phos., Visit 25 (Month 92), n=25: number analyzed (Participants) | 25
  Alk. Phos., Visit 25 (Month 92), n=25 | 1.5 (21.27)
  Alk. Phos., Visit 26 (Month 96), n=26: number analyzed (Participants) | 26
  Alk. Phos., Visit 26 (Month 96), n=26 | 4.8 (23.10)
  Alk. Phos., Visit 27 (Month 100), n=20: number analyzed (Participants) | 20
  Alk. Phos., Visit 27 (Month 100), n=20 | 4.1 (14.67)
  Alk. Phos., Visit 28 (Month 104), n=16: number analyzed (Participants) | 16
  Alk. Phos., Visit 28 (Month 104), n=16 | 8.6 (21.80)
  Alk. Phos., Visit 29 (Month 108), n=13: number analyzed (Participants) | 13
  Alk. Phos., Visit 29 (Month 108), n=13 | 6.6 (17.94)
  Alk. Phos., Visit 30 (Month 112), n=4: number analyzed (Participants) | 4
  Alk. Phos., Visit 30 (Month 112), n=4 | 1.8 (14.57)
  Alk. Phos., Visit 31 (Month 116), n=3: number analyzed (Participants) | 3
  Alk. Phos., Visit 31 (Month 116), n=3 | 3.0 (3.61)
  Alk. Phos., Visit 32 (Month 120), n=1: number analyzed (Participants) | 1
  Alk. Phos., Visit 32 (Month 120), n=1 | 1.0 (NA) — Standard deviation could not be calculated as only 1 participant was analyzed.
  Alk. Phos., Follow up, n=261: number analyzed (Participants) | 261
  Alk. Phos., Follow up, n=261 | -0.4 (18.15)
  ALT, Visit 1 (Month 1), n=352: number analyzed (Participants) | 352
  ALT, Visit 1 (Month 1), n=352 | 2.6 (20.05)
  ALT, Visit 1a (Month 2), n=1: number analyzed (Participants) | 1
  ALT, Visit 1a (Month 2), n=1 | -24.0 (NA) — Standard deviation could not be calculated as only 1 participant was analyzed.
  ALT, Visit 2 (Month 3), n=322: number analyzed (Participants) | 322
  ALT, Visit 2 (Month 3), n=322 | 1.5 (16.57)
  ALT, Visit 2a (Month 4), n=1: number analyzed (Participants) | 1
  ALT, Visit 2a (Month 4), n=1 | 45.0 (NA) — Standard deviation could not be calculated as only 1 participant was analyzed.
  ALT, Visit 3 (Month 6), n=278: number analyzed (Participants) | 278
  ALT, Visit 3 (Month 6), n=278 | 1.3 (13.99)
  ALT, Visit 4 (Month 9), n=246: number analyzed (Participants) | 246
  ALT, Visit 4 (Month 9), n=246 | -0.2 (10.94)
  ALT, Visit 5 (Month 12), n=227: number analyzed (Participants) | 227
  ALT, Visit 5 (Month 12), n=227 | 3.4 (28.91)
  ALT, Visit 6 (Month 16), n=200: number analyzed (Participants) | 200
  ALT, Visit 6 (Month 16), n=200 | 1.3 (12.56)
  ALT, Visit 7 (Month 20), n=174: number analyzed (Participants) | 174
  ALT, Visit 7 (Month 20), n=174 | 1.2 (17.23)
  ALT, Visit 8 (Month 24), n=163: number analyzed (Participants) | 163
  ALT, Visit 8 (Month 24), n=163 | 0.5 (11.03)
  ALT, Visit 9 (Month 28), n=141: number analyzed (Participants) | 141
  ALT, Visit 9 (Month 28), n=141 | 1.7 (16.40)
  ALT, Visit 10 (Month 32), n=126: number analyzed (Participants) | 126
  ALT, Visit 10 (Month 32), n=126 | 1.0 (9.95)
  ALT, Visit 11 (Month 36), n=115: number analyzed (Participants) | 115
  ALT, Visit 11 (Month 36), n=115 | 0.1 (8.11)
  ALT, Visit 12 (Month 40), n=107: number analyzed (Participants) | 107
  ALT, Visit 12 (Month 40), n=107 | 0.9 (8.49)
  ALT, Visit 13 (Month 44), n=101: number analyzed (Participants) | 101
  ALT, Visit 13 (Month 44), n=101 | 0.6 (8.39)
  ALT, Visit 14 (Month 48), n=99: number analyzed (Participants) | 99
  ALT, Visit 14 (Month 48), n=99 | 0.5 (8.47)
  ALT, Visit 15 (Month 52), n=88: number analyzed (Participants) | 88
  ALT, Visit 15 (Month 52), n=88 | 0.9 (9.83)
  ALT, Visit 16 (Month 56), n=75: number analyzed (Participants) | 75
  ALT, Visit 16 (Month 56), n=75 | 1.3 (9.16)
  ALT, Visit 17 (Month 60), n=89: number analyzed (Participants) | 89
  ALT, Visit 17 (Month 60), n=89 | 0.0 (8.06)
  ALT, Visit 18 (Month 64), n=54: number analyzed (Participants) | 54
  ALT, Visit 18 (Month 64), n=54 | -0.8 (7.12)
  ALT, Visit 19 (Month 68), n=50: number analyzed (Participants) | 50
  ALT, Visit 19 (Month 68), n=50 | -0.5 (7.57)
  ALT, Visit 20 (Month 72), n=58: number analyzed (Participants) | 58
  ALT, Visit 20 (Month 72), n=58 | 0.6 (10.70)
  ALT, Visit 21 (Month 76), n=39: number analyzed (Participants) | 39
  ALT, Visit 21 (Month 76), n=39 | 0.3 (10.65)
  ALT, Visit 22 (Month 80), n=35: number analyzed (Participants) | 35
  ALT, Visit 22 (Month 80), n=35 | 0.1 (16.27)
  ALT, Visit 23 (Month 84), n=32: number analyzed (Participants) | 32
  ALT, Visit 23 (Month 84), n=32 | -2.3 (7.95)
  ALT, Visit 24 (Month 88), n=28: number analyzed (Participants) | 28
  ALT, Visit 24 (Month 88), n=28 | -4.1 (9.45)
  ALT, Visit 25 (Month 92), n=25: number analyzed (Participants) | 25
  ALT, Visit 25 (Month 92), n=25 | -4.2 (9.99)
  ALT, Visit 26 (Month 96), n=26: number analyzed (Participants) | 26
  ALT, Visit 26 (Month 96), n=26 | -1.6 (11.74)
  ALT, Visit 27 (Month 100), n=20: number analyzed (Participants) | 20
  ALT, Visit 27 (Month 100), n=20 | -3.2 (6.76)
  ALT, Visit 28 (Month 104), n=16: number analyzed (Participants) | 16
  ALT, Visit 28 (Month 104), n=16 | -3.1 (12.15)
  ALT, Visit 29 (Month 108), n=13: number analyzed (Participants) | 13
  ALT, Visit 29 (Month 108), n=13 | -3.6 (8.65)
  ALT, Visit 30 (Month 112), n=4: number analyzed (Participants) | 4
  ALT, Visit 30 (Month 112), n=4 | -5.3 (11.84)
  ALT, Visit 31 (Month 116), n=3: number analyzed (Participants) | 3
  ALT, Visit 31 (Month 116), n=3 | 2.3 (18.15)
  ALT, Visit 32 (Month 120), n=1: number analyzed (Participants) | 1
  ALT, Visit 32 (Month 120), n=1 | 1.0 (NA) — Standard deviation could not be calculated as only 1 participant was analyzed.
  ALT, Follow up, n=259: number analyzed (Participants) | 259
  ALT, Follow up, n=259 | 5.5 (64.04)
  AST, Visit 1 (Month 1), n=352: number analyzed (Participants) | 352
  AST, Visit 1 (Month 1), n=352 | 2.1 (13.00)
  AST, Visit 1a (Month 2), n=1: number analyzed (Participants) | 1
  AST, Visit 1a (Month 2), n=1 | -65.0 (NA) — Standard deviation could not be calculated as only 1 participant was analyzed.
  AST, Visit 2 (Month 3), n=322: number analyzed (Participants) | 322
  AST, Visit 2 (Month 3), n=322 | 1.8 (14.76)
  AST, Visit 2a (Month 4), n=1: number analyzed (Participants) | 1
  AST, Visit 2a (Month 4), n=1 | 24.0 (NA) — Standard deviation could not be calculated as only 1 participant was analyzed.
  AST, Visit 3 (Month 6), n=278: number analyzed (Participants) | 278
  AST, Visit 3 (Month 6), n=278 | 1.0 (9.60)
  AST, Visit 4 (Month 9), n=246: number analyzed (Participants) | 246
  AST, Visit 4 (Month 9), n=246 | 0.7 (8.90)
  AST, Visit 5 (Month 12), n=227: number analyzed (Participants) | 227
  AST, Visit 5 (Month 12), n=227 | 3.0 (16.88)
  AST, Visit 6 (Month 16), n=200: number analyzed (Participants) | 200
  AST, Visit 6 (Month 16), n=200 | 1.7 (7.95)
  AST, Visit 7 (Month 20), n=174: number analyzed (Participants) | 174
  AST, Visit 7 (Month 20), n=174 | 2.7 (10.53)
  AST, Visit 8 (Month 24), n=162: number analyzed (Participants) | 162
  AST, Visit 8 (Month 24), n=162 | 2.7 (8.42)
  AST, Visit 9 (Month 28), n=141: number analyzed (Participants) | 141
  AST, Visit 9 (Month 28), n=141 | 3.3 (11.36)
  AST, Visit 10 (Month 32), n=126: number analyzed (Participants) | 126
  AST, Visit 10 (Month 32), n=126 | 3.3 (7.36)
  AST, Visit 11 (Month 36), n=115: number analyzed (Participants) | 115
  AST, Visit 11 (Month 36), n=115 | 3.2 (7.77)
  AST, Visit 12 (Month 40), n=106: number analyzed (Participants) | 106
  AST, Visit 12 (Month 40), n=106 | 3.6 (8.78)
  AST, Visit 13 (Month 44), n=101: number analyzed (Participants) | 101
  AST, Visit 13 (Month 44), n=101 | 3.7 (8.37)
  AST, Visit 14 (Month 48), n=99: number analyzed (Participants) | 99
  AST, Visit 14 (Month 48), n=99 | 3.9 (7.67)
  AST, Visit 15 (Month 52), n=87: number analyzed (Participants) | 87
  AST, Visit 15 (Month 52), n=87 | 2.7 (8.15)
  AST, Visit 16 (Month 56), n=74: number analyzed (Participants) | 74
  AST, Visit 16 (Month 56), n=74 | 3.7 (8.77)
  AST, Visit 17 (Month 60), n=89: number analyzed (Participants) | 89
  AST, Visit 17 (Month 60), n=89 | 3.6 (6.57)
  AST, Visit 18 (Month 64), n=54: number analyzed (Participants) | 54
  AST, Visit 18 (Month 64), n=54 | 2.1 (8.24)
  AST, Visit 19 (Month 68), n=50: number analyzed (Participants) | 50
  AST, Visit 19 (Month 68), n=50 | 2.3 (7.22)
  AST, Visit 20 (Month 72), n=58: number analyzed (Participants) | 58
  AST, Visit 20 (Month 72), n=58 | 4.0 (10.35)
  AST, Visit 21 (Month 76), n=39: number analyzed (Participants) | 39
  AST, Visit 21 (Month 76), n=39 | 3.9 (10.22)
  AST, Visit 22 (Month 80), n=35: number analyzed (Participants) | 35
  AST, Visit 22 (Month 80), n=35 | 3.8 (11.96)
  AST, Visit 23 (Month 84), n=32: number analyzed (Participants) | 32
  AST, Visit 23 (Month 84), n=32 | 1.9 (9.96)
  AST, Visit 24 (Month 88), n=28: number analyzed (Participants) | 28
  AST, Visit 24 (Month 88), n=28 | 3.5 (11.21)
  AST, Visit 25 (Month 92), n=25: number analyzed (Participants) | 25
  AST, Visit 25 (Month 92), n=25 | 1.3 (9.09)
  AST, Visit 26 (Month 96), n=26: number analyzed (Participants) | 26
  AST, Visit 26 (Month 96), n=26 | 2.5 (9.78)
  AST, Visit 27 (Month 100), n=20: number analyzed (Participants) | 20
  AST, Visit 27 (Month 100), n=20 | 1.6 (7.67)
  AST, Visit 28 (Month 104), n=16: number analyzed (Participants) | 16
  AST, Visit 28 (Month 104), n=16 | 3.2 (10.71)
  AST, Visit 29 (Month 108), n=13: number analyzed (Participants) | 13
  AST, Visit 29 (Month 108), n=13 | 0.7 (8.70)
  AST, Visit 30 (Month 112), n=4: number analyzed (Participants) | 4
  AST, Visit 30 (Month 112), n=4 | -4.5 (10.60)
  AST, Visit 31 (Month 116), n=3: number analyzed (Participants) | 3
  AST, Visit 31 (Month 116), n=3 | 2.7 (23.03)
  AST, Visit 32 (Month 120), n=1: number analyzed (Participants) | 1
  AST, Visit 32 (Month 120), n=1 | 7.0 (NA) — Standard deviation could not be calculated as only 1 participant was analyzed.
  AST, Follow up, n=257: number analyzed (Participants) | 257
  AST, Follow up, n=257 | 3.4 (36.36)

10. Primary Outcome: Change From Baseline in Bicarbonate, Calcium, Chloride, Cholesterol, Non-fasting Glucose, Phosphorus, Potassium, Sodium and Urea
Description: Clinical chemistry parameters included bicarbonate, calcium, chloride, cholesterol, Non-fasting Glucose, phosphorus, potassium, sodium and urea. Approximately 7-milliliter sample of blood was drawn for clinical chemistry assays. The clinical laboratory evaluations were performed at all study visits during the Open-Label Treatment Phase. Baseline assessment in this OLE study was defined as the last assessment of that endpoint in VRX-RET-E22-302 taken prior to the first active treatment with retigabine. Change from Baseline was calculated by subtracting the Baseline value from the post Baseline values. NA indicates standard deviation could not be calculated as only 1 participant was analyzed. Only those participants with data available at the specified time points were analyzed (represented by n=X in the category titles).
Time Frame: Baseline and up to 122 months
Population: Safety Population
Measure: Mean (Standard Deviation); unit: Millimoles per liter
Arm/Group | Retigabine
Number analyzed (Participants) | 376
Millimoles per liter
  Bicarbonate, Visit 1 (Month 1), n=344: number analyzed (Participants) | 344
  Bicarbonate, Visit 1 (Month 1), n=344 | -0.2 (3.02)
  Bicarbonate, Visit 1a (Month 2), n=1: number analyzed (Participants) | 1
  Bicarbonate, Visit 1a (Month 2), n=1 | -2.0 (NA) — Standard deviation could not be calculated as only 1 participant was analyzed.
  Bicarbonate, Visit 2 (Month 3), n=316: number analyzed (Participants) | 316
  Bicarbonate, Visit 2 (Month 3), n=316 | -0.3 (3.34)
  Bicarbonate, Visit 3 (Month 6), n=272: number analyzed (Participants) | 272
  Bicarbonate, Visit 3 (Month 6), n=272 | 0.0 (3.06)
  Bicarbonate, Visit 4 (Month 9), n=243: number analyzed (Participants) | 243
  Bicarbonate, Visit 4 (Month 9), n=243 | -0.3 (3.22)
  Bicarbonate, Visit 5 (Month 12), n=221: number analyzed (Participants) | 221
  Bicarbonate, Visit 5 (Month 12), n=221 | -0.8 (3.18)
  Bicarbonate, Visit 6 (Month 16), n=196: number analyzed (Participants) | 196
  Bicarbonate, Visit 6 (Month 16), n=196 | -0.2 (3.11)
  Bicarbonate, Visit 7 (Month 20), n=171: number analyzed (Participants) | 171
  Bicarbonate, Visit 7 (Month 20), n=171 | -0.2 (3.22)
  Bicarbonate, Visit 8 (Month 24), n=159: number analyzed (Participants) | 159
  Bicarbonate, Visit 8 (Month 24), n=159 | -0.2 (3.26)
  Bicarbonate, Visit 9 (Month 28), n=140: number analyzed (Participants) | 140
  Bicarbonate, Visit 9 (Month 28), n=140 | -0.1 (3.44)
  Bicarbonate, Visit 10 (Month 32), n=126: number analyzed (Participants) | 126
  Bicarbonate, Visit 10 (Month 32), n=126 | -0.5 (3.74)
  Bicarbonate, Visit 11 (Month 36), n=116: number analyzed (Participants) | 116
  Bicarbonate, Visit 11 (Month 36), n=116 | -0.4 (3.54)
  Bicarbonate, Visit 12 (Month 40), n=107: number analyzed (Participants) | 107
  Bicarbonate, Visit 12 (Month 40), n=107 | 0.0 (3.52)
  Bicarbonate, Visit 13 (Month 44), n=100: number analyzed (Participants) | 100
  Bicarbonate, Visit 13 (Month 44), n=100 | 0.4 (3.41)
  Bicarbonate, Visit 14 (Month 48), n=101: number analyzed (Participants) | 101
  Bicarbonate, Visit 14 (Month 48), n=101 | -0.1 (3.56)
  Bicarbonate, Visit 15 (Month 52), n=86: number analyzed (Participants) | 86
  Bicarbonate, Visit 15 (Month 52), n=86 | 0.5 (3.77)
  Bicarbonate, Visit 16 (Month 56), n=76: number analyzed (Participants) | 76
  Bicarbonate, Visit 16 (Month 56), n=76 | -0.1 (3.07)
  Bicarbonate, Visit 17 (Month 60), n=90: number analyzed (Participants) | 90
  Bicarbonate, Visit 17 (Month 60), n=90 | -0.1 (3.45)
  Bicarbonate, Visit 18 (Month 64), n=55: number analyzed (Participants) | 55
  Bicarbonate, Visit 18 (Month 64), n=55 | -0.7 (3.93)
  Bicarbonate, Visit 19 (Month 68), n=49: number analyzed (Participants) | 49
  Bicarbonate, Visit 19 (Month 68), n=49 | -1.1 (4.11)
  Bicarbonate, Visit 20 (Month 72), n=56: number analyzed (Participants) | 56
  Bicarbonate, Visit 20 (Month 72), n=56 | -1.2 (3.81)
  Bicarbonate, Visit 21 (Month 76), n=39: number analyzed (Participants) | 39
  Bicarbonate, Visit 21 (Month 76), n=39 | -0.2 (3.58)
  Bicarbonate, Visit 22 (Month 80), n=35: number analyzed (Participants) | 35
  Bicarbonate, Visit 22 (Month 80), n=35 | -1.0 (3.24)
  Bicarbonate, Visit 23 (Month 84), n=32: number analyzed (Participants) | 32
  Bicarbonate, Visit 23 (Month 84), n=32 | -1.3 (3.17)
  Bicarbonate, Visit 24 (Month 88), n=28: number analyzed (Participants) | 28
  Bicarbonate, Visit 24 (Month 88), n=28 | -0.7 (3.56)
  Bicarbonate, Visit 25 (Month 92), n=25: number analyzed (Participants) | 25
  Bicarbonate, Visit 25 (Month 92), n=25 | -1.8 (3.15)
  Bicarbonate, Visit 26 (Month 96), n=25: number analyzed (Participants) | 25
  Bicarbonate, Visit 26 (Month 96), n=25 | -1.0 (3.48)
  Bicarbonate, Visit 27 (Month 100), n=20: number analyzed (Participants) | 20
  Bicarbonate, Visit 27 (Month 100), n=20 | -1.3 (3.91)
  Bicarbonate, Visit 28 (Month 104), n=15: number analyzed (Participants) | 15
  Bicarbonate, Visit 28 (Month 104), n=15 | -1.9 (3.70)
  Bicarbonate, Visit 29 (Month 108), n=13: number analyzed (Participants) | 13
  Bicarbonate, Visit 29 (Month 108), n=13 | -1.8 (2.35)
  Bicarbonate, Visit 30 (Month 112), n=4: number analyzed (Participants) | 4
  Bicarbonate, Visit 30 (Month 112), n=4 | -2.0 (1.41)
  Bicarbonate, Visit 31 (Month 116), n=3: number analyzed (Participants) | 3
  Bicarbonate, Visit 31 (Month 116), n=3 | 3.3 (6.11)
  Bicarbonate, Visit 32 (Month 120), n=1: number analyzed (Participants) | 1
  Bicarbonate, Visit 32 (Month 120), n=1 | 2.0 (NA) — Standard deviation could not be calculated as only 1 participant was analyzed.
  Bicarbonate, Follow up, n=256: number analyzed (Participants) | 256
  Bicarbonate, Follow up, n=256 | -1.0 (3.19)
  Calcium, Visit 1 (Month 1), n=352: number analyzed (Participants) | 352
  Calcium, Visit 1 (Month 1), n=352 | 0.000 (0.1187)
  Calcium, Visit 1a (Month 2), n=1: number analyzed (Participants) | 1
  Calcium, Visit 1a (Month 2), n=1 | -0.250 (NA) — Standard deviation could not be calculated as only 1 participant was analyzed.
  Calcium, Visit 2 (Month 3), n=322: number analyzed (Participants) | 322
  Calcium, Visit 2 (Month 3), n=322 | 0.008 (0.1146)
  Calcium, Visit 2a (Month 4), n=1: number analyzed (Participants) | 1
  Calcium, Visit 2a (Month 4), n=1 | -0.100 (NA) — Standard deviation could not be calculated as only 1 participant was analyzed.
  Calcium, Visit 3 (Month 6), n=279: number analyzed (Participants) | 279
  Calcium, Visit 3 (Month 6), n=279 | 0.018 (0.1169)
  Calcium, Visit 4 (Month 9), n=248: number analyzed (Participants) | 248
  Calcium, Visit 4 (Month 9), n=248 | 0.022 (0.1187)
  Calcium, Visit 5 (Month 12), n=228: number analyzed (Participants) | 228
  Calcium, Visit 5 (Month 12), n=228 | 0.010 (0.1269)
  Calcium, Visit 6 (Month 16), n=200: number analyzed (Participants) | 200
  Calcium, Visit 6 (Month 16), n=200 | 0.005 (0.1168)
  Calcium, Visit 7 (Month 20), n=176: number analyzed (Participants) | 176
  Calcium, Visit 7 (Month 20), n=176 | 0.005 (0.1118)
  Calcium, Visit 8 (Month 24), n=163: number analyzed (Participants) | 163
  Calcium, Visit 8 (Month 24), n=163 | 0.014 (0.1193)
  Calcium, Visit 9 (Month 28), n=142: number analyzed (Participants) | 142
  Calcium, Visit 9 (Month 28), n=142 | 0.015 (0.1154)
  Calcium, Visit 10 (Month 32), n=126: number analyzed (Participants) | 126
  Calcium, Visit 10 (Month 32), n=126 | 0.023 (0.1161)
  Calcium, Visit 11 (Month 36), n=116: number analyzed (Participants) | 116
  Calcium, Visit 11 (Month 36), n=116 | 0.017 (0.1274)
  Calcium, Visit 12 (Month 40), n=108: number analyzed (Participants) | 108
  Calcium, Visit 12 (Month 40), n=108 | 0.035 (0.1239)
  Calcium, Visit 13 (Month 44), n=101: number analyzed (Participants) | 101
  Calcium, Visit 13 (Month 44), n=101 | 0.028 (0.1168)
  Calcium, Visit 14 (Month 48), n=101: number analyzed (Participants) | 101
  Calcium, Visit 14 (Month 48), n=101 | 0.025 (0.1176)
  Calcium, Visit 15 (Month 52), n=88: number analyzed (Participants) | 88
  Calcium, Visit 15 (Month 52), n=88 | 0.020 (0.1225)
  Calcium, Visit 16 (Month 56), n=76: number analyzed (Participants) | 76
  Calcium, Visit 16 (Month 56), n=76 | 0.016 (0.1227)
  Calcium, Visit 17 (Month 60), n=90: number analyzed (Participants) | 90
  Calcium, Visit 17 (Month 60), n=90 | 0.008 (0.1172)
  Calcium, Visit 18 (Month 64), n=55: number analyzed (Participants) | 55
  Calcium, Visit 18 (Month 64), n=55 | -0.007 (0.1270)
  Calcium, Visit 19 (Month 68), n=51: number analyzed (Participants) | 51
  Calcium, Visit 19 (Month 68), n=51 | 0.019 (0.1177)
  Calcium, Visit 20 (Month 72), n=58: number analyzed (Participants) | 58
  Calcium, Visit 20 (Month 72), n=58 | -0.012 (0.1298)
  Calcium, Visit 21 (Month 76), n=40: number analyzed (Participants) | 40
  Calcium, Visit 21 (Month 76), n=40 | 0.020 (0.1257)
  Calcium, Visit 22 (Month 80), n=35: number analyzed (Participants) | 35
  Calcium, Visit 22 (Month 80), n=35 | 0.079 (0.1531)
  Calcium, Visit 23 (Month 84), n=32: number analyzed (Participants) | 32
  Calcium, Visit 23 (Month 84), n=32 | 0.038 (0.1113)
  Calcium, Visit 24 (Month 88), n=28: number analyzed (Participants) | 28
  Calcium, Visit 24 (Month 88), n=28 | 0.034 (0.1497)
  Calcium, Visit 25 (Month 92), n=25: number analyzed (Participants) | 25
  Calcium, Visit 25 (Month 92), n=25 | 0.089 (0.1560)
  Calcium, Visit 26 (Month 96), n=26: number analyzed (Participants) | 26
  Calcium, Visit 26 (Month 96), n=26 | 0.075 (0.1636)
  Calcium, Visit 27 (Month 100), n=20: number analyzed (Participants) | 20
  Calcium, Visit 27 (Month 100), n=20 | 0.121 (0.1552)
  Calcium, Visit 28 (Month 104), n=16: number analyzed (Participants) | 16
  Calcium, Visit 28 (Month 104), n=16 | 0.091 (0.1653)
  Calcium, Visit 29 (Month 108), n=13: number analyzed (Participants) | 13
  Calcium, Visit 29 (Month 108), n=13 | 0.080 (0.1297)
  Calcium, Visit 30 (Month 112), n=4: number analyzed (Participants) | 4
  Calcium, Visit 30 (Month 112), n=4 | 0.133 (0.1063)
  Calcium, Visit 31 (Month 116), n=3: number analyzed (Participants) | 3
  Calcium, Visit 31 (Month 116), n=3 | 0.053 (0.1124)
  Calcium, Visit 32 (Month 120), n=1: number analyzed (Participants) | 1
  Calcium, Visit 32 (Month 120), n=1 | -0.040 (NA) — Standard deviation could not be calculated as only 1 participant was analyzed.
  Calcium, Follow up, n=261: number analyzed (Participants) | 261
  Calcium, Follow up, n=261 | 0.031 (0.1245)
  Chloride, Visit 1 (Month 1), n=352: number analyzed (Participants) | 352
  Chloride, Visit 1 (Month 1), n=352 | 0.1 (3.48)
  Chloride, Visit 1a (Month 2), n=1: number analyzed (Participants) | 1
  Chloride, Visit 1a (Month 2), n=1 | 1.0 (NA) — Standard deviation could not be calculated as only 1 participant was analyzed.
  Chloride, Visit 2 (Month 3), n=322: number analyzed (Participants) | 322
  Chloride, Visit 2 (Month 3), n=322 | 0.3 (3.49)
  Chloride, Visit 2a (Month 4), n=1: number analyzed (Participants) | 1
  Chloride, Visit 2a (Month 4), n=1 | 2.0 (NA) — Standard deviation could not be calculated as only 1 participant was analyzed.
  Chloride, Visit 3 (Month 6), n=279: number analyzed (Participants) | 279
  Chloride, Visit 3 (Month 6), n=279 | 0.9 (3.52)
  Chloride, Visit 4 (Month 9), n=248: number analyzed (Participants) | 248
  Chloride, Visit 4 (Month 9), n=248 | 1.0 (3.46)
  Chloride, Visit 5 (Month 12), n=228: number analyzed (Participants) | 228
  Chloride, Visit 5 (Month 12), n=228 | 1.2 (3.75)
  Chloride, Visit 6 (Month 16), n=200: number analyzed (Participants) | 200
  Chloride, Visit 6 (Month 16), n=200 | 1.8 (3.73)
  Chloride, Visit 7 (Month 20), n=176: number analyzed (Participants) | 176
  Chloride, Visit 7 (Month 20), n=176 | 2.0 (4.09)
  Chloride, Visit 8 (Month 24), n=164: number analyzed (Participants) | 164
  Chloride, Visit 8 (Month 24), n=164 | 1.8 (4.42)
  Chloride, Visit 9 (Month 28), n=143: number analyzed (Participants) | 143
  Chloride, Visit 9 (Month 28), n=143 | 2.1 (4.45)
  Chloride, Visit 10 (Month 32), n=127: number analyzed (Participants) | 127
  Chloride, Visit 10 (Month 32), n=127 | 1.3 (4.22)
  Chloride, Visit 11 (Month 36), n=118: number analyzed (Participants) | 118
  Chloride, Visit 11 (Month 36), n=118 | 1.3 (4.55)
  Chloride, Visit 12 (Month 40), n=108: number analyzed (Participants) | 108
  Chloride, Visit 12 (Month 40), n=108 | 2.4 (4.68)
  Chloride, Visit 13 (Month 44), n=103: number analyzed (Participants) | 103
  Chloride, Visit 13 (Month 44), n=103 | 2.2 (4.59)
  Chloride, Visit 14 (Month 48), n=102: number analyzed (Participants) | 102
  Chloride, Visit 14 (Month 48), n=102 | 1.2 (4.91)
  Chloride, Visit 15 (Month 52), n=89: number analyzed (Participants) | 89
  Chloride, Visit 15 (Month 52), n=89 | 2.0 (4.63)
  Chloride, Visit 16 (Month 56), n=76: number analyzed (Participants) | 76
  Chloride, Visit 16 (Month 56), n=76 | 1.6 (4.51)
  Chloride, Visit 17 (Month 60), n=91: number analyzed (Participants) | 91
  Chloride, Visit 17 (Month 60), n=91 | 1.3 (5.16)
  Chloride, Visit 18 (Month 64), n=55: number analyzed (Participants) | 55
  Chloride, Visit 18 (Month 64), n=55 | 2.3 (3.33)
  Chloride, Visit 19 (Month 68), n=51: number analyzed (Participants) | 51
  Chloride, Visit 19 (Month 68), n=51 | 0.9 (4.22)
  Chloride, Visit 20 (Month 72), n=58: number analyzed (Participants) | 58
  Chloride, Visit 20 (Month 72), n=58 | 0.2 (5.33)
  Chloride, Visit 21 (Month 76), n=40: number analyzed (Participants) | 40
  Chloride, Visit 21 (Month 76), n=40 | 0.6 (4.11)
  Chloride, Visit 22 (Month 80), n=35: number analyzed (Participants) | 35
  Chloride, Visit 22 (Month 80), n=35 | 0.8 (3.30)
  Chloride, Visit 23 (Month 84), n=32: number analyzed (Participants) | 32
  Chloride, Visit 23 (Month 84), n=32 | 1.1 (4.33)
  Chloride, Visit 24 (Month 88), n=28: number analyzed (Participants) | 28
  Chloride, Visit 24 (Month 88), n=28 | 0.8 (3.94)
  Chloride, Visit 25 (Month 92), n=25: number analyzed (Participants) | 25
  Chloride, Visit 25 (Month 92), n=25 | -0.4 (5.97)
  Chloride, Visit 26 (Month 96), n=26: number analyzed (Participants) | 26
  Chloride, Visit 26 (Month 96), n=26 | -0.4 (4.56)
  Chloride, Visit 27 (Month 100), n=20: number analyzed (Participants) | 20
  Chloride, Visit 27 (Month 100), n=20 | 0.1 (5.31)
  Chloride, Visit 28 (Month 104), n=16: number analyzed (Participants) | 16
  Chloride, Visit 28 (Month 104), n=16 | -1.1 (4.86)
  Chloride, Visit 29 (Month 108), n=13: number analyzed (Participants) | 13
  Chloride, Visit 29 (Month 108), n=13 | -1.0 (5.66)
  Chloride,Visit 30 (Month 112), n=4: number analyzed (Participants) | 4
  Chloride,Visit 30 (Month 112), n=4 | -3.0 (4.24)
  Chloride,Visit 31 (Month 116), n=3: number analyzed (Participants) | 3
  Chloride,Visit 31 (Month 116), n=3 | -2.3 (5.03)
  Chloride, Visit 32 (Month 120), n=1: number analyzed (Participants) | 1
  Chloride, Visit 32 (Month 120), n=1 | -3.0 (NA) — Standard deviation could not be calculated as only 1 participant was analyzed.
  Chloride, Follow up, n=261: number analyzed (Participants) | 261
  Chloride, Follow up, n=261 | 0.3 (4.03)
  Cholesterol, Visit 1 (Month 1), n=352: number analyzed (Participants) | 352
  Cholesterol, Visit 1 (Month 1), n=352 | 0.066 (0.6255)
  Cholesterol, Visit 1a (Month 2), n=1: number analyzed (Participants) | 1
  Cholesterol, Visit 1a (Month 2), n=1 | -0.360 (NA) — Standard deviation could not be calculated as only 1 participant was analyzed.
  Cholesterol, Visit 2 (Month 3), n=322: number analyzed (Participants) | 322
  Cholesterol, Visit 2 (Month 3), n=322 | 0.108 (0.6368)
  Cholesterol, Visit 2a (Month 4), n=1: number analyzed (Participants) | 1
  Cholesterol, Visit 2a (Month 4), n=1 | -0.470 (NA) — Standard deviation could not be calculated as only 1 participant was analyzed.
  Cholesterol, Visit 3 (Month 6), n=279: number analyzed (Participants) | 279
  Cholesterol, Visit 3 (Month 6), n=279 | 0.062 (0.6978)
  Cholesterol, Visit 4 (Month 9), n=248: number analyzed (Participants) | 248
  Cholesterol, Visit 4 (Month 9), n=248 | 0.062 (0.7238)
  Cholesterol, Visit 5 (Month 12), n=228: number analyzed (Participants) | 228
  Cholesterol, Visit 5 (Month 12), n=228 | 0.075 (0.7074)
  Cholesterol, Visit 6 (Month 16), n=200: number analyzed (Participants) | 200
  Cholesterol, Visit 6 (Month 16), n=200 | 0.101 (0.7601)
  Cholesterol, Visit 7 (Month 20), n=176: number analyzed (Participants) | 176
  Cholesterol, Visit 7 (Month 20), n=176 | 0.001 (0.7820)
  Cholesterol, Visit 8 (Month 24), n=163: number analyzed (Participants) | 163
  Cholesterol, Visit 8 (Month 24), n=163 | 0.087 (0.8471)
  Cholesterol, Visit 9 (Month 28), n=142: number analyzed (Participants) | 142
  Cholesterol, Visit 9 (Month 28), n=142 | -0.001 (0.7732)
  Cholesterol, Visit 10 (Month 32), n=126: number analyzed (Participants) | 126
  Cholesterol, Visit 10 (Month 32), n=126 | -0.028 (0.8520)
  Cholesterol, Visit 11 (Month 36), n=116: number analyzed (Participants) | 116
  Cholesterol, Visit 11 (Month 36), n=116 | -0.087 (0.7823)
  Cholesterol, Visit 12 (Month 40), n=108: number analyzed (Participants) | 108
  Cholesterol, Visit 12 (Month 40), n=108 | -0.001 (0.7830)
  Cholesterol, Visit 13 (Month 44), n=101: number analyzed (Participants) | 101
  Cholesterol, Visit 13 (Month 44), n=101 | -0.043 (0.8053)
  Cholesterol, Visit 14 (Month 48), n=101: number analyzed (Participants) | 101
  Cholesterol, Visit 14 (Month 48), n=101 | -0.128 (0.7505)
  Cholesterol, Visit 15 (Month 52), n=88: number analyzed (Participants) | 88
  Cholesterol, Visit 15 (Month 52), n=88 | -0.057 (0.7427)
  Cholesterol, Visit 16 (Month 56), n=76: number analyzed (Participants) | 76
  Cholesterol, Visit 16 (Month 56), n=76 | 0.026 (0.7354)
  Cholesterol, Visit 17 (Month 60), n=90: number analyzed (Participants) | 90
  Cholesterol, Visit 17 (Month 60), n=90 | 0.016 (0.8209)
  Cholesterol, Visit 18 (Month 64), n=55: number analyzed (Participants) | 55
  Cholesterol, Visit 18 (Month 64), n=55 | 0.054 (0.7474)
  Cholesterol, Visit 19 (Month 68), n=50: number analyzed (Participants) | 50
  Cholesterol, Visit 19 (Month 68), n=50 | 0.074 (0.8943)
  Cholesterol, Visit 20 (Month 72), n=58: number analyzed (Participants) | 58
  Cholesterol, Visit 20 (Month 72), n=58 | -0.048 (0.8221)
  Cholesterol, Visit 21 (Month 76), n=40: number analyzed (Participants) | 40
  Cholesterol, Visit 21 (Month 76), n=40 | 0.103 (0.9056)
  Cholesterol, Visit 22 (Month 80), n=35: number analyzed (Participants) | 35
  Cholesterol, Visit 22 (Month 80), n=35 | 0.096 (0.8671)
  Cholesterol, Visit 23 (Month 84), n=32: number analyzed (Participants) | 32
  Cholesterol, Visit 23 (Month 84), n=32 | 0.077 (0.9637)
  Cholesterol, Visit 24 (Month 88), n=28: number analyzed (Participants) | 28
  Cholesterol, Visit 24 (Month 88), n=28 | 0.310 (0.8553)
  Cholesterol, Visit 25 (Month 92), n=25: number analyzed (Participants) | 25
  Cholesterol, Visit 25 (Month 92), n=25 | 0.327 (0.8143)
  Cholesterol, Visit 26 (Month 96), n=26: number analyzed (Participants) | 26
  Cholesterol, Visit 26 (Month 96), n=26 | 0.489 (1.0353)
  Cholesterol, Visit 27 (Month 100), n=20: number analyzed (Participants) | 20
  Cholesterol, Visit 27 (Month 100), n=20 | 0.370 (0.6675)
  Cholesterol, Visit 28 (Month 104), n=16: number analyzed (Participants) | 16
  Cholesterol, Visit 28 (Month 104), n=16 | 0.354 (0.6488)
  Cholesterol, Visit 29 (Month 108), n=13: number analyzed (Participants) | 13
  Cholesterol, Visit 29 (Month 108), n=13 | 0.141 (1.0346)
  Cholesterol, Visit 30 (Month 112), n=4: number analyzed (Participants) | 4
  Cholesterol, Visit 30 (Month 112), n=4 | 1.775 (0.9858)
  Cholesterol, Visit 31 (Month 116), n=3: number analyzed (Participants) | 3
  Cholesterol, Visit 31 (Month 116), n=3 | 1.123 (0.8723)
  Cholesterol, Visit 32 (Month 120), n=1: number analyzed (Participants) | 1
  Cholesterol, Visit 32 (Month 120), n=1 | 0.050 (NA) — Standard deviation could not be calculated as only 1 participant was analyzed.
  Cholesterol, Follow up, n=261: number analyzed (Participants) | 261
  Cholesterol, Follow up, n=261 | -0.070 (0.7047)
  Non-fasting Glucose, Visit 1 (Month 1), n=351: number analyzed (Participants) | 351
  Non-fasting Glucose, Visit 1 (Month 1), n=351 | 0.06 (0.885)
  Non-fasting Glucose, Visit 1a (Month 2), n=1: number analyzed (Participants) | 1
  Non-fasting Glucose, Visit 1a (Month 2), n=1 | -0.30 (NA) — Standard deviation could not be calculated as only 1 participant was analyzed.
  Non-fasting Glucose, Visit 2 (Month 3), n=321: number analyzed (Participants) | 321
  Non-fasting Glucose, Visit 2 (Month 3), n=321 | 0.17 (1.002)
  Non-fasting Glucose, Visit 2a (Month 4), n=1: number analyzed (Participants) | 1
  Non-fasting Glucose, Visit 2a (Month 4), n=1 | 0.40 (NA) — Standard deviation could not be calculated as only 1 participant was analyzed.
  Non-fasting Glucose, Visit 3 (Month 6), n=278: number analyzed (Participants) | 278
  Non-fasting Glucose, Visit 3 (Month 6), n=278 | 0.12 (0.804)
  Non-fasting Glucose, Visit 4 (Month 9), n=247: number analyzed (Participants) | 247
  Non-fasting Glucose, Visit 4 (Month 9), n=247 | 0.16 (1.066)
  Non-fasting Glucose, Visit 5 (Month 12), n=227: number analyzed (Participants) | 227
  Non-fasting Glucose, Visit 5 (Month 12), n=227 | 0.16 (0.906)
  Non-fasting Glucose, Visit 6 (Month 16), n=199: number analyzed (Participants) | 199
  Non-fasting Glucose, Visit 6 (Month 16), n=199 | 0.10 (0.851)
  Non-fasting Glucose, Visit 7 (Month 20), n=176: number analyzed (Participants) | 176
  Non-fasting Glucose, Visit 7 (Month 20), n=176 | 0.02 (0.843)
  Non-fasting Glucose, Visit 8 (Month 24), n=161: number analyzed (Participants) | 161
  Non-fasting Glucose, Visit 8 (Month 24), n=161 | 0.12 (0.858)
  Non-fasting Glucose, Visit 9 (Month 28), n=142: number analyzed (Participants) | 142
  Non-fasting Glucose, Visit 9 (Month 28), n=142 | 0.04 (0.842)
  Non-fasting Glucose, Visit 10 (Month 32), n=126: number analyzed (Participants) | 126
  Non-fasting Glucose, Visit 10 (Month 32), n=126 | 0.03 (0.976)
  Non-fasting Glucose, Visit 11 (Month 36), n=115: number analyzed (Participants) | 115
  Non-fasting Glucose, Visit 11 (Month 36), n=115 | 0.08 (0.951)
  Non-fasting Glucose, Visit 12 (Month 40), n=108: number analyzed (Participants) | 108
  Non-fasting Glucose, Visit 12 (Month 40), n=108 | 0.06 (0.938)
  Non-fasting Glucose, Visit 13 (Month 44), n=100: number analyzed (Participants) | 100
  Non-fasting Glucose, Visit 13 (Month 44), n=100 | 0.07 (0.912)
  Non-fasting Glucose, Visit 14 (Month 48), n=101: number analyzed (Participants) | 101
  Non-fasting Glucose, Visit 14 (Month 48), n=101 | -0.04 (0.881)
  Non-fasting Glucose, Visit 15 (Month 52), n=88: number analyzed (Participants) | 88
  Non-fasting Glucose, Visit 15 (Month 52), n=88 | 0.08 (0.745)
  Non-fasting Glucose, Visit 16 (Month 56), n=75: number analyzed (Participants) | 75
  Non-fasting Glucose, Visit 16 (Month 56), n=75 | 0.19 (0.931)
  Non-fasting Glucose, Visit 17 (Month 60), n=89: number analyzed (Participants) | 89
  Non-fasting Glucose, Visit 17 (Month 60), n=89 | 0.08 (0.773)
  Non-fasting Glucose, Visit 18 (Month 64), n=55: number analyzed (Participants) | 55
  Non-fasting Glucose, Visit 18 (Month 64), n=55 | 0.14 (1.125)
  Non-fasting Glucose, Visit 19 (Month 68), n=49: number analyzed (Participants) | 49
  Non-fasting Glucose, Visit 19 (Month 68), n=49 | 0.05 (0.816)
  Non-fasting Glucose, Visit 20 (Month 72), n=58: number analyzed (Participants) | 58
  Non-fasting Glucose, Visit 20 (Month 72), n=58 | 0.16 (0.878)
  Non-fasting Glucose, Visit 21 (Month 76), n=40: number analyzed (Participants) | 40
  Non-fasting Glucose, Visit 21 (Month 76), n=40 | 0.03 (0.895)
  Non-fasting Glucose, Visit 22 (Month 80), n=35: number analyzed (Participants) | 35
  Non-fasting Glucose, Visit 22 (Month 80), n=35 | 0.29 (1.116)
  Non-fasting Glucose, Visit 23 (Month 84), n=32: number analyzed (Participants) | 32
  Non-fasting Glucose, Visit 23 (Month 84), n=32 | -0.01 (0.903)
  Non-fasting Glucose, Visit 24 (Month 88), n=28: number analyzed (Participants) | 28
  Non-fasting Glucose, Visit 24 (Month 88), n=28 | 0.14 (1.017)
  Non-fasting Glucose, Visit 25 (Month 92), n=25: number analyzed (Participants) | 25
  Non-fasting Glucose, Visit 25 (Month 92), n=25 | 0.28 (1.105)
  Non-fasting Glucose, Visit 26 (Month 96), n=26: number analyzed (Participants) | 26
  Non-fasting Glucose, Visit 26 (Month 96), n=26 | 0.50 (1.381)
  Non-fasting Glucose, Visit 27 (Month 100), n=20: number analyzed (Participants) | 20
  Non-fasting Glucose, Visit 27 (Month 100), n=20 | 0.18 (1.022)
  Non-fasting Glucose, Visit 28 (Month 104), n=16: number analyzed (Participants) | 16
  Non-fasting Glucose, Visit 28 (Month 104), n=16 | 0.74 (0.916)
  Non-fasting Glucose, Visit 29 (Month 108), n=13: number analyzed (Participants) | 13
  Non-fasting Glucose, Visit 29 (Month 108), n=13 | 0.25 (0.989)
  Non-fasting Glucose, Visit 30 (Month 112), n=4: number analyzed (Participants) | 4
  Non-fasting Glucose, Visit 30 (Month 112), n=4 | 0.65 (0.839)
  Non-fasting Glucose, Visit 31 (Month 116), n=3: number analyzed (Participants) | 3
  Non-fasting Glucose, Visit 31 (Month 116), n=3 | 0.70 (1.127)
  Non-fasting Glucose, Visit 32 (Month 120), n=1: number analyzed (Participants) | 1
  Non-fasting Glucose, Visit 32 (Month 120), n=1 | -0.30 (NA) — Standard deviation could not be calculated as only 1 participant was analyzed.
  Non-fasting Glucose, Follow up, n=259: number analyzed (Participants) | 259
  Non-fasting Glucose, Follow up, n=259 | 0.18 (1.068)
  Phosphorus, Visit 1 (Month 1), n=351: number analyzed (Participants) | 351
  Phosphorus, Visit 1 (Month 1), n=351 | 0.017 (0.1991)
  Phosphorus, Visit 1a (Month 2), n=1: number analyzed (Participants) | 1
  Phosphorus, Visit 1a (Month 2), n=1 | 0.030 (NA) — Standard deviation could not be calculated as only 1 participant was analyzed.
  Phosphorus, Visit 2 (Month 3), n=320: number analyzed (Participants) | 320
  Phosphorus, Visit 2 (Month 3), n=320 | 0.014 (0.2011)
  Phosphorus, Visit 2a (Month 4), n=1: number analyzed (Participants) | 1
  Phosphorus, Visit 2a (Month 4), n=1 | 0.160 (NA) — Standard deviation could not be calculated as only 1 participant was analyzed.
  Phosphorus, Visit 3 (Month 6), n=278: number analyzed (Participants) | 278
  Phosphorus, Visit 3 (Month 6), n=278 | -0.001 (0.2125)
  Phosphorus, Visit 4 (Month 9), n=247: number analyzed (Participants) | 247
  Phosphorus, Visit 4 (Month 9), n=247 | -0.009 (0.1912)
  Phosphorus, Visit 5 (Month 12), n=227: number analyzed (Participants) | 227
  Phosphorus, Visit 5 (Month 12), n=227 | -0.016 (0.2130)
  Phosphorus, Visit 6 (Month 16), n=199: number analyzed (Participants) | 199
  Phosphorus, Visit 6 (Month 16), n=199 | -0.023 (0.1994)
  Phosphorus, Visit 7 (Month 20), n=176: number analyzed (Participants) | 176
  Phosphorus, Visit 7 (Month 20), n=176 | -0.022 (0.2224)
  Phosphorus, Visit 8 (Month 24), n=161: number analyzed (Participants) | 161
  Phosphorus, Visit 8 (Month 24), n=161 | -0.012 (0.2332)
  Phosphorus, Visit 9 (Month 28), n=142: number analyzed (Participants) | 142
  Phosphorus, Visit 9 (Month 28), n=142 | -0.011 (0.2146)
  Phosphorus, Visit 10 (Month 32), n=126: number analyzed (Participants) | 126
  Phosphorus, Visit 10 (Month 32), n=126 | -0.005 (0.2231)
  Phosphorus, Visit 11 (Month 36), n=115: number analyzed (Participants) | 115
  Phosphorus, Visit 11 (Month 36), n=115 | -0.026 (0.2284)
  Phosphorus, Visit 12 (Month 40), n=108: number analyzed (Participants) | 108
  Phosphorus, Visit 12 (Month 40), n=108 | -0.030 (0.2585)
  Phosphorus, Visit 13 (Month 44), n=100: number analyzed (Participants) | 100
  Phosphorus, Visit 13 (Month 44), n=100 | -0.026 (0.2241)
  Phosphorus, Visit 14 (Month 48), n=101: number analyzed (Participants) | 101
  Phosphorus, Visit 14 (Month 48), n=101 | -0.050 (0.2331)
  Phosphorus, Visit 15 (Month 52), n=88: number analyzed (Participants) | 88
  Phosphorus, Visit 15 (Month 52), n=88 | -0.054 (0.2207)
  Phosphorus, Visit 16 (Month 56), n=75: number analyzed (Participants) | 75
  Phosphorus, Visit 16 (Month 56), n=75 | -0.052 (0.2465)
  Phosphorus, Visit 17 (Month 60), n=89: number analyzed (Participants) | 89
  Phosphorus, Visit 17 (Month 60), n=89 | -0.047 (0.2419)
  Phosphorus, Visit 18 (Month 64), n=55: number analyzed (Participants) | 55
  Phosphorus, Visit 18 (Month 64), n=55 | -0.059 (0.2540)
  Phosphorus, Visit 19 (Month 68), n=49: number analyzed (Participants) | 49
  Phosphorus, Visit 19 (Month 68), n=49 | -0.047 (0.2905)
  Phosphorus, Visit 20 (Month 72), n=58: number analyzed (Participants) | 58
  Phosphorus, Visit 20 (Month 72), n=58 | -0.076 (0.2502)
  Phosphorus, Visit 21 (Month 76), n=40: number analyzed (Participants) | 40
  Phosphorus, Visit 21 (Month 76), n=40 | -0.074 (0.2503)
  Phosphorus, Visit 22 (Month 80), n=35: number analyzed (Participants) | 35
  Phosphorus, Visit 22 (Month 80), n=35 | -0.071 (0.2930)
  Phosphorus, Visit 23 (Month 84), n=32: number analyzed (Participants) | 32
  Phosphorus, Visit 23 (Month 84), n=32 | -0.068 (0.3006)
  Phosphorus, Visit 24 (Month 88), n=28: number analyzed (Participants) | 28
  Phosphorus, Visit 24 (Month 88), n=28 | -0.115 (0.3460)
  Phosphorus, Visit 25 (Month 92), n=25: number analyzed (Participants) | 25
  Phosphorus, Visit 25 (Month 92), n=25 | -0.130 (0.3251)
  Phosphorus, Visit 26 (Month 96), n=26: number analyzed (Participants) | 26
  Phosphorus, Visit 26 (Month 96), n=26 | -0.098 (0.2820)
  Phosphorus, Visit 27 (Month 100), n=20: number analyzed (Participants) | 20
  Phosphorus, Visit 27 (Month 100), n=20 | -0.197 (0.3030)
  Phosphorus, Visit 28 (Month 104), n=16: number analyzed (Participants) | 16
  Phosphorus, Visit 28 (Month 104), n=16 | -0.261 (0.2665)
  Phosphorus, Visit 29 (Month 108), n=13: number analyzed (Participants) | 13
  Phosphorus, Visit 29 (Month 108), n=13 | -0.300 (0.1534)
  Phosphorus, Visit 30 (Month 112), n=4: number analyzed (Participants) | 4
  Phosphorus, Visit 30 (Month 112), n=4 | -0.065 (0.0603)
  Phosphorus, Visit 31 (Month 116), n=3: number analyzed (Participants) | 3
  Phosphorus, Visit 31 (Month 116), n=3 | -0.260 (0.0000)
  Phosphorus, Visit 32 (Month 120), n=1: number analyzed (Participants) | 1
  Phosphorus, Visit 32 (Month 120), n=1 | -0.320 (NA) — Standard deviation could not be calculated as only 1 participant was analyzed.
  Phosphorus, Follow up, n=260: number analyzed (Participants) | 260
  Phosphorus, Follow up, n=260 | -0.038 (0.2237)
  Potassium, Visit 1 (Month 1), n=351: number analyzed (Participants) | 351
  Potassium, Visit 1 (Month 1), n=351 | -0.02 (0.426)
  Potassium, Visit 1a (Month 2), n=1: number analyzed (Participants) | 1
  Potassium, Visit 1a (Month 2), n=1 | -0.40 (NA) — Standard deviation could not be calculated as only 1 participant was analyzed.
  Potassium, Visit 2 (Month 3), n=322: number analyzed (Participants) | 322
  Potassium, Visit 2 (Month 3), n=322 | -0.05 (0.410)
  Potassium, Visit 2a (Month 4), n=1: number analyzed (Participants) | 1
  Potassium, Visit 2a (Month 4), n=1 | 0.40 (NA) — Standard deviation could not be calculated as only 1 participant was analyzed.
  Potassium, Visit 3 (Month 6), n=279: number analyzed (Participants) | 279
  Potassium, Visit 3 (Month 6), n=279 | -0.04 (0.424)
  Potassium, Visit 4 (Month 9), n=247: number analyzed (Participants) | 247
  Potassium, Visit 4 (Month 9), n=247 | -0.08 (0.427)
  Potassium, Visit 5 (Month 12), n=230: number analyzed (Participants) | 230
  Potassium, Visit 5 (Month 12), n=230 | -0.07 (0.440)
  Potassium, Visit 6 (Month 16), n=199: number analyzed (Participants) | 199
  Potassium, Visit 6 (Month 16), n=199 | 0.00 (0.436)
  Potassium, Visit 7 (Month 20), n=174: number analyzed (Participants) | 174
  Potassium, Visit 7 (Month 20), n=174 | -0.02 (0.434)
  Potassium, Visit 8 (Month 24), n=162: number analyzed (Participants) | 162
  Potassium, Visit 8 (Month 24), n=162 | -0.03 (0.430)
  Potassium, Visit 9 (Month 28), n=143: number analyzed (Participants) | 143
  Potassium, Visit 9 (Month 28), n=143 | -0.01 (0.434)
  Potassium, Visit 10 (Month 32), n=127: number analyzed (Participants) | 127
  Potassium, Visit 10 (Month 32), n=127 | -0.01 (0.451)
  Potassium, Visit 11 (Month 36), n=116: number analyzed (Participants) | 116
  Potassium, Visit 11 (Month 36), n=116 | -0.01 (0.457)
  Potassium, Visit 12 (Month 40), n=108: number analyzed (Participants) | 108
  Potassium, Visit 12 (Month 40), n=108 | -0.05 (0.475)
  Potassium, Visit 13 (Month 44), n=102: number analyzed (Participants) | 102
  Potassium, Visit 13 (Month 44), n=102 | -0.06 (0.466)
  Potassium, Visit 14 (Month 48), n=101: number analyzed (Participants) | 101
  Potassium, Visit 14 (Month 48), n=101 | -0.01 (0.443)
  Potassium, Visit 15 (Month 52), n=89: number analyzed (Participants) | 89
  Potassium, Visit 15 (Month 52), n=89 | -0.01 (0.436)
  Potassium, Visit 16 (Month 56), n=75: number analyzed (Participants) | 75
  Potassium, Visit 16 (Month 56), n=75 | 0.00 (0.506)
  Potassium, Visit 17 (Month 60), n=89: number analyzed (Participants) | 89
  Potassium, Visit 17 (Month 60), n=89 | -0.05 (0.477)
  Potassium, Visit 18 (Month 64), n=55: number analyzed (Participants) | 55
  Potassium, Visit 18 (Month 64), n=55 | -0.12 (0.468)
  Potassium, Visit 19 (Month 68), n=50: number analyzed (Participants) | 50
  Potassium, Visit 19 (Month 68), n=50 | -0.03 (0.484)
  Potassium, Visit 20 (Month 72), n=58: number analyzed (Participants) | 58
  Potassium, Visit 20 (Month 72), n=58 | -0.10 (0.485)
  Potassium, Visit 21 (Month 76), n=39: number analyzed (Participants) | 39
  Potassium, Visit 21 (Month 76), n=39 | -0.11 (0.469)
  Potassium, Visit 22 (Month 80), n=35: number analyzed (Participants) | 35
  Potassium, Visit 22 (Month 80), n=35 | -0.08 (0.461)
  Potassium, Visit 23 (Month 84), n=32: number analyzed (Participants) | 32
  Potassium, Visit 23 (Month 84), n=32 | 0.01 (0.523)
  Potassium, Visit 24 (Month 88), n=28: number analyzed (Participants) | 28
  Potassium, Visit 24 (Month 88), n=28 | -0.05 (0.517)
  Potassium, Visit 25 (Month 92), n=25: number analyzed (Participants) | 25
  Potassium, Visit 25 (Month 92), n=25 | -0.01 (0.488)
  Potassium, Visit 26 (Month 96), n=26: number analyzed (Participants) | 26
  Potassium, Visit 26 (Month 96), n=26 | -0.02 (0.603)
  Potassium, Visit 27 (Month 100), n=20: number analyzed (Participants) | 20
  Potassium, Visit 27 (Month 100), n=20 | -0.09 (0.609)
  Potassium, Visit 28 (Month 104), n=16: number analyzed (Participants) | 16
  Potassium, Visit 28 (Month 104), n=16 | -0.18 (0.481)
  Potassium, Visit 29 (Month 108), n=13: number analyzed (Participants) | 13
  Potassium, Visit 29 (Month 108), n=13 | -0.09 (0.647)
  Potassium, Visit 30 (Month 112), n=4: number analyzed (Participants) | 4
  Potassium, Visit 30 (Month 112), n=4 | -0.38 (0.574)
  Potassium, Visit 31 (Month 116), n=3: number analyzed (Participants) | 3
  Potassium, Visit 31 (Month 116), n=3 | -0.83 (0.611)
  Potassium, Visit 32 (Month 120), n=1: number analyzed (Participants) | 1
  Potassium, Visit 32 (Month 120), n=1 | -0.30 (NA) — Standard deviation could not be calculated as only 1 participant was analyzed.
  Potassium, Follow up, n=258: number analyzed (Participants) | 258
  Potassium, Follow up, n=258 | -0.02 (0.456)
  Sodium, Visit 1 (Month 1), n=352: number analyzed (Participants) | 352
  Sodium, Visit 1 (Month 1), n=352 | -0.3 (3.60)
  Sodium, Visit 1a (Month 2), n=1: number analyzed (Participants) | 1
  Sodium, Visit 1a (Month 2), n=1 | 0.0 (NA) — Standard deviation could not be calculated as only 1 participant was analyzed.
  Sodium, Visit 2 (Month 3), n=324: number analyzed (Participants) | 324
  Sodium, Visit 2 (Month 3), n=324 | -0.1 (3.52)
  Sodium, Visit 2a (Month 4), n=1: number analyzed (Participants) | 1
  Sodium, Visit 2a (Month 4), n=1 | 1.0 (NA) — Standard deviation could not be calculated as only 1 participant was analyzed.
  Sodium, Visit 3 (Month 6), n=280: number analyzed (Participants) | 280
  Sodium, Visit 3 (Month 6), n=280 | 0.8 (3.49)
  Sodium, Visit 4 (Month 9), n=248: number analyzed (Participants) | 248
  Sodium, Visit 4 (Month 9), n=248 | 0.5 (3.50)
  Sodium, Visit 5 (Month 12), n=231: number analyzed (Participants) | 231
  Sodium, Visit 5 (Month 12), n=231 | 0.6 (3.84)
  Sodium, Visit 6 (Month 16), n=200: number analyzed (Participants) | 200
  Sodium, Visit 6 (Month 16), n=200 | 0.9 (3.81)
  Sodium, Visit 7 (Month 20), n=176: number analyzed (Participants) | 176
  Sodium, Visit 7 (Month 20), n=176 | 1.1 (3.88)
  Sodium, Visit 8 (Month 24), n=164: number analyzed (Participants) | 164
  Sodium, Visit 8 (Month 24), n=164 | 1.0 (4.38)
  Sodium, Visit 9 (Month 28), n=143: number analyzed (Participants) | 143
  Sodium, Visit 9 (Month 28), n=143 | 1.6 (4.36)
  Sodium, Visit 10 (Month 32), n=127: number analyzed (Participants) | 127
  Sodium, Visit 10 (Month 32), n=127 | 1.2 (4.08)
  Sodium, Visit 11 (Month 36), n=118: number analyzed (Participants) | 118
  Sodium, Visit 11 (Month 36), n=118 | 1.3 (5.15)
  Sodium, Visit 12 (Month 40), n=108: number analyzed (Participants) | 108
  Sodium, Visit 12 (Month 40), n=108 | 1.9 (4.25)
  Sodium, Visit 13 (Month 44), n=103: number analyzed (Participants) | 103
  Sodium, Visit 13 (Month 44), n=103 | 1.7 (4.06)
  Sodium, Visit 14 (Month 48), n=102: number analyzed (Participants) | 102
  Sodium, Visit 14 (Month 48), n=102 | 1.1 (4.44)
  Sodium, Visit 15 (Month 52), n=89: number analyzed (Participants) | 89
  Sodium, Visit 15 (Month 52), n=89 | 1.8 (4.29)
  Sodium, Visit 16 (Month 56), n=76: number analyzed (Participants) | 76
  Sodium, Visit 16 (Month 56), n=76 | 1.7 (3.75)
  Sodium, Visit 17 (Month 60), n=91: number analyzed (Participants) | 91
  Sodium, Visit 17 (Month 60), n=91 | 1.8 (4.62)
  Sodium, Visit 18 (Month 64), n=55: number analyzed (Participants) | 55
  Sodium, Visit 18 (Month 64), n=55 | 2.7 (3.32)
  Sodium, Visit 19 (Month 68), n=51: number analyzed (Participants) | 51
  Sodium, Visit 19 (Month 68), n=51 | 2.2 (3.63)
  Sodium, Visit 20 (Month 72), n=58: number analyzed (Participants) | 58
  Sodium, Visit 20 (Month 72), n=58 | 1.0 (4.46)
  Sodium, Visit 21 (Month 76), n=40: number analyzed (Participants) | 40
  Sodium, Visit 21 (Month 76), n=40 | 2.2 (3.82)
  Sodium, Visit 22 (Month 80), n=35: number analyzed (Participants) | 35
  Sodium, Visit 22 (Month 80), n=35 | 2.0 (3.11)
  Sodium, Visit 23 (Month 84), n=32: number analyzed (Participants) | 32
  Sodium, Visit 23 (Month 84), n=32 | 2.4 (3.72)
  Sodium, Visit 24 (Month 88), n=28: number analyzed (Participants) | 28
  Sodium, Visit 24 (Month 88), n=28 | 1.9 (3.85)
  Sodium, Visit 25 (Month 92), n=25: number analyzed (Participants) | 25
  Sodium, Visit 25 (Month 92), n=25 | 1.4 (5.45)
  Sodium, Visit 26 (Month 96), n=26: number analyzed (Participants) | 26
  Sodium, Visit 26 (Month 96), n=26 | 1.8 (4.48)
  Sodium, Visit 27 (Month 100), n=20: number analyzed (Participants) | 20
  Sodium, Visit 27 (Month 100), n=20 | 1.8 (4.76)
  Sodium, Visit 28 (Month 104), n=16: number analyzed (Participants) | 16
  Sodium, Visit 28 (Month 104), n=16 | 0.9 (3.14)
  Sodium, Visit 29 (Month 108), n=13: number analyzed (Participants) | 13
  Sodium, Visit 29 (Month 108), n=13 | 0.5 (4.58)
  Sodium, Visit 30 (Month 112), n=4: number analyzed (Participants) | 4
  Sodium, Visit 30 (Month 112), n=4 | -0.3 (5.85)
  Sodium, Visit 31 (Month 116), n=3: number analyzed (Participants) | 3
  Sodium, Visit 31 (Month 116), n=3 | 0.7 (3.79)
  Sodium, Visit 32 (Month 120), n=1: number analyzed (Participants) | 1
  Sodium, Visit 32 (Month 120), n=1 | -5.0 (NA) — Standard deviation could not be calculated as only 1 participant was analyzed.
  Sodium, Follow up, n=261: number analyzed (Participants) | 261
  Sodium, Follow up, n=261 | 0.3 (3.91)
  Urea, Visit 1 (Month 1), n=351: number analyzed (Participants) | 351
  Urea, Visit 1 (Month 1), n=351 | 0.583 (1.2933)
  Urea, Visit 1a (Month 2), n=1: number analyzed (Participants) | 1
  Urea, Visit 1a (Month 2), n=1 | 2.860 (NA) — Standard deviation could not be calculated as only 1 participant was analyzed.
  Urea, Visit 2 (Month 3), n=322: number analyzed (Participants) | 322
  Urea, Visit 2 (Month 3), n=322 | 0.606 (1.2846)
  Urea, Visit 2a (Month 4), n=1: number analyzed (Participants) | 1
  Urea, Visit 2a (Month 4), n=1 | 1.780 (NA) — Standard deviation could not be calculated as only 1 participant was analyzed.
  Urea, Visit 3 (Month 6), n=279: number analyzed (Participants) | 279
  Urea, Visit 3 (Month 6), n=279 | 0.623 (1.3294)
  Urea, Visit 4 (Month 9), n=248: number analyzed (Participants) | 248
  Urea, Visit 4 (Month 9), n=248 | 0.642 (1.3781)
  Urea, Visit 5 (Month 12), n=228: number analyzed (Participants) | 228
  Urea, Visit 5 (Month 12), n=228 | 0.599 (1.3323)
  Urea, Visit 6 (Month 16), n=200: number analyzed (Participants) | 200
  Urea, Visit 6 (Month 16), n=200 | 0.656 (1.3598)
  Urea, Visit 7 (Month 20), n=176: number analyzed (Participants) | 176
  Urea, Visit 7 (Month 20), n=176 | 0.750 (1.3893)
  Urea, Visit 8 (Month 24), n=163: number analyzed (Participants) | 163
  Urea, Visit 8 (Month 24), n=163 | 0.652 (1.5332)
  Urea, Visit 9 (Month 28), n=142: number analyzed (Participants) | 142
  Urea, Visit 9 (Month 28), n=142 | 0.578 (1.3512)
  Urea, Visit 10 (Month 32), n=126: number analyzed (Participants) | 126
  Urea, Visit 10 (Month 32), n=126 | 0.748 (1.5680)
  Urea, Visit 11 (Month 36), n=117: number analyzed (Participants) | 117
  Urea, Visit 11 (Month 36), n=117 | 0.552 (1.6650)
  Urea, Visit 12 (Month 40), n=108: number analyzed (Participants) | 108
  Urea, Visit 12 (Month 40), n=108 | 0.794 (1.5456)
  Urea, Visit 13 (Month 44), n=102: number analyzed (Participants) | 102
  Urea, Visit 13 (Month 44), n=102 | 0.697 (1.5664)
  Urea, Visit 14 (Month 48), n=101: number analyzed (Participants) | 101
  Urea, Visit 14 (Month 48), n=101 | 0.792 (1.7321)
  Urea, Visit 15 (Month 52), n=88: number analyzed (Participants) | 88
  Urea, Visit 15 (Month 52), n=88 | 0.828 (1.4226)
  Urea, Visit 16 (Month 56), n=76: number analyzed (Participants) | 76
  Urea, Visit 16 (Month 56), n=76 | 0.742 (1.3964)
  Urea, Visit 17 (Month 60), n=90: number analyzed (Participants) | 90
  Urea, Visit 17 (Month 60), n=90 | 0.778 (1.5392)
  Urea, Visit 18 (Month 64), n=55: number analyzed (Participants) | 55
  Urea, Visit 18 (Month 64), n=55 | 0.766 (1.5980)
  Urea, Visit 19 (Month 68), n=51: number analyzed (Participants) | 51
  Urea, Visit 19 (Month 68), n=51 | 0.791 (1.3485)
  Urea, Visit 20 (Month 72), n=58: number analyzed (Participants) | 58
  Urea, Visit 20 (Month 72), n=58 | 0.794 (1.5895)
  Urea, Visit 21 (Month 76), n=40: number analyzed (Participants) | 40
  Urea, Visit 21 (Month 76), n=40 | 1.152 (1.3824)
  Urea, Visit 22 (Month 80), n=35: number analyzed (Participants) | 35
  Urea, Visit 22 (Month 80), n=35 | 0.939 (1.2432)
  Urea, Visit 23 (Month 84), n=32: number analyzed (Participants) | 32
  Urea, Visit 23 (Month 84), n=32 | 0.781 (1.3376)
  Urea, Visit 24 (Month 88), n=28: number analyzed (Participants) | 28
  Urea, Visit 24 (Month 88), n=28 | 0.791 (1.0485)
  Urea, Visit 25 (Month 92), n=25: number analyzed (Participants) | 25
  Urea, Visit 25 (Month 92), n=25 | 0.529 (1.6380)
  Urea, Visit 26 (Month 96), n=26: number analyzed (Participants) | 26
  Urea, Visit 26 (Month 96), n=26 | 0.811 (1.4025)
  Urea, Visit 27 (Month 100), n=20: number analyzed (Participants) | 20
  Urea, Visit 27 (Month 100), n=20 | 0.501 (1.1668)
  Urea, Visit 28 (Month 104), n=16: number analyzed (Participants) | 16
  Urea, Visit 28 (Month 104), n=16 | 0.536 (0.9589)
  Urea, Visit 29 (Month 108), n=13: number analyzed (Participants) | 13
  Urea, Visit 29 (Month 108), n=13 | 0.523 (1.2418)
  Urea, Visit 30 (Month 112), n=4: number analyzed (Participants) | 4
  Urea, Visit 30 (Month 112), n=4 | 0.983 (1.0297)
  Urea, Visit 31 (Month 116), n=3: number analyzed (Participants) | 3
  Urea, Visit 31 (Month 116), n=3 | 0.837 (1.6082)
  Urea, Visit 32 (Month 120), n=1: number analyzed (Participants) | 1
  Urea, Visit 32 (Month 120), n=1 | -1.070 (NA) — Standard deviation could not be calculated as only 1 participant was analyzed.
  Urea, Follow up, n=260: number analyzed (Participants) | 260
  Urea, Follow up, n=260 | 0.158 (1.2473)

11. Primary Outcome: Change From Baseline in Creatinine, Total Bilirubin and Uric Acid
Description: Clinical chemistry parameters included creatinine, total bilirubin and uric acid. The clinical laboratory evaluations were performed at all study visits during the Open-Label Treatment Phase. Baseline assessment in this OLE study was defined as the last assessment of that endpoint in VRX-RET-E22-302 taken prior to the first active treatment with retigabine. Change from Baseline was calculated by subtracting the Baseline value from the post Baseline values. NA indicates standard deviation could not be calculated as only 1 participant was analyzed. Only those participants with data available at the specified time points were analyzed (represented by n=X in the category titles).
Time Frame: Baseline and up to 122 months
Population: Safety Population
Measure: Mean (Standard Deviation); unit: Micromoles per liter
Arm/Group | Retigabine
Number analyzed (Participants) | 376
Micromoles per liter
  Creatinine, Visit 1 (Month 1), n=351: number analyzed (Participants) | 351
  Creatinine, Visit 1 (Month 1), n=351 | 1.8 (12.85)
  Creatinine, Visit 1a (Month 2), n=1: number analyzed (Participants) | 1
  Creatinine, Visit 1a (Month 2), n=1 | 0.0 (NA) — Standard deviation could not be calculated as only 1 participant was analyzed.
  Creatinine, Visit 2 (Month 3), n=320: number analyzed (Participants) | 320
  Creatinine, Visit 2 (Month 3), n=320 | 0.9 (8.49)
  Creatinine, Visit 2a (Month 4), n=1: number analyzed (Participants) | 1
  Creatinine, Visit 2a (Month 4), n=1 | 9.0 (NA) — Standard deviation could not be calculated as only 1 participant was analyzed.
  Creatinine, Visit 3 (Month 6), n=278: number analyzed (Participants) | 278
  Creatinine, Visit 3 (Month 6), n=278 | 0.7 (8.89)
  Creatinine, Visit 4 (Month 9), n=247: number analyzed (Participants) | 247
  Creatinine, Visit 4 (Month 9), n=247 | 0.1 (9.04)
  Creatinine, Visit 5 (Month 12), n=227: number analyzed (Participants) | 227
  Creatinine, Visit 5 (Month 12), n=227 | 0.0 (9.33)
  Creatinine, Visit 6 (Month 16), n=199: number analyzed (Participants) | 199
  Creatinine, Visit 6 (Month 16), n=199 | 0.8 (10.14)
  Creatinine, Visit 7 (Month 20), n=176: number analyzed (Participants) | 176
  Creatinine, Visit 7 (Month 20), n=176 | 0.6 (9.84)
  Creatinine, Visit 8 (Month 24), n=161: number analyzed (Participants) | 161
  Creatinine, Visit 8 (Month 24), n=161 | 0.0 (8.81)
  Creatinine, Visit 9 (Month 28), n=142: number analyzed (Participants) | 142
  Creatinine, Visit 9 (Month 28), n=142 | -0.2 (9.98)
  Creatinine, Visit 10 (Month 32), n=126: number analyzed (Participants) | 126
  Creatinine, Visit 10 (Month 32), n=126 | 1.3 (10.98)
  Creatinine, Visit 11 (Month 36), n=115: number analyzed (Participants) | 115
  Creatinine, Visit 11 (Month 36), n=115 | -0.3 (10.13)
  Creatinine, Visit 12 (Month 40), n=108: number analyzed (Participants) | 108
  Creatinine, Visit 12 (Month 40), n=108 | 0.8 (10.30)
  Creatinine, Visit 13 (Month 44), n=101: number analyzed (Participants) | 101
  Creatinine, Visit 13 (Month 44), n=101 | 0.5 (10.70)
  Creatinine, Visit 14 (Month 48), n=101: number analyzed (Participants) | 101
  Creatinine, Visit 14 (Month 48), n=101 | -0.3 (10.49)
  Creatinine, Visit 15 (Month 52), n=88: number analyzed (Participants) | 88
  Creatinine, Visit 15 (Month 52), n=88 | 0.8 (9.55)
  Creatinine, Visit 16 (Month 56), n=75: number analyzed (Participants) | 75
  Creatinine, Visit 16 (Month 56), n=75 | 1.1 (22.92)
  Creatinine, Visit 17 (Month 60), n=89: number analyzed (Participants) | 89
  Creatinine, Visit 17 (Month 60), n=89 | -1.6 (10.31)
  Creatinine, Visit 18 (Month 64), n=55: number analyzed (Participants) | 55
  Creatinine, Visit 18 (Month 64), n=55 | -0.7 (11.09)
  Creatinine, Visit 19 (Month 68), n=50: number analyzed (Participants) | 50
  Creatinine, Visit 19 (Month 68), n=50 | -0.9 (13.22)
  Creatinine, Visit 20 (Month 72), n=58: number analyzed (Participants) | 58
  Creatinine, Visit 20 (Month 72), n=58 | -3.6 (11.31)
  Creatinine, Visit 21 (Month 76), n=40: number analyzed (Participants) | 40
  Creatinine, Visit 21 (Month 76), n=40 | -0.7 (13.10)
  Creatinine, Visit 22 (Month 80), n=35: number analyzed (Participants) | 35
  Creatinine, Visit 22 (Month 80), n=35 | -2.2 (11.98)
  Creatinine, Visit 23 (Month 84), n=32: number analyzed (Participants) | 32
  Creatinine, Visit 23 (Month 84), n=32 | -1.4 (12.50)
  Creatinine, Visit 24 (Month 88), n=28: number analyzed (Participants) | 28
  Creatinine, Visit 24 (Month 88), n=28 | -4.1 (12.03)
  Creatinine, Visit 25 (Month 92), n=25: number analyzed (Participants) | 25
  Creatinine, Visit 25 (Month 92), n=25 | -3.2 (10.84)
  Creatinine, Visit 26 (Month 96), n=26: number analyzed (Participants) | 26
  Creatinine, Visit 26 (Month 96), n=26 | -2.6 (13.67)
  Creatinine, Visit 27 (Month 100), n=20: number analyzed (Participants) | 20
  Creatinine, Visit 27 (Month 100), n=20 | -3.9 (11.05)
  Creatinine, Visit 28 (Month 104), n=16: number analyzed (Participants) | 16
  Creatinine, Visit 28 (Month 104), n=16 | -4.2 (10.63)
  Creatinine, Visit 29 (Month 108), n=13: number analyzed (Participants) | 13
  Creatinine, Visit 29 (Month 108), n=13 | -7.7 (13.98)
  Creatinine, Visit 30 (Month 112), n=4: number analyzed (Participants) | 4
  Creatinine, Visit 30 (Month 112), n=4 | -6.3 (6.85)
  Creatinine, Visit 31 (Month 116), n=3: number analyzed (Participants) | 3
  Creatinine, Visit 31 (Month 116), n=3 | -18.7 (8.50)
  Creatinine, Visit 32 (Month 120), n=1: number analyzed (Participants) | 1
  Creatinine, Visit 32 (Month 120), n=1 | -19.0 (NA) — Standard deviation could not be calculated as only 1 participant was analyzed.
  Creatinine, Follow up, n=260: number analyzed (Participants) | 260
  Creatinine, Follow up, n=260 | 0.6 (9.99)
  Total Bilirubin, Visit 1 (Month 1), n=351: number analyzed (Participants) | 351
  Total Bilirubin, Visit 1 (Month 1), n=351 | 3.5 (3.41)
  Total Bilirubin, Visit 1a (Month 2), n=1: number analyzed (Participants) | 1
  Total Bilirubin, Visit 1a (Month 2), n=1 | 0.0 (NA) — Standard deviation could not be calculated as only 1 participant was analyzed.
  Total Bilirubin, Visit 2 (Month 3), n=322: number analyzed (Participants) | 322
  Total Bilirubin, Visit 2 (Month 3), n=322 | 3.5 (3.57)
  Total Bilirubin, Visit 2a (Month 4), n=1: number analyzed (Participants) | 1
  Total Bilirubin, Visit 2a (Month 4), n=1 | 6.0 (NA) — Standard deviation could not be calculated as only 1 participant was analyzed.
  Total Bilirubin, Visit 3 (Month 6), n=278: number analyzed (Participants) | 278
  Total Bilirubin, Visit 3 (Month 6), n=278 | 3.6 (3.62)
  Total Bilirubin, Visit 4 (Month 9), n=245: number analyzed (Participants) | 245
  Total Bilirubin, Visit 4 (Month 9), n=245 | 3.5 (3.63)
  Total Bilirubin, Visit 5 (Month 12), n=227: number analyzed (Participants) | 227
  Total Bilirubin, Visit 5 (Month 12), n=227 | 3.4 (3.56)
  Total Bilirubin, Visit 6 (Month 16), n=200: number analyzed (Participants) | 200
  Total Bilirubin, Visit 6 (Month 16), n=200 | 3.6 (3.69)
  Total Bilirubin, Visit 7 (Month 20), n=176: number analyzed (Participants) | 176
  Total Bilirubin, Visit 7 (Month 20), n=176 | 3.7 (3.60)
  Total Bilirubin, Visit 8 (Month 24), n=162: number analyzed (Participants) | 162
  Total Bilirubin, Visit 8 (Month 24), n=162 | 3.8 (3.70)
  Total Bilirubin, Visit 9 (Month 28), n=141: number analyzed (Participants) | 141
  Total Bilirubin, Visit 9 (Month 28), n=141 | 3.7 (3.57)
  Total Bilirubin, Visit 10 (Month 32), n=126: number analyzed (Participants) | 126
  Total Bilirubin, Visit 10 (Month 32), n=126 | 4.1 (3.68)
  Total Bilirubin, Visit 11 (Month 36), n=116: number analyzed (Participants) | 116
  Total Bilirubin, Visit 11 (Month 36), n=116 | 4.0 (3.82)
  Total Bilirubin, Visit 12 (Month 40), n=107: number analyzed (Participants) | 107
  Total Bilirubin, Visit 12 (Month 40), n=107 | 3.7 (3.44)
  Total Bilirubin, Visit 13 (Month 44), n=101: number analyzed (Participants) | 101
  Total Bilirubin, Visit 13 (Month 44), n=101 | 3.9 (3.46)
  Total Bilirubin, Visit 14 (Month 48), n=100: number analyzed (Participants) | 100
  Total Bilirubin, Visit 14 (Month 48), n=100 | 3.7 (3.67)
  Total Bilirubin, Visit 15 (Month 52), n=88: number analyzed (Participants) | 88
  Total Bilirubin, Visit 15 (Month 52), n=88 | 3.7 (3.37)
  Total Bilirubin, Visit 16 (Month 56), n=76: number analyzed (Participants) | 76
  Total Bilirubin, Visit 16 (Month 56), n=76 | 3.6 (3.47)
  Total Bilirubin, Visit 17 (Month 60), n=90: number analyzed (Participants) | 90
  Total Bilirubin, Visit 17 (Month 60), n=90 | 3.8 (3.36)
  Total Bilirubin, Visit 18 (Month 64), n=55: number analyzed (Participants) | 55
  Total Bilirubin, Visit 18 (Month 64), n=55 | 3.7 (3.68)
  Total Bilirubin, Visit 19 (Month 68), n=51: number analyzed (Participants) | 51
  Total Bilirubin, Visit 19 (Month 68), n=51 | 3.1 (4.12)
  Total Bilirubin, Visit 20 (Month 72), n=58: number analyzed (Participants) | 58
  Total Bilirubin, Visit 20 (Month 72), n=58 | 3.3 (3.69)
  Total Bilirubin, Visit 21 (Month 76), n=40: number analyzed (Participants) | 40
  Total Bilirubin, Visit 21 (Month 76), n=40 | 3.7 (4.02)
  Total Bilirubin, Visit 22 (Month 80), n=35: number analyzed (Participants) | 35
  Total Bilirubin, Visit 22 (Month 80), n=35 | 3.2 (4.22)
  Total Bilirubin, Visit 23 (Month 84), n=32: number analyzed (Participants) | 32
  Total Bilirubin, Visit 23 (Month 84), n=32 | 3.4 (4.01)
  Total Bilirubin, Visit 24 (Month 88), n=28: number analyzed (Participants) | 28
  Total Bilirubin, Visit 24 (Month 88), n=28 | 3.6 (5.04)
  Total Bilirubin, Visit 25 (Month 92), n=25: number analyzed (Participants) | 25
  Total Bilirubin, Visit 25 (Month 92), n=25 | 5.5 (4.57)
  Total Bilirubin, Visit 26 (Month 96), n=26: number analyzed (Participants) | 26
  Total Bilirubin, Visit 26 (Month 96), n=26 | 5.5 (6.59)
  Total Bilirubin, Visit 27 (Month 100), n=20: number analyzed (Participants) | 20
  Total Bilirubin, Visit 27 (Month 100), n=20 | 5.2 (6.29)
  Total Bilirubin, Visit 28 (Month 104), n=16: number analyzed (Participants) | 16
  Total Bilirubin, Visit 28 (Month 104), n=16 | 5.8 (5.01)
  Total Bilirubin, Visit 29 (Month 108), n=13: number analyzed (Participants) | 13
  Total Bilirubin, Visit 29 (Month 108), n=13 | 5.5 (8.32)
  Total Bilirubin, Visit 30 (Month 112), n=4: number analyzed (Participants) | 4
  Total Bilirubin, Visit 30 (Month 112), n=4 | 5.0 (3.65)
  Total Bilirubin, Visit 31 (Month 116), n=3: number analyzed (Participants) | 3
  Total Bilirubin, Visit 31 (Month 116), n=3 | 2.7 (6.03)
  Total Bilirubin, Visit 32 (Month 120), n=1: number analyzed (Participants) | 1
  Total Bilirubin, Visit 32 (Month 120), n=1 | 11.0 (NA) — Standard deviation could not be calculated as only 1 participant was analyzed.
  Total Bilirubin, Follow up, n=258: number analyzed (Participants) | 258
  Total Bilirubin, Follow up, n=258 | 0.0 (2.92)
  Uric acid, Visit 1 (Month 1), n=352: number analyzed (Participants) | 352
  Uric acid, Visit 1 (Month 1), n=352 | 2.1 (38.02)
  Uric acid, Visit 1a (Month 2), n=1: number analyzed (Participants) | 1
  Uric acid, Visit 1a (Month 2), n=1 | 41.0 (NA) — Standard deviation could not be calculated as only 1 participant was analyzed
  Uric acid, Visit 2 (Month 3), n=322: number analyzed (Participants) | 322
  Uric acid, Visit 2 (Month 3), n=322 | 5.5 (42.30)
  Uric acid, Visit 2a (Month 4), n=1: number analyzed (Participants) | 1
  Uric acid, Visit 2a (Month 4), n=1 | 107.0 (NA) — Standard deviation could not be calculated as only 1 participant was analyzed
  Uric acid, Visit 3 (Month 6), n=279: number analyzed (Participants) | 279
  Uric acid, Visit 3 (Month 6), n=279 | 4.3 (44.39)
  Uric acid, Visit 4 (Month 9), n=248: number analyzed (Participants) | 248
  Uric acid, Visit 4 (Month 9), n=248 | 7.8 (41.60)
  Uric acid, Visit 5 (Month 12), n=228: number analyzed (Participants) | 228
  Uric acid, Visit 5 (Month 12), n=228 | 5.3 (45.90)
  Uric acid, Visit 6 (Month 16), n=200: number analyzed (Participants) | 200
  Uric acid, Visit 6 (Month 16), n=200 | 7.9 (49.61)
  Uric acid, Visit 7 (Month 20), n=176: number analyzed (Participants) | 176
  Uric acid, Visit 7 (Month 20), n=176 | 8.8 (50.55)
  Uric acid, Visit 8 (Month 24), n=163: number analyzed (Participants) | 163
  Uric acid, Visit 8 (Month 24), n=163 | 10.1 (54.77)
  Uric acid, Visit 9 (Month 28), n=142: number analyzed (Participants) | 142
  Uric acid, Visit 9 (Month 28), n=142 | 7.7 (59.32)
  Uric acid, Visit 10 (Month 32), n=126: number analyzed (Participants) | 126
  Uric acid, Visit 10 (Month 32), n=126 | 8.7 (55.37)
  Uric acid, Visit 11 (Month 36), n=116: number analyzed (Participants) | 116
  Uric acid, Visit 11 (Month 36), n=116 | 9.8 (55.78)
  Uric acid, Visit 12 (Month 40), n=108: number analyzed (Participants) | 108
  Uric acid, Visit 12 (Month 40), n=108 | 13.8 (64.68)
  Uric acid, Visit 13 (Month 44), n=101: number analyzed (Participants) | 101
  Uric acid, Visit 13 (Month 44), n=101 | 13.4 (61.73)
  Uric acid, Visit 14 (Month 48), n=101: number analyzed (Participants) | 101
  Uric acid, Visit 14 (Month 48), n=101 | 6.8 (61.69)
  Uric acid, Visit 15 (Month 52), n=88: number analyzed (Participants) | 88
  Uric acid, Visit 15 (Month 52), n=88 | 14.2 (69.08)
  Uric acid, Visit 16 (Month 56), n=76: number analyzed (Participants) | 76
  Uric acid, Visit 16 (Month 56), n=76 | 12.0 (60.26)
  Uric acid, Visit 17 (Month 60), n=90: number analyzed (Participants) | 90
  Uric acid, Visit 17 (Month 60), n=90 | 14.7 (61.14)
  Uric acid, Visit 18 (Month 64), n=55: number analyzed (Participants) | 55
  Uric acid, Visit 18 (Month 64), n=55 | 14.8 (58.21)
  Uric acid, Visit 19 (Month 68), n=50: number analyzed (Participants) | 50
  Uric acid, Visit 19 (Month 68), n=50 | 25.2 (62.64)
  Uric acid, Visit 20 (Month 72), n=58: number analyzed (Participants) | 58
  Uric acid, Visit 20 (Month 72), n=58 | 14.4 (62.38)
  Uric acid, Visit 21 (Month 76), n=40: number analyzed (Participants) | 40
  Uric acid, Visit 21 (Month 76), n=40 | 25.5 (67.33)
  Uric acid, Visit 22 (Month 80), n=35: number analyzed (Participants) | 35
  Uric acid, Visit 22 (Month 80), n=35 | 18.3 (63.64)
  Uric acid, Visit 23 (Month 84), n=32: number analyzed (Participants) | 32
  Uric acid, Visit 23 (Month 84), n=32 | 21.4 (60.20)
  Uric acid, Visit 24 (Month 88), n=28: number analyzed (Participants) | 28
  Uric acid, Visit 24 (Month 88), n=28 | 14.0 (72.96)
  Uric acid, Visit 25 (Month 92), n=25: number analyzed (Participants) | 25
  Uric acid, Visit 25 (Month 92), n=25 | 29.6 (79.56)
  Uric acid, Visit 26 (Month 96), n=26: number analyzed (Participants) | 26
  Uric acid, Visit 26 (Month 96), n=26 | 14.3 (69.23)
  Uric acid, Visit 27 (Month 100), n=20: number analyzed (Participants) | 20
  Uric acid, Visit 27 (Month 100), n=20 | 14.2 (71.63)
  Uric acid, Visit 28 (Month 104), n=16: number analyzed (Participants) | 16
  Uric acid, Visit 28 (Month 104), n=16 | -1.8 (59.67)
  Uric acid, Visit 29 (Month 108), n=13: number analyzed (Participants) | 13
  Uric acid, Visit 29 (Month 108), n=13 | 9.2 (74.02)
  Uric acid, Visit 30 (Month 112), n=4: number analyzed (Participants) | 4
  Uric acid, Visit 30 (Month 112), n=4 | 46.3 (87.78)
  Uric acid, Visit 31 (Month 116), n=3: number analyzed (Participants) | 3
  Uric acid, Visit 31 (Month 116), n=3 | -8.0 (37.24)
  Uric acid, Visit 32 (Month 120), n=1: number analyzed (Participants) | 1
  Uric acid, Visit 32 (Month 120), n=1 | -23.0 (NA) — Standard deviation could not be calculated as only 1 participant was analyzed
  Uric acid, Follow up, n=261: number analyzed (Participants) | 261
  Uric acid, Follow up, n=261 | 11.7 (45.09)

12. Primary Outcome: Change From Baseline in Total Protein
Description: Clinical chemistry parameter included total protein. The clinical laboratory evaluation were performed at all study visits during the Open-Label Treatment Phase. Baseline assessment in this OLE study was defined as the last assessment of that endpoint in VRX-RET-E22-302 taken prior to the first active treatment with retigabine. Change from Baseline was calculated by subtracting the Baseline value from the post Baseline values. NA indicates standard deviation could not be calculated as only 1 participant was analyzed. Only those participants with data available at the specified time points were analyzed (represented by n=X in the category titles).
Time Frame: Baseline and up to 122 months
Population: Safety Population
Measure: Mean (Standard Deviation); unit: Grams per liter
Arm/Group | Retigabine
Number analyzed (Participants) | 376
Grams per liter
  Total Protein, Visit 1 (Month 1), n=352: number analyzed (Participants) | 352
  Total Protein, Visit 1 (Month 1), n=352 | -1.1 (4.32)
  Total Protein, Visit 1a (Month 2), n=1: number analyzed (Participants) | 1
  Total Protein, Visit 1a (Month 2), n=1 | -12.0 (NA) — Standard deviation could not be calculated as only 1 participant was analyzed.
  Total Protein, Visit 2 (Month 3), n=322: number analyzed (Participants) | 322
  Total Protein, Visit 2 (Month 3), n=322 | -0.8 (4.34)
  Total Protein, Visit 2a (Month 4), n=1: number analyzed (Participants) | 1
  Total Protein, Visit 2a (Month 4), n=1 | -3.0 (NA) — Standard deviation could not be calculated as only 1 participant was analyzed.
  Total Protein, Visit 3 (Month 6), n=279: number analyzed (Participants) | 279
  Total Protein, Visit 3 (Month 6), n=279 | -1.1 (4.18)
  Total Protein, Visit 4 (Month 9), n=248: number analyzed (Participants) | 248
  Total Protein, Visit 4 (Month 9), n=248 | -1.8 (5.42)
  Total Protein, Visit 5 (Month 12), n=228: number analyzed (Participants) | 228
  Total Protein, Visit 5 (Month 12), n=228 | -1.6 (4.34)
  Total Protein, Visit 6 (Month 16), n=200: number analyzed (Participants) | 200
  Total Protein, Visit 6 (Month 16), n=200 | -1.3 (4.24)
  Total Protein, Visit 7 (Month 20), n=176: number analyzed (Participants) | 176
  Total Protein, Visit 7 (Month 20), n=176 | -1.8 (4.19)
  Total Protein, Visit 8 (Month 24), n=163: number analyzed (Participants) | 163
  Total Protein, Visit 8 (Month 24), n=163 | -1.5 (4.25)
  Total Protein, Visit 9 (Month 28), n=142: number analyzed (Participants) | 142
  Total Protein, Visit 9 (Month 28), n=142 | -1.5 (4.22)
  Total Protein, Visit 10 (Month 32), n=126: number analyzed (Participants) | 126
  Total Protein, Visit 10 (Month 32), n=126 | -1.3 (4.62)
  Total Protein, Visit 11 (Month 36), n=116: number analyzed (Participants) | 116
  Total Protein, Visit 11 (Month 36), n=116 | -2.1 (4.35)
  Total Protein, Visit 12 (Month 40), n=108: number analyzed (Participants) | 108
  Total Protein, Visit 12 (Month 40), n=108 | -1.9 (4.36)
  Total Protein, Visit 13 (Month 44), n=101: number analyzed (Participants) | 101
  Total Protein, Visit 13 (Month 44), n=101 | -1.8 (4.10)
  Total Protein, Visit 14 (Month 48), n=101: number analyzed (Participants) | 101
  Total Protein, Visit 14 (Month 48), n=101 | -2.0 (4.37)
  Total Protein, Visit 15 (Month 52), n=88: number analyzed (Participants) | 88
  Total Protein, Visit 15 (Month 52), n=88 | -1.9 (4.81)
  Total Protein, Visit 16 (Month 56), n=76: number analyzed (Participants) | 76
  Total Protein, Visit 16 (Month 56), n=76 | -2.1 (4.18)
  Total Protein, Visit 17 (Month 60), n=90: number analyzed (Participants) | 90
  Total Protein, Visit 17 (Month 60), n=90 | -2.4 (4.29)
  Total Protein, Visit 18 (Month 64), n=55: number analyzed (Participants) | 55
  Total Protein, Visit 18 (Month 64), n=55 | -2.2 (4.12)
  Total Protein, Visit 19 (Month 68), n=50: number analyzed (Participants) | 50
  Total Protein, Visit 19 (Month 68), n=50 | -2.2 (3.95)
  Total Protein, Visit 20 (Month 72), n=58: number analyzed (Participants) | 58
  Total Protein, Visit 20 (Month 72), n=58 | -3.0 (4.85)
  Total Protein, Visit 21 (Month 76), n=40: number analyzed (Participants) | 40
  Total Protein, Visit 21 (Month 76), n=40 | -1.8 (4.01)
  Total Protein, Visit 22 (Month 80), n=35: number analyzed (Participants) | 35
  Total Protein, Visit 22 (Month 80), n=35 | -0.6 (5.09)
  Total Protein, Visit 23 (Month 84), n=32: number analyzed (Participants) | 32
  Total Protein, Visit 23 (Month 84), n=32 | -2.2 (4.38)
  Total Protein, Visit 24 (Month 88), n=28: number analyzed (Participants) | 28
  Total Protein, Visit 24 (Month 88), n=28 | -1.9 (4.63)
  Total Protein, Visit 25 (Month 92), n=25: number analyzed (Participants) | 25
  Total Protein, Visit 25 (Month 92), n=25 | -1.2 (4.82)
  Total Protein, Visit 26 (Month 96), n=26: number analyzed (Participants) | 26
  Total Protein, Visit 26 (Month 96), n=26 | -1.1 (5.32)
  Total Protein, Visit 27 (Month 100), n=20: number analyzed (Participants) | 20
  Total Protein, Visit 27 (Month 100), n=20 | -0.9 (4.08)
  Total Protein, Visit 28 (Month 104), n=16: number analyzed (Participants) | 16
  Total Protein, Visit 28 (Month 104), n=16 | -0.2 (4.68)
  Total Protein, Visit 29 (Month 108), n=13: number analyzed (Participants) | 13
  Total Protein, Visit 29 (Month 108), n=13 | -2.1 (4.57)
  Total Protein, Visit 30 (Month 112), n=4: number analyzed (Participants) | 4
  Total Protein, Visit 30 (Month 112), n=4 | 0.8 (2.36)
  Total Protein, Visit 31 (Month 116), n=3: number analyzed (Participants) | 3
  Total Protein, Visit 31 (Month 116), n=3 | -4.7 (0.58)
  Total Protein, Visit 32 (Month 120), n=1: number analyzed (Participants) | 1
  Total Protein, Visit 32 (Month 120), n=1 | -4.0 (NA) — Standard deviation could not be calculated as only 1 participant was analyzed.
  Total Protein, Follow up, n=261: number analyzed (Participants) | 261
  Total Protein, Follow up, n=261 | -1.1 (4.75)

13. Primary Outcome: Change From Baseline in Basophils, Eosinophils, Lymphocytes, Monocytes, Neutrophils, Platelet Count, White Blood Cells (WBC)
Description: Hematology parameters included eosinophils, basophils lymphocytes, monocytes, neutrophils, platelet count , and WBC. The clinical laboratory evaluations were performed at all study visits during the Open-Label Treatment Phase. Baseline assessment in this OLE study was defined as the last assessment of that endpoint in VRX-RET-E22-302 taken prior to the first active treatment with retigabine. Change from Baseline was calculated by subtracting the Baseline value from the post Baseline values. NA indicates standard deviation could not be calculated as only 1 participant was analyzed. Only those participants with data available at the specified time points were analyzed (represented by n=X in the category titles).
Time Frame: Baseline and up to 122 months
Population: Safety Population
Measure: Mean (Standard Deviation); unit: 10^9 cells per Liter
Arm/Group | Retigabine
Number analyzed (Participants) | 376
10^9 cells per Liter
  Basophils, Visit 1 (Month 1), n=345: number analyzed (Participants) | 345
  Basophils, Visit 1 (Month 1), n=345 | 0.003 (0.0261)
  Basophils, Visit 1a (Month 2), n=64: number analyzed (Participants) | 64
  Basophils, Visit 1a (Month 2), n=64 | 0.013 (0.0340)
  Basophils, Visit 2 (Month 3), n=309: number analyzed (Participants) | 309
  Basophils, Visit 2 (Month 3), n=309 | 0.001 (0.0251)
  Basophils, Visit 2a (Month 4), n=82: number analyzed (Participants) | 82
  Basophils, Visit 2a (Month 4), n=82 | 0.021 (0.0488)
  Basophils, Visit 3 (Month 6), n=273: number analyzed (Participants) | 273
  Basophils, Visit 3 (Month 6), n=273 | 0.003 (0.0340)
  Basophils, Visit 3a (Month 8), n=97: number analyzed (Participants) | 97
  Basophils, Visit 3a (Month 8), n=97 | 0.005 (0.0300)
  Basophils, Visit 4 (Month 9), n=239: number analyzed (Participants) | 239
  Basophils, Visit 4 (Month 9), n=239 | 0.000 (0.0222)
  Basophils, Visit 4a (Month 10), n=111: number analyzed (Participants) | 111
  Basophils, Visit 4a (Month 10), n=111 | 0.003 (0.0276)
  Basophils, Visit 5 (Month 12), n=225: number analyzed (Participants) | 225
  Basophils, Visit 5 (Month 12), n=225 | 0.002 (0.0188)
  Basophils, Visit 6 (Month 16), n=198: number analyzed (Participants) | 198
  Basophils, Visit 6 (Month 16), n=198 | 0.002 (0.0215)
  Basophils, Visit 7 (Month 20), n=173: number analyzed (Participants) | 173
  Basophils, Visit 7 (Month 20), n=173 | 0.003 (0.0230)
  Basophils, Visit 8 (Month 24), n=159: number analyzed (Participants) | 159
  Basophils, Visit 8 (Month 24), n=159 | 0.001 (0.0205)
  Basophils, Visit 9 (Month 28), n=139: number analyzed (Participants) | 139
  Basophils, Visit 9 (Month 28), n=139 | 0.005 (0.0200)
  Basophils, Visit 10 (Month 32), n=125: number analyzed (Participants) | 125
  Basophils, Visit 10 (Month 32), n=125 | 0.008 (0.0229)
  Basophils, Visit 11 (Month 36), n=112: number analyzed (Participants) | 112
  Basophils, Visit 11 (Month 36), n=112 | 0.005 (0.0200)
  Basophils, Visit 12 (Month 40), n=108: number analyzed (Participants) | 108
  Basophils, Visit 12 (Month 40), n=108 | 0.007 (0.0253)
  Basophils, Visit 13 (Month 44), n=98: number analyzed (Participants) | 98
  Basophils, Visit 13 (Month 44), n=98 | 0.002 (0.0157)
  Basophils, Visit 14 (Month 48), n=100: number analyzed (Participants) | 100
  Basophils, Visit 14 (Month 48), n=100 | 0.002 (0.0201)
  Basophils, Visit 15 (Month 52), n=88: number analyzed (Participants) | 88
  Basophils, Visit 15 (Month 52), n=88 | 0.005 (0.0249)
  Basophils, Visit 16 (Month 56), n=75: number analyzed (Participants) | 75
  Basophils, Visit 16 (Month 56), n=75 | 0.006 (0.0245)
  Basophils, Visit 17 (Month 60), n=89: number analyzed (Participants) | 89
  Basophils, Visit 17 (Month 60), n=89 | 0.006 (0.0186)
  Basophils, Visit 18 (Month 64), n=51: number analyzed (Participants) | 51
  Basophils, Visit 18 (Month 64), n=51 | 0.005 (0.0334)
  Basophils, Visit 19 (Month 68), n=50: number analyzed (Participants) | 50
  Basophils, Visit 19 (Month 68), n=50 | 0.006 (0.0184)
  Basophils, Visit 20 (Month 72), n=54: number analyzed (Participants) | 54
  Basophils, Visit 20 (Month 72), n=54 | 0.005 (0.0173)
  Basophils, Visit 21 (Month 76), n=39: number analyzed (Participants) | 39
  Basophils, Visit 21 (Month 76), n=39 | 0.009 (0.0226)
  Basophils, Visit 22 (Month 80), n=35: number analyzed (Participants) | 35
  Basophils, Visit 22 (Month 80), n=35 | 0.004 (0.0140)
  Basophils, Visit 23 (Month 84), n=32: number analyzed (Participants) | 32
  Basophils, Visit 23 (Month 84), n=32 | 0.009 (0.0178)
  Basophils, Visit 24 (Month 88), n=27: number analyzed (Participants) | 27
  Basophils, Visit 24 (Month 88), n=27 | 0.004 (0.0189)
  Basophils, Visit 25 (Month 92), n=25: number analyzed (Participants) | 25
  Basophils, Visit 25 (Month 92), n=25 | 0.013 (0.0281)
  Basophils, Visit 26 (Month 96), n=24: number analyzed (Participants) | 24
  Basophils, Visit 26 (Month 96), n=24 | 0.010 (0.0254)
  Basophils, Visit 27 (Month 100), n=20: number analyzed (Participants) | 20
  Basophils, Visit 27 (Month 100), n=20 | 0.010 (0.0192)
  Basophils, Visit 28 (Month 104), n=16: number analyzed (Participants) | 16
  Basophils, Visit 28 (Month 104), n=16 | 0.008 (0.0118)
  Basophils, Visit 29 (Month 108), n=13: number analyzed (Participants) | 13
  Basophils, Visit 29 (Month 108), n=13 | 0.005 (0.0156)
  Basophils, Visit 30 (Month 112), n=4: number analyzed (Participants) | 4
  Basophils, Visit 30 (Month 112), n=4 | 0.003 (0.0171)
  Basophils, Visit 31 (Month 116), n=3: number analyzed (Participants) | 3
  Basophils, Visit 31 (Month 116), n=3 | -0.003 (0.0153)
  Basophils, Visit 32 (Month 120), n=1: number analyzed (Participants) | 1
  Basophils, Visit 32 (Month 120), n=1 | -0.020 (NA) — Standard deviation could not be calculated as only 1 participant was analyzed.
  Basophils, Follow up, n=252: number analyzed (Participants) | 252
  Basophils, Follow up, n=252 | 0.001 (0.0236)
  Eosinophils, Visit 1 (Month 1), n=345: number analyzed (Participants) | 345
  Eosinophils, Visit 1 (Month 1), n=345 | -0.006 (0.1045)
  Eosinophils, Visit 1a (Month 2), n=64: number analyzed (Participants) | 64
  Eosinophils, Visit 1a (Month 2), n=64 | -0.018 (0.0982)
  Eosinophils, Visit 2 (Month 3), n=309: number analyzed (Participants) | 309
  Eosinophils, Visit 2 (Month 3), n=309 | -0.006 (0.1061)
  Eosinophils, Visit 2a (Month 4), n=82: number analyzed (Participants) | 82
  Eosinophils, Visit 2a (Month 4), n=82 | -0.002 (0.1274)
  Eosinophils, Visit 3 (Month 6), n=273: number analyzed (Participants) | 273
  Eosinophils, Visit 3 (Month 6), n=273 | -0.009 (0.0941)
  Eosinophils, Visit 3a (Month 8), n=97: number analyzed (Participants) | 97
  Eosinophils, Visit 3a (Month 8), n=97 | -0.010 (0.1142)
  Eosinophils, Visit 4 (Month 9), n=239: number analyzed (Participants) | 239
  Eosinophils, Visit 4 (Month 9), n=239 | 0.001 (0.1148)
  Eosinophils, Visit 4a (Month 10), n=111: number analyzed (Participants) | 111
  Eosinophils, Visit 4a (Month 10), n=111 | -0.003 (0.1126)
  Eosinophils, Visit 5 (Month 12), n=225: number analyzed (Participants) | 225
  Eosinophils, Visit 5 (Month 12), n=225 | -0.005 (0.1160)
  Eosinophils, Visit 6 (Month 16), n=198: number analyzed (Participants) | 198
  Eosinophils, Visit 6 (Month 16), n=198 | -0.012 (0.1015)
  Eosinophils, Visit 7 (Month 20), n=173: number analyzed (Participants) | 173
  Eosinophils, Visit 7 (Month 20), n=173 | -0.008 (0.1070)
  Eosinophils, Visit 8 (Month 24), n=159: number analyzed (Participants) | 159
  Eosinophils, Visit 8 (Month 24), n=159 | -0.007 (0.0989)
  Eosinophils, Visit 9 (Month 28), n=139: number analyzed (Participants) | 139
  Eosinophils, Visit 9 (Month 28), n=139 | -0.013 (0.0972)
  Eosinophils, Visit 10 (Month 32), n=125: number analyzed (Participants) | 125
  Eosinophils, Visit 10 (Month 32), n=125 | -0.007 (0.0997)
  Eosinophils, Visit 11 (Month 36), n=112: number analyzed (Participants) | 112
  Eosinophils, Visit 11 (Month 36), n=112 | -0.004 (0.1042)
  Eosinophils, Visit 12 (Month 40), n=108: number analyzed (Participants) | 108
  Eosinophils, Visit 12 (Month 40), n=108 | -0.006 (0.1044)
  Eosinophils, Visit 13 (Month 44), n=98: number analyzed (Participants) | 98
  Eosinophils, Visit 13 (Month 44), n=98 | -0.007 (0.0962)
  Eosinophils, Visit 14 (Month 48), n=100: number analyzed (Participants) | 100
  Eosinophils, Visit 14 (Month 48), n=100 | -0.018 (0.0973)
  Eosinophils, Visit 15 (Month 52), n=88: number analyzed (Participants) | 88
  Eosinophils, Visit 15 (Month 52), n=88 | -0.008 (0.1115)
  Eosinophils, Visit 16 (Month 56), n=75: number analyzed (Participants) | 75
  Eosinophils, Visit 16 (Month 56), n=75 | -0.008 (0.1051)
  Eosinophils, Visit 17 (Month 60), n=88: number analyzed (Participants) | 88
  Eosinophils, Visit 17 (Month 60), n=88 | 0.009 (0.1214)
  Eosinophils, Visit 18 (Month 64), n=51: number analyzed (Participants) | 51
  Eosinophils, Visit 18 (Month 64), n=51 | -0.001 (0.1298)
  Eosinophils, Visit 19 (Month 68), n=50: number analyzed (Participants) | 50
  Eosinophils, Visit 19 (Month 68), n=50 | -0.008 (0.1335)
  Eosinophils, Visit 20 (Month 72), n=54: number analyzed (Participants) | 54
  Eosinophils, Visit 20 (Month 72), n=54 | -0.002 (0.1235)
  Eosinophils, Visit 21 (Month 76), n=39: number analyzed (Participants) | 39
  Eosinophils, Visit 21 (Month 76), n=39 | 0.000 (0.1365)
  Eosinophils, Visit 22 (Month 80), n=35: number analyzed (Participants) | 35
  Eosinophils, Visit 22 (Month 80), n=35 | 0.000 (0.1352)
  Eosinophils, Visit 23 (Month 84), n=32: number analyzed (Participants) | 32
  Eosinophils, Visit 23 (Month 84), n=32 | 0.015 (0.1251)
  Eosinophils, Visit 24 (Month 88), n=27: number analyzed (Participants) | 27
  Eosinophils, Visit 24 (Month 88), n=27 | -0.022 (0.1272)
  Eosinophils, Visit 25 (Month 92), n=25: number analyzed (Participants) | 25
  Eosinophils, Visit 25 (Month 92), n=25 | -0.004 (0.1064)
  Eosinophils, Visit 26 (Month 96), n=24: number analyzed (Participants) | 24
  Eosinophils, Visit 26 (Month 96), n=24 | -0.007 (0.1082)
  Eosinophils, Visit 27 (Month 100), n=20: number analyzed (Participants) | 20
  Eosinophils, Visit 27 (Month 100), n=20 | 0.032 (0.1637)
  Eosinophils, Visit 28 (Month 104), n=16: number analyzed (Participants) | 16
  Eosinophils, Visit 28 (Month 104), n=16 | 0.041 (0.1509)
  Eosinophils, Visit 29 (Month 108), n=13: number analyzed (Participants) | 13
  Eosinophils, Visit 29 (Month 108), n=13 | 0.062 (0.1678)
  Eosinophils, Visit 30 (Month 112), n=4: number analyzed (Participants) | 4
  Eosinophils, Visit 30 (Month 112), n=4 | 0.185 (0.1933)
  Eosinophils, Visit 31 (Month 116), n=3: number analyzed (Participants) | 3
  Eosinophils, Visit 31 (Month 116), n=3 | 0.043 (0.0603)
  Eosinophils, Visit 32 (Month 120), n=1: number analyzed (Participants) | 1
  Eosinophils, Visit 32 (Month 120), n=1 | -0.020 (NA) — : Standard deviation could not be calculated as only 1 participant was analyzed.
  Eosinophils, Follow up, n=252: number analyzed (Participants) | 252
  Eosinophils, Follow up, n=252 | -0.010 (0.1082)
  Lymphocytes, Visit 1 (Month 1), n=345: number analyzed (Participants) | 345
  Lymphocytes, Visit 1 (Month 1), n=345 | -0.127 (0.4854)
  Lymphocytes, Visit 1a (Month 2), n=64: number analyzed (Participants) | 64
  Lymphocytes, Visit 1a (Month 2), n=64 | -0.029 (0.5459)
  Lymphocytes, Visit 2 (Month 3), n=309: number analyzed (Participants) | 309
  Lymphocytes, Visit 2 (Month 3), n=309 | -0.147 (0.4446)
  Lymphocytes, Visit 2a (Month 4), n=82: number analyzed (Participants) | 82
  Lymphocytes, Visit 2a (Month 4), n=82 | -0.089 (0.5561)
  Lymphocytes, Visit 3 (Month 6), n=273: number analyzed (Participants) | 273
  Lymphocytes, Visit 3 (Month 6), n=273 | -0.124 (0.4476)
  Lymphocytes, Visit 3a (Month 8), n=97: number analyzed (Participants) | 97
  Lymphocytes, Visit 3a (Month 8), n=97 | -0.104 (0.4733)
  Lymphocytes, Visit 4 (Month 9), n=239: number analyzed (Participants) | 239
  Lymphocytes, Visit 4 (Month 9), n=239 | -0.137 (0.4833)
  Lymphocytes, Visit 4a (Month 10), n=111: number analyzed (Participants) | 111
  Lymphocytes, Visit 4a (Month 10), n=111 | 0.007 (0.4505)
  Lymphocytes, Visit 5 (Month 12), n=225: number analyzed (Participants) | 225
  Lymphocytes, Visit 5 (Month 12), n=225 | -0.118 (0.4839)
  Lymphocytes, Visit 6 (Month 16), n=198: number analyzed (Participants) | 198
  Lymphocytes, Visit 6 (Month 16), n=198 | -0.130 (0.4605)
  Lymphocytes, Visit 7 (Month 20), n=173: number analyzed (Participants) | 173
  Lymphocytes, Visit 7 (Month 20), n=173 | -0.103 (0.4656)
  Lymphocytes, Visit 8 (Month 24), n=159: number analyzed (Participants) | 159
  Lymphocytes, Visit 8 (Month 24), n=159 | -0.091 (0.4387)
  Lymphocytes, Visit 9 (Month 28), n=139: number analyzed (Participants) | 139
  Lymphocytes, Visit 9 (Month 28), n=139 | -0.099 (0.4582)
  Lymphocytes, Visit 10 (Month 32), n=125: number analyzed (Participants) | 125
  Lymphocytes, Visit 10 (Month 32), n=125 | -0.103 (0.4502)
  Lymphocytes, Visit 11 (Month 36), n=112: number analyzed (Participants) | 112
  Lymphocytes, Visit 11 (Month 36), n=112 | -0.135 (0.4232)
  Lymphocytes, Visit 12 (Month 40), n=108: number analyzed (Participants) | 108
  Lymphocytes, Visit 12 (Month 40), n=108 | -0.114 (0.5521)
  Lymphocytes, Visit 13 (Month 44), n=98: number analyzed (Participants) | 98
  Lymphocytes, Visit 13 (Month 44), n=98 | -0.057 (0.4896)
  Lymphocytes, Visit 14 (Month 48), n=100: number analyzed (Participants) | 100
  Lymphocytes, Visit 14 (Month 48), n=100 | -0.117 (0.4672)
  Lymphocytes, Visit 15 (Month 52), n=88: number analyzed (Participants) | 88
  Lymphocytes, Visit 15 (Month 52), n=88 | -0.055 (0.4918)
  Lymphocytes, Visit 16 (Month 56), n=75: number analyzed (Participants) | 75
  Lymphocytes, Visit 16 (Month 56), n=75 | -0.049 (0.5077)
  Lymphocytes, Visit 17 (Month 60), n=88: number analyzed (Participants) | 88
  Lymphocytes, Visit 17 (Month 60), n=88 | -0.034 (0.5568)
  Lymphocytes, Visit 18 (Month 64), n=51: number analyzed (Participants) | 51
  Lymphocytes, Visit 18 (Month 64), n=51 | 0.004 (0.5778)
  Lymphocytes, Visit 19 (Month 68), n=50: number analyzed (Participants) | 50
  Lymphocytes, Visit 19 (Month 68), n=50 | 0.077 (0.5280)
  Lymphocytes, Visit 20 (Month 72), n=54: number analyzed (Participants) | 54
  Lymphocytes, Visit 20 (Month 72), n=54 | 0.000 (0.5129)
  Lymphocytes, Visit 21 (Month 76), n=39: number analyzed (Participants) | 39
  Lymphocytes, Visit 21 (Month 76), n=39 | 0.113 (0.5493)
  Lymphocytes, Visit 22 (Month 80), n=35: number analyzed (Participants) | 35
  Lymphocytes, Visit 22 (Month 80), n=35 | 0.110 (0.5896)
  Lymphocytes, Visit 23 (Month 84), n=32: number analyzed (Participants) | 32
  Lymphocytes, Visit 23 (Month 84), n=32 | 0.166 (0.4766)
  Lymphocytes, Visit 24 (Month 88), n=27: number analyzed (Participants) | 27
  Lymphocytes, Visit 24 (Month 88), n=27 | 0.133 (0.5958)
  Lymphocytes, Visit 25 (Month 92), n=25: number analyzed (Participants) | 25
  Lymphocytes, Visit 25 (Month 92), n=25 | 0.144 (0.3940)
  Lymphocytes, Visit 26 (Month 96), n=24: number analyzed (Participants) | 24
  Lymphocytes, Visit 26 (Month 96), n=24 | -0.001 (0.6195)
  Lymphocytes, Visit 27 (Month 100), n=20: number analyzed (Participants) | 20
  Lymphocytes, Visit 27 (Month 100), n=20 | 0.172 (0.5272)
  Lymphocytes, Visit 28 (Month 104), n=16: number analyzed (Participants) | 16
  Lymphocytes, Visit 28 (Month 104), n=16 | 0.141 (0.5226)
  Lymphocytes, Visit 29 (Month 108), n=13: number analyzed (Participants) | 13
  Lymphocytes, Visit 29 (Month 108), n=13 | 0.193 (0.5144)
  Lymphocytes, Visit 30 (Month 112), n=4: number analyzed (Participants) | 4
  Lymphocytes, Visit 30 (Month 112), n=4 | 0.278 (0.8945)
  Lymphocytes, Visit 31 (Month 116), n=3: number analyzed (Participants) | 3
  Lymphocytes, Visit 31 (Month 116), n=3 | 0.367 (0.4038)
  Lymphocytes, Visit 32 (Month 120), n=1: number analyzed (Participants) | 1
  Lymphocytes, Visit 32 (Month 120), n=1 | -0.130 (NA) — : Standard deviation could not be calculated as only 1 participant was analyzed.
  Lymphocytes, Follow up, n=252: number analyzed (Participants) | 252
  Lymphocytes, Follow up, n=252 | 0.022 (0.5031)
  Monocytes, Visit 1 (Month 1), n=345: number analyzed (Participants) | 345
  Monocytes, Visit 1 (Month 1), n=345 | 0.024 (0.1425)
  Monocytes, Visit 1a (Month 2), n=64: number analyzed (Participants) | 64
  Monocytes, Visit 1a (Month 2), n=64 | 0.085 (0.1846)
  Monocytes, Visit 2 (Month 3), n=309: number analyzed (Participants) | 309
  Monocytes, Visit 2 (Month 3), n=309 | 0.017 (0.1580)
  Monocytes, Visit 2a (Month 4), n=82: number analyzed (Participants) | 82
  Monocytes, Visit 2a (Month 4), n=82 | 0.071 (0.1850)
  Monocytes, Visit 3 (Month 6), n=273: number analyzed (Participants) | 273
  Monocytes, Visit 3 (Month 6), n=273 | 0.022 (0.1610)
  Monocytes, Visit 3a (Month 8), n=97: number analyzed (Participants) | 97
  Monocytes, Visit 3a (Month 8), n=97 | 0.073 (0.1581)
  Monocytes, Visit 4 (Month 9), n=239: number analyzed (Participants) | 239
  Monocytes, Visit 4 (Month 9), n=239 | 0.022 (0.1518)
  Monocytes, Visit 4a (Month 10), n=111: number analyzed (Participants) | 111
  Monocytes, Visit 4a (Month 10), n=111 | 0.080 (0.1653)
  Monocytes, Visit 5 (Month 12), n=225: number analyzed (Participants) | 225
  Monocytes, Visit 5 (Month 12), n=225 | 0.028 (0.1563)
  Monocytes, Visit 6 (Month 16), n=198: number analyzed (Participants) | 198
  Monocytes, Visit 6 (Month 16), n=198 | 0.023 (0.1598)
  Monocytes, Visit 7 (Month 20), n=173: number analyzed (Participants) | 173
  Monocytes, Visit 7 (Month 20), n=173 | 0.019 (0.1661)
  Monocytes, Visit 8 (Month 24), n=159: number analyzed (Participants) | 159
  Monocytes, Visit 8 (Month 24), n=159 | 0.038 (0.1840)
  Monocytes, Visit 9 (Month 28), n=139: number analyzed (Participants) | 139
  Monocytes, Visit 9 (Month 28), n=139 | 0.056 (0.1646)
  Monocytes, Visit 10 (Month 32), n=125: number analyzed (Participants) | 125
  Monocytes, Visit 10 (Month 32), n=125 | 0.047 (0.1597)
  Monocytes, Visit 11 (Month 36), n=112: number analyzed (Participants) | 112
  Monocytes, Visit 11 (Month 36), n=112 | 0.049 (0.1649)
  Monocytes, Visit 12 (Month 40), n=108: number analyzed (Participants) | 108
  Monocytes, Visit 12 (Month 40), n=108 | 0.040 (0.1750)
  Monocytes, Visit 13 (Month 44), n=98: number analyzed (Participants) | 98
  Monocytes, Visit 13 (Month 44), n=98 | 0.037 (0.1780)
  Monocytes, Visit 14 (Month 48), n=100: number analyzed (Participants) | 100
  Monocytes, Visit 14 (Month 48), n=100 | 0.033 (0.1442)
  Monocytes, Visit 15 (Month 52), n=88: number analyzed (Participants) | 88
  Monocytes, Visit 15 (Month 52), n=88 | 0.065 (0.1720)
  Monocytes, Visit 16 (Month 56), n=75: number analyzed (Participants) | 75
  Monocytes, Visit 16 (Month 56), n=75 | 0.043 (0.1632)
  Monocytes, Visit 17 (Month 60), n=88: number analyzed (Participants) | 88
  Monocytes, Visit 17 (Month 60), n=88 | 0.044 (0.1736)
  Monocytes, Visit 18 (Month 64), n=51: number analyzed (Participants) | 51
  Monocytes, Visit 18 (Month 64), n=51 | 0.028 (0.1644)
  Monocytes, Visit 19 (Month 68), n=50: number analyzed (Participants) | 50
  Monocytes, Visit 19 (Month 68), n=50 | 0.027 (0.1253)
  Monocytes, Visit 20 (Month 72), n=54: number analyzed (Participants) | 54
  Monocytes, Visit 20 (Month 72), n=54 | 0.039 (0.1201)
  Monocytes, Visit 21 (Month 76), n=39: number analyzed (Participants) | 39
  Monocytes, Visit 21 (Month 76), n=39 | 0.078 (0.2002)
  Monocytes, Visit 22 (Month 80), n=35: number analyzed (Participants) | 35
  Monocytes, Visit 22 (Month 80), n=35 | 0.046 (0.1629)
  Monocytes, Visit 23 (Month 84), n=32: number analyzed (Participants) | 32
  Monocytes, Visit 23 (Month 84), n=32 | 0.064 (0.1596)
  Monocytes, Visit 24 (Month 88), n=27: number analyzed (Participants) | 27
  Monocytes, Visit 24 (Month 88), n=27 | 0.065 (0.2083)
  Monocytes, Visit 25 (Month 92), n=25: number analyzed (Participants) | 25
  Monocytes, Visit 25 (Month 92), n=25 | 0.057 (0.1956)
  Monocytes, Visit 26 (Month 96), n=24: number analyzed (Participants) | 24
  Monocytes, Visit 26 (Month 96), n=24 | 0.035 (0.1405)
  Monocytes, Visit 27 (Month 100), n=20: number analyzed (Participants) | 20
  Monocytes, Visit 27 (Month 100), n=20 | 0.119 (0.1604)
  Monocytes, Visit 28 (Month 104), n=16: number analyzed (Participants) | 16
  Monocytes, Visit 28 (Month 104), n=16 | 0.039 (0.1903)
  Monocytes, Visit 29 (Month 108), n=13: number analyzed (Participants) | 13
  Monocytes, Visit 29 (Month 108), n=13 | 0.068 (0.2342)
  Monocytes, Visit 30 (Month 112), n=4: number analyzed (Participants) | 4
  Monocytes, Visit 30 (Month 112), n=4 | 0.030 (0.1985)
  Monocytes, Visit 31 (Month 116), n=3: number analyzed (Participants) | 3
  Monocytes, Visit 31 (Month 116), n=3 | -0.007 (0.0850)
  Monocytes, Visit 32 (Month 120), n=1: number analyzed (Participants) | 1
  Monocytes, Visit 32 (Month 120), n=1 | 0.080 (NA) — Standard deviation could not be calculated as only 1 participant was analyzed.
  Monocytes, Follow up, n=252: number analyzed (Participants) | 252
  Monocytes, Follow up, n=252 | 0.022 (0.1754)
  Neutrophils, Visit 1 (Month 1), n=345: number analyzed (Participants) | 345
  Neutrophils, Visit 1 (Month 1), n=345 | -0.143 (1.3093)
  Neutrophils, Visit 1a (Month 2), n=64: number analyzed (Participants) | 64
  Neutrophils, Visit 1a (Month 2), n=64 | -0.142 (1.3123)
  Neutrophils, Visit 2 (Month 3), n=309: number analyzed (Participants) | 309
  Neutrophils, Visit 2 (Month 3), n=309 | -0.045 (1.1768)
  Neutrophils, Visit 2a (Month 4), n=82: number analyzed (Participants) | 82
  Neutrophils, Visit 2a (Month 4), n=82 | 0.075 (1.4826)
  Neutrophils, Visit 3 (Month 6), n=273: number analyzed (Participants) | 273
  Neutrophils, Visit 3 (Month 6), n=273 | -0.087 (1.3700)
  Neutrophils, Visit 3a (Month 8), n=97: number analyzed (Participants) | 97
  Neutrophils, Visit 3a (Month 8), n=97 | -0.098 (1.3412)
  Neutrophils, Visit 4 (Month 9), n=239: number analyzed (Participants) | 239
  Neutrophils, Visit 4 (Month 9), n=239 | 0.032 (1.1933)
  Neutrophils, Visit 4a (Month 10), n=111: number analyzed (Participants) | 111
  Neutrophils, Visit 4a (Month 10), n=111 | 0.203 (1.3922)
  Neutrophils, Visit 5 (Month 12), n=225: number analyzed (Participants) | 225
  Neutrophils, Visit 5 (Month 12), n=225 | 0.015 (1.6014)
  Neutrophils, Visit 6 (Month 16), n=198: number analyzed (Participants) | 198
  Neutrophils, Visit 6 (Month 16), n=198 | 0.086 (1.3107)
  Neutrophils, Visit 7 (Month 20), n=173: number analyzed (Participants) | 173
  Neutrophils, Visit 7 (Month 20), n=173 | 0.121 (1.2780)
  Neutrophils, Visit 8 (Month 24), n=159: number analyzed (Participants) | 159
  Neutrophils, Visit 8 (Month 24), n=159 | 0.368 (1.4584)
  Neutrophils, Visit 9 (Month 28), n=139: number analyzed (Participants) | 139
  Neutrophils, Visit 9 (Month 28), n=139 | 0.188 (1.2575)
  Neutrophils, Visit 10 (Month 32), n=125: number analyzed (Participants) | 125
  Neutrophils, Visit 10 (Month 32), n=125 | 0.118 (1.1824)
  Neutrophils, Visit 11 (Month 36), n=112: number analyzed (Participants) | 112
  Neutrophils, Visit 11 (Month 36), n=112 | 0.057 (1.2868)
  Neutrophils, Visit 12 (Month 40), n=108: number analyzed (Participants) | 108
  Neutrophils, Visit 12 (Month 40), n=108 | 0.196 (1.1770)
  Neutrophils, Visit 13 (Month 44), n=98: number analyzed (Participants) | 98
  Neutrophils, Visit 13 (Month 44), n=98 | 0.243 (1.4180)
  Neutrophils, Visit 14 (Month 48), n=100: number analyzed (Participants) | 100
  Neutrophils, Visit 14 (Month 48), n=100 | 0.095 (1.2410)
  Neutrophils, Visit 15 (Month 52), n=88: number analyzed (Participants) | 88
  Neutrophils, Visit 15 (Month 52), n=88 | 0.432 (1.4504)
  Neutrophils, Visit 16 (Month 56), n=75: number analyzed (Participants) | 75
  Neutrophils, Visit 16 (Month 56), n=75 | 0.412 (1.4045)
  Neutrophils, Visit 17 (Month 60), n=88: number analyzed (Participants) | 88
  Neutrophils, Visit 17 (Month 60), n=88 | 0.416 (1.3905)
  Neutrophils, Visit 18 (Month 64), n=51: number analyzed (Participants) | 51
  Neutrophils, Visit 18 (Month 64), n=51 | 0.296 (1.2674)
  Neutrophils, Visit 19 (Month 68), n=50: number analyzed (Participants) | 50
  Neutrophils, Visit 19 (Month 68), n=50 | 0.436 (1.0379)
  Neutrophils, Visit 20 (Month 72), n=54: number analyzed (Participants) | 54
  Neutrophils, Visit 20 (Month 72), n=54 | 0.552 (1.3322)
  Neutrophils, Visit 21 (Month 76), n=39: number analyzed (Participants) | 39
  Neutrophils, Visit 21 (Month 76), n=39 | 0.639 (1.5548)
  Neutrophils, Visit 22 (Month 80), n=35: number analyzed (Participants) | 35
  Neutrophils, Visit 22 (Month 80), n=35 | 0.346 (1.3809)
  Neutrophils, Visit 23 (Month 84), n=32: number analyzed (Participants) | 32
  Neutrophils, Visit 23 (Month 84), n=32 | 0.560 (1.4536)
  Neutrophils, Visit 24 (Month 88), n=27: number analyzed (Participants) | 27
  Neutrophils, Visit 24 (Month 88), n=27 | 0.366 (1.8672)
  Neutrophils, Visit 25 (Month 92), n=25: number analyzed (Participants) | 25
  Neutrophils, Visit 25 (Month 92), n=25 | 0.130 (1.9387)
  Neutrophils, Visit 26 (Month 96), n=24: number analyzed (Participants) | 24
  Neutrophils, Visit 26 (Month 96), n=24 | 0.707 (1.7085)
  Neutrophils, Visit 27 (Month 100), n=20: number analyzed (Participants) | 20
  Neutrophils, Visit 27 (Month 100), n=20 | 0.247 (1.6045)
  Neutrophils, Visit 28 (Month 104), n=16: number analyzed (Participants) | 16
  Neutrophils, Visit 28 (Month 104), n=16 | 0.458 (1.1406)
  Neutrophils, Visit 29 (Month 108), n=13: number analyzed (Participants) | 13
  Neutrophils, Visit 29 (Month 108), n=13 | -0.027 (1.4607)
  Neutrophils, Visit 30 (Month 112), n=4: number analyzed (Participants) | 4
  Neutrophils, Visit 30 (Month 112), n=4 | 0.658 (1.2219)
  Neutrophils, Visit 31 (Month 116), n=3: number analyzed (Participants) | 3
  Neutrophils, Visit 31 (Month 116), n=3 | 0.297 (0.5320)
  Neutrophils, Visit 32 (Month 120), n=1: number analyzed (Participants) | 1
  Neutrophils, Visit 32 (Month 120), n=1 | 0.470 (NA) — Standard deviation could not be calculated as only 1 participant was analyzed
  Neutrophils, Follow up, n=252: number analyzed (Participants) | 252
  Neutrophils, Follow up, n=252 | -0.010 (1.5258)
  Platelet Count, Visit 1 (Month 1), n=345: number analyzed (Participants) | 345
  Platelet Count, Visit 1 (Month 1), n=345 | 0.9 (40.69)
  Platelet count, Visit 1a (Month 2), n=65: number analyzed (Participants) | 65
  Platelet count, Visit 1a (Month 2), n=65 | 6.4 (41.67)
  Platelet count, Visit 2 (Month 3), n=311: number analyzed (Participants) | 311
  Platelet count, Visit 2 (Month 3), n=311 | 0.7 (37.59)
  Platelet count, Visit 2a (Month 4), n=82: number analyzed (Participants) | 82
  Platelet count, Visit 2a (Month 4), n=82 | 12.7 (37.26)
  Platelet count, Visit 3 (Month 6), n=273: number analyzed (Participants) | 273
  Platelet count, Visit 3 (Month 6), n=273 | -1.7 (41.28)
  Platelet count, Visit 3a (Month 8), n=99: number analyzed (Participants) | 99
  Platelet count, Visit 3a (Month 8), n=99 | -5.3 (31.49)
  Platelet count, Visit 4 (Month 9), n=241: number analyzed (Participants) | 241
  Platelet count, Visit 4 (Month 9), n=241 | -7.1 (37.88)
  Platelet count, Visit 4a (Month 10), n=108: number analyzed (Participants) | 108
  Platelet count, Visit 4a (Month 10), n=108 | -2.8 (38.71)
  Platelet count, Visit 5 (Month 12), n=225: number analyzed (Participants) | 225
  Platelet count, Visit 5 (Month 12), n=225 | -8.6 (35.57)
  Platelet count, Visit 6 (Month 16), n=196: number analyzed (Participants) | 196
  Platelet count, Visit 6 (Month 16), n=196 | -9.0 (43.09)
  Platelet count, Visit 7 (Month 20), n=171: number analyzed (Participants) | 171
  Platelet count, Visit 7 (Month 20), n=171 | -15.8 (41.13)
  Platelet count, Visit 8 (Month 24), n=162: number analyzed (Participants) | 162
  Platelet count, Visit 8 (Month 24), n=162 | -17.3 (44.99)
  Platelet count, Visit 9 (Month 28), n=137: number analyzed (Participants) | 137
  Platelet count, Visit 9 (Month 28), n=137 | -18.0 (44.47)
  Platelet count, Visit 10 (Month 32), n=124: number analyzed (Participants) | 124
  Platelet count, Visit 10 (Month 32), n=124 | -20.8 (38.96)
  Platelet count, Visit 11 (Month 36), n=114: number analyzed (Participants) | 114
  Platelet count, Visit 11 (Month 36), n=114 | -25.8 (42.66)
  Platelet count, Visit 12 (Month 40), n=108: number analyzed (Participants) | 108
  Platelet count, Visit 12 (Month 40), n=108 | -24.3 (39.96)
  Platelet count, Visit 13 (Month 44), n=98: number analyzed (Participants) | 98
  Platelet count, Visit 13 (Month 44), n=98 | -22.4 (37.92)
  Platelet count, Visit 14 (Month 48), n=98: number analyzed (Participants) | 98
  Platelet count, Visit 14 (Month 48), n=98 | -25.2 (37.88)
  Platelet count, Visit 15 (Month 52), n=84: number analyzed (Participants) | 84
  Platelet count, Visit 15 (Month 52), n=84 | -22.3 (40.93)
  Platelet count, Visit 16 (Month 56), n=75: number analyzed (Participants) | 75
  Platelet count, Visit 16 (Month 56), n=75 | -17.1 (50.19)
  Platelet count, Visit 17 (Month 60), n=88: number analyzed (Participants) | 88
  Platelet count, Visit 17 (Month 60), n=88 | -18.6 (46.11)
  Platelet count, Visit 18 (Month 64), n=54: number analyzed (Participants) | 54
  Platelet count, Visit 18 (Month 64), n=54 | -23.1 (38.78)
  Platelet count, Visit 19 (Month 68), n=50: number analyzed (Participants) | 50
  Platelet count, Visit 19 (Month 68), n=50 | -17.7 (42.66)
  Platelet count, Visit 20 (Month 72), n=53: number analyzed (Participants) | 53
  Platelet count, Visit 20 (Month 72), n=53 | -20.4 (51.90)
  Platelet count, Visit 21 (Month 76), n=40: number analyzed (Participants) | 40
  Platelet count, Visit 21 (Month 76), n=40 | -11.1 (55.97)
  Platelet count, Visit 22 (Month 80), n=34: number analyzed (Participants) | 34
  Platelet count, Visit 22 (Month 80), n=34 | -10.0 (57.22)
  Platelet count, Visit 23 (Month 84), n=31: number analyzed (Participants) | 31
  Platelet count, Visit 23 (Month 84), n=31 | -7.0 (50.20)
  Platelet count, Visit 24 (Month 88), n=25: number analyzed (Participants) | 25
  Platelet count, Visit 24 (Month 88), n=25 | -22.1 (29.77)
  Platelet count, Visit 25 (Month 92), n=25: number analyzed (Participants) | 25
  Platelet count, Visit 25 (Month 92), n=25 | -16.8 (40.54)
  Platelet count, Visit 26 (Month 96), n=24: number analyzed (Participants) | 24
  Platelet count, Visit 26 (Month 96), n=24 | -4.9 (43.76)
  Platelet count, Visit 27 (Month 100), n=20: number analyzed (Participants) | 20
  Platelet count, Visit 27 (Month 100), n=20 | 1.9 (45.98)
  Platelet count, Visit 28 (Month 104), n=16: number analyzed (Participants) | 16
  Platelet count, Visit 28 (Month 104), n=16 | -6.3 (44.81)
  Platelet count, Visit 29 (Month 108), n=13: number analyzed (Participants) | 13
  Platelet count, Visit 29 (Month 108), n=13 | -9.5 (41.54)
  Platelet count, Visit 30 (Month 112), n=4: number analyzed (Participants) | 4
  Platelet count, Visit 30 (Month 112), n=4 | 10.0 (32.44)
  Platelet count, Visit 31 (Month 116), n=3: number analyzed (Participants) | 3
  Platelet count, Visit 31 (Month 116), n=3 | -5.7 (30.09)
  Platelet count, Visit 32 (Month 120), n=1: number analyzed (Participants) | 1
  Platelet count, Visit 32 (Month 120), n=1 | 25.0 (NA) — Standard deviation could not be calculated as only 1 participant was analyzed.
  Platelet count, Follow up, n=249: number analyzed (Participants) | 249
  Platelet count, Follow up, n=249 | -9.4 (49.63)
  WBC, Visit 1 (Month 1), n=349: number analyzed (Participants) | 349
  WBC, Visit 1 (Month 1), n=349 | -0.25 (1.403)
  WBC, Visit 1a (Month 2), n=65: number analyzed (Participants) | 65
  WBC, Visit 1a (Month 2), n=65 | -0.11 (1.478)
  WBC, Visit 2 (Month 3), n=315: number analyzed (Participants) | 315
  WBC, Visit 2 (Month 3), n=315 | -0.22 (1.371)
  WBC, Visit 2a (Month 4), n=82: number analyzed (Participants) | 82
  WBC, Visit 2a (Month 4), n=82 | 0.07 (1.648)
  WBC, Visit 3 (Month 6), n=278: number analyzed (Participants) | 278
  WBC, Visit 3 (Month 6), n=278 | -0.20 (1.531)
  WBC, Visit 3a (Month 8), n=99: number analyzed (Participants) | 99
  WBC, Visit 3a (Month 8), n=99 | -0.15 (1.537)
  WBC, Visit 4 (Month 9), n=244: number analyzed (Participants) | 244
  WBC, Visit 4 (Month 9), n=244 | -0.08 (1.356)
  WBC, Visit 4a (Month 10), n=113: number analyzed (Participants) | 113
  WBC, Visit 4a (Month 10), n=113 | 0.28 (1.608)
  WBC, Visit 5 (Month 12), n=226: number analyzed (Participants) | 226
  WBC, Visit 5 (Month 12), n=226 | -0.09 (1.690)
  WBC, Visit 6 (Month 16), n=199: number analyzed (Participants) | 199
  WBC, Visit 6 (Month 16), n=199 | -0.06 (1.385)
  WBC, Visit 7 (Month 20), n=174: number analyzed (Participants) | 174
  WBC, Visit 7 (Month 20), n=174 | 0.01 (1.468)
  WBC, Visit 8 (Month 24), n=164: number analyzed (Participants) | 164
  WBC, Visit 8 (Month 24), n=164 | 0.25 (1.655)
  WBC, Visit 9 (Month 28), n=142: number analyzed (Participants) | 142
  WBC, Visit 9 (Month 28), n=142 | 0.10 (1.367)
  WBC, Visit 10 (Month 32), n=126: number analyzed (Participants) | 126
  WBC, Visit 10 (Month 32), n=126 | 0.09 (1.374)
  WBC, Visit 11 (Month 36), n=115: number analyzed (Participants) | 115
  WBC, Visit 11 (Month 36), n=115 | -0.05 (1.387)
  WBC, Visit 12 (Month 40), n=109: number analyzed (Participants) | 109
  WBC, Visit 12 (Month 40), n=109 | 0.10 (1.514)
  WBC, Visit 13 (Month 44), n=98: number analyzed (Participants) | 98
  WBC, Visit 13 (Month 44), n=98 | 0.21 (1.687)
  WBC, Visit 14 (Month 48), n=101: number analyzed (Participants) | 101
  WBC, Visit 14 (Month 48), n=101 | -0.01 (1.381)
  WBC, Visit 15 (Month 52), n=88: number analyzed (Participants) | 88
  WBC, Visit 15 (Month 52), n=88 | 0.43 (1.648)
  WBC, Visit 16 (Month 56), n=76: number analyzed (Participants) | 76
  WBC, Visit 16 (Month 56), n=76 | 0.37 (1.603)
  WBC, Visit 17 (Month 60), n=89: number analyzed (Participants) | 89
  WBC, Visit 17 (Month 60), n=89 | 0.41 (1.663)
  WBC, Visit 18 (Month 64), n=54: number analyzed (Participants) | 54
  WBC, Visit 18 (Month 64), n=54 | 0.33 (1.613)
  WBC, Visit 19 (Month 68), n=50: number analyzed (Participants) | 50
  WBC, Visit 19 (Month 68), n=50 | 0.54 (1.376)
  WBC, Visit 20 (Month 72), n=55: number analyzed (Participants) | 55
  WBC, Visit 20 (Month 72), n=55 | 0.57 (1.532)
  WBC, Visit 21 (Month 76), n=40: number analyzed (Participants) | 40
  WBC, Visit 21 (Month 76), n=40 | 0.81 (1.940)
  WBC, Visit 22 (Month 80), n=35: number analyzed (Participants) | 35
  WBC, Visit 22 (Month 80), n=35 | 0.52 (1.622)
  WBC, Visit 23 (Month 84), n=32: number analyzed (Participants) | 32
  WBC, Visit 23 (Month 84), n=32 | 0.83 (1.599)
  WBC, Visit 24 (Month 88), n=27: number analyzed (Participants) | 27
  WBC, Visit 24 (Month 88), n=27 | 0.57 (1.964)
  WBC, Visit 25 (Month 92), n=25: number analyzed (Participants) | 25
  WBC, Visit 25 (Month 92), n=25 | 0.34 (2.114)
  WBC, Visit 26 (Month 96), n=24: number analyzed (Participants) | 24
  WBC, Visit 26 (Month 96), n=24 | 0.75 (1.670)
  WBC, Visit 27 (Month 100), n=20: number analyzed (Participants) | 20
  WBC, Visit 27 (Month 100), n=20 | 0.59 (1.809)
  WBC, Visit 28 (Month 104), n=16: number analyzed (Participants) | 16
  WBC, Visit 28 (Month 104), n=16 | 0.70 (1.372)
  WBC, Visit 29 (Month 108), n=13: number analyzed (Participants) | 13
  WBC, Visit 29 (Month 108), n=13 | 0.30 (1.614)
  WBC, Visit 30 (Month 112), n=4: number analyzed (Participants) | 4
  WBC, Visit 30 (Month 112), n=4 | 1.18 (1.864)
  WBC, Visit 31 (Month 116), n=3: number analyzed (Participants) | 3
  WBC, Visit 31 (Month 116), n=3 | 0.70 (0.800)
  WBC, Visit 32 (Month 120), n=1: number analyzed (Participants) | 1
  WBC, Visit 32 (Month 120), n=1 | 0.40 (NA) — Standard deviation could not be calculated as only 1 participant was analyzed.
  WBC, Follow up, n=255: number analyzed (Participants) | 255
  WBC, Follow up, n=255 | 0.02 (1.738)

14. Primary Outcome: Change From Baseline in Hematocrit
Description: Blood samples for the assessment of clinical laboratory parameter hematocrit were collected at all study visits during the Open-Label Treatment Phase. Baseline assessment in this OLE study was defined as the last assessment of that endpoint in VRX-RET-E22-302 taken prior to the first active treatment with retigabine. Change from Baseline was calculated by subtracting the Baseline value from the post Baseline values. NA indicates standard deviation could not be calculated as only 1 participant was analyzed. Only those participants with data available at the specified time points were analyzed (represented by n=X in the category titles).
Time Frame: Baseline and up to 122 months
Population: Safety Population
Measure: Mean (Standard Deviation); unit: Percentage of red blood cells in blood
Arm/Group | Retigabine
Number analyzed (Participants) | 376
Percentage of red blood cells in blood
  Hematocrit, Visit 1 (Month 1), n=340: number analyzed (Participants) | 340
  Hematocrit, Visit 1 (Month 1), n=340 | -0.009 (0.0215)
  Hematocrit, Visit 1a (Month 2), n=63: number analyzed (Participants) | 63
  Hematocrit, Visit 1a (Month 2), n=63 | -0.005 (0.0227)
  Hematocrit, Visit 2 (Month 3), n=308: number analyzed (Participants) | 308
  Hematocrit, Visit 2 (Month 3), n=308 | -0.004 (0.0229)
  Hematocrit, Visit 2a (Month 4), n=79: number analyzed (Participants) | 79
  Hematocrit, Visit 2a (Month 4), n=79 | -0.012 (0.0230)
  Hematocrit, Visit 3 (Month 6), n=274: number analyzed (Participants) | 274
  Hematocrit, Visit 3 (Month 6), n=274 | -0.005 (0.0244)
  Hematocrit, Visit 3a (Month 8), n=95: number analyzed (Participants) | 95
  Hematocrit, Visit 3a (Month 8), n=95 | -0.009 (0.0264)
  Hematocrit, Visit 4 (Month 9), n=231: number analyzed (Participants) | 231
  Hematocrit, Visit 4 (Month 9), n=231 | -0.002 (0.0263)
  Hematocrit, Visit 4a (Month 10), n=111: number analyzed (Participants) | 111
  Hematocrit, Visit 4a (Month 10), n=111 | -0.004 (0.0254)
  Hematocrit, Visit 5 (Month 12), n=223: number analyzed (Participants) | 223
  Hematocrit, Visit 5 (Month 12), n=223 | -0.004 (0.0256)
  Hematocrit, Visit 6 (Month 16), n=196: number analyzed (Participants) | 196
  Hematocrit, Visit 6 (Month 16), n=196 | -0.003 (0.0270)
  Hematocrit, Visit 7 (Month 20), n=166: number analyzed (Participants) | 166
  Hematocrit, Visit 7 (Month 20), n=166 | -0.001 (0.0255)
  Hematocrit, Visit 8 (Month 24), n=160: number analyzed (Participants) | 160
  Hematocrit, Visit 8 (Month 24), n=160 | 0.000 (0.0275)
  Hematocrit, Visit 9 (Month 28), n=141: number analyzed (Participants) | 141
  Hematocrit, Visit 9 (Month 28), n=141 | 0.005 (0.0260)
  Hematocrit, Visit 10 (Month 32), n=122: number analyzed (Participants) | 122
  Hematocrit, Visit 10 (Month 32), n=122 | 0.004 (0.0285)
  Hematocrit, Visit 11 (Month 36), n=113: number analyzed (Participants) | 113
  Hematocrit, Visit 11 (Month 36), n=113 | -0.001 (0.0301)
  Haematocrit, Visit 12 (Month 40), n=106: number analyzed (Participants) | 106
  Haematocrit, Visit 12 (Month 40), n=106 | 0.006 (0.0301)
  Hematocrit, Visit 13 (Month 44), n=95: number analyzed (Participants) | 95
  Hematocrit, Visit 13 (Month 44), n=95 | 0.003 (0.0274)
  Hematocrit, Visit 14 (Month 48), n=100: number analyzed (Participants) | 100
  Hematocrit, Visit 14 (Month 48), n=100 | -0.003 (0.0286)
  Hematocrit, Visit 15 (Month 52), n=88: number analyzed (Participants) | 88
  Hematocrit, Visit 15 (Month 52), n=88 | -0.001 (0.0289)
  Hematocrit, Visit 16 (Month 56), n=74: number analyzed (Participants) | 74
  Hematocrit, Visit 16 (Month 56), n=74 | -0.001 (0.0230)
  Haematocrit, Visit 17 (Month 60), n=88: number analyzed (Participants) | 88
  Haematocrit, Visit 17 (Month 60), n=88 | 0.000 (0.0314)
  Hematocrit, Visit 18 (Month 64), n=51: number analyzed (Participants) | 51
  Hematocrit, Visit 18 (Month 64), n=51 | 0.009 (0.0270)
  Hematocrit, Visit 19 (Month 68), n=50: number analyzed (Participants) | 50
  Hematocrit, Visit 19 (Month 68), n=50 | 0.008 (0.0278)
  Hematocrit, Visit 20 (Month 72), n=55: number analyzed (Participants) | 55
  Hematocrit, Visit 20 (Month 72), n=55 | 0.004 (0.0287)
  Hematocrit, Visit 21 (Month 76), n=39: number analyzed (Participants) | 39
  Hematocrit, Visit 21 (Month 76), n=39 | 0.010 (0.0377)
  Hematocrit, Visit 22 (Month 80), n=34: number analyzed (Participants) | 34
  Hematocrit, Visit 22 (Month 80), n=34 | 0.015 (0.0303)
  Hematocrit, Visit 23 (Month 84), n=30: number analyzed (Participants) | 30
  Hematocrit, Visit 23 (Month 84), n=30 | 0.000 (0.0344)
  Hematocrit, Visit 24 (Month 88), n=26: number analyzed (Participants) | 26
  Hematocrit, Visit 24 (Month 88), n=26 | 0.005 (0.0294)
  Hematocrit, Visit 25 (Month 92), n=24: number analyzed (Participants) | 24
  Hematocrit, Visit 25 (Month 92), n=24 | 0.016 (0.0264)
  Hematocrit, Visit 26 (Month 96), n=24: number analyzed (Participants) | 24
  Hematocrit, Visit 26 (Month 96), n=24 | 0.013 (0.0258)
  Hematocrit, Visit 27 (Month 100), n=20: number analyzed (Participants) | 20
  Hematocrit, Visit 27 (Month 100), n=20 | 0.016 (0.0201)
  Hematocrit, Visit 28 (Month 104), n=16: number analyzed (Participants) | 16
  Hematocrit, Visit 28 (Month 104), n=16 | 0.016 (0.0203)
  Hematocrit, Visit 29 (Month 108), n=13: number analyzed (Participants) | 13
  Hematocrit, Visit 29 (Month 108), n=13 | -0.002 (0.0268)
  Hematocrit, Visit 30 (Month 112), n=4: number analyzed (Participants) | 4
  Hematocrit, Visit 30 (Month 112), n=4 | 0.000 (0.0365)
  Hematocrit, Visit 31 (Month 116), n=3: number analyzed (Participants) | 3
  Hematocrit, Visit 31 (Month 116), n=3 | 0.033 (0.0666)
  Hematocrit, Visit 32 (Month 120), n=1: number analyzed (Participants) | 1
  Hematocrit, Visit 32 (Month 120), n=1 | 0.080 (NA) — Standard deviation could not be calculated as only 1 participant was analyzed.
  Hematocrit,Follow up, n=253: number analyzed (Participants) | 253
  Hematocrit,Follow up, n=253 | 0.003 (0.0262)

15. Primary Outcome: Change From Baseline in Hemoglobin
Description: The hematology parameters included hemoglobin. The clinical laboratory evaluations were performed at all study visits during the Open-Label Treatment Phase. Baseline assessment in this OLE study was defined as the last assessment of that endpoint in VRX-RET-E22-302 taken prior to the first active treatment with retigabine. Change from Baseline was calculated by subtracting the Baseline value from the post Baseline values. NA indicates standard deviation could not be calculated as only 1 participant was analyzed. Only those participants with data available at the specified time points were analyzed (represented by n=X in the category titles).
Time Frame: Baseline and up to 122 months
Population: Safety Population
Measure: Mean (Standard Deviation); unit: Grams per liter
Arm/Group | Retigabine
Number analyzed (Participants) | 376
Grams per liter
  Hemoglobin, Visit 1 (Month 1), n=349: number analyzed (Participants) | 349
  Hemoglobin, Visit 1 (Month 1), n=349 | -2.6 (6.96)
  Hemoglobin, Visit 1a (Month 2), n=65: number analyzed (Participants) | 65
  Hemoglobin, Visit 1a (Month 2), n=65 | -1.8 (7.30)
  Hemoglobin, Visit 2 (Month 3), n=316: number analyzed (Participants) | 316
  Hemoglobin, Visit 2 (Month 3), n=316 | -0.8 (7.89)
  Hemoglobin, Visit 2a (Month 4), n=82: number analyzed (Participants) | 82
  Hemoglobin, Visit 2a (Month 4), n=82 | -3.3 (8.11)
  Hemoglobin, Visit 3 (Month 6), n=279: number analyzed (Participants) | 279
  Hemoglobin, Visit 3 (Month 6), n=279 | -1.3 (8.21)
  Hemoglobin, Visit 3a (Month 8), n=99: number analyzed (Participants) | 99
  Hemoglobin, Visit 3a (Month 8), n=99 | -3.0 (8.70)
  Hemoglobin, Visit 4 (Month 9), n=244: number analyzed (Participants) | 244
  Hemoglobin, Visit 4 (Month 9), n=244 | -0.7 (8.87)
  Hemoglobin, Visit 4a (Month 10), n=113: number analyzed (Participants) | 113
  Hemoglobin, Visit 4a (Month 10), n=113 | -2.0 (8.41)
  Hemoglobin, Visit 5 (Month 12), n=226: number analyzed (Participants) | 226
  Hemoglobin, Visit 5 (Month 12), n=226 | -1.4 (8.64)
  Hemoglobin, Visit 6 (Month 16), n=199: number analyzed (Participants) | 199
  Hemoglobin, Visit 6 (Month 16), n=199 | -0.4 (8.83)
  Hemoglobin, Visit 7 (Month 20), n=174: number analyzed (Participants) | 174
  Hemoglobin, Visit 7 (Month 20), n=174 | -0.6 (9.01)
  Hemoglobin, Visit 8 (Month 24), n=164: number analyzed (Participants) | 164
  Hemoglobin, Visit 8 (Month 24), n=164 | -0.3 (8.58)
  Hemoglobin, Visit 9 (Month 28), n=142: number analyzed (Participants) | 142
  Hemoglobin, Visit 9 (Month 28), n=142 | 1.2 (8.99)
  Hemoglobin, Visit 10 (Month 32), n=126: number analyzed (Participants) | 126
  Hemoglobin, Visit 10 (Month 32), n=126 | 0.3 (9.58)
  Hemoglobin, Visit 11 (Month 36), n=115: number analyzed (Participants) | 115
  Hemoglobin, Visit 11 (Month 36), n=115 | -1.0 (10.12)
  Hemoglobin, Visit 12 (Month 40), n=109: number analyzed (Participants) | 109
  Hemoglobin, Visit 12 (Month 40), n=109 | 0.4 (9.78)
  Hemoglobin, Visit 13 (Month 44), n=98: number analyzed (Participants) | 98
  Hemoglobin, Visit 13 (Month 44), n=98 | -0.1 (9.44)
  Hemoglobin, Visit 14 (Month 48), n=101: number analyzed (Participants) | 101
  Hemoglobin, Visit 14 (Month 48), n=101 | -1.6 (9.57)
  Hemoglobin, Visit 15 (Month 52), n=88: number analyzed (Participants) | 88
  Hemoglobin, Visit 15 (Month 52), n=88 | -1.6 (9.75)
  Hemoglobin, Visit 16 (Month 56), n=76: number analyzed (Participants) | 76
  Hemoglobin, Visit 16 (Month 56), n=76 | -2.3 (7.47)
  Hemoglobin, Visit 17 (Month 60), n=89: number analyzed (Participants) | 89
  Hemoglobin, Visit 17 (Month 60), n=89 | -2.4 (10.14)
  Hemoglobin, Visit 18 (Month 64), n=54: number analyzed (Participants) | 54
  Hemoglobin, Visit 18 (Month 64), n=54 | -1.1 (8.76)
  Hemoglobin, Visit 19 (Month 68), n=50: number analyzed (Participants) | 50
  Hemoglobin, Visit 19 (Month 68), n=50 | -0.4 (9.42)
  Hemoglobin, Visit 20 (Month 72), n=55: number analyzed (Participants) | 55
  Hemoglobin, Visit 20 (Month 72), n=55 | -2.5 (10.78)
  Hemoglobin, Visit 21 (Month 76), n=40: number analyzed (Participants) | 40
  Hemoglobin, Visit 21 (Month 76), n=40 | -1.5 (11.67)
  Hemoglobin, Visit 22 (Month 80), n=35: number analyzed (Participants) | 35
  Hemoglobin, Visit 22 (Month 80), n=35 | -0.8 (9.66)
  Hemoglobin, Visit 23 (Month 84), n=32: number analyzed (Participants) | 32
  Hemoglobin, Visit 23 (Month 84), n=32 | -3.6 (11.61)
  Hemoglobin, Visit 24 (Month 88), n=27: number analyzed (Participants) | 27
  Hemoglobin, Visit 24 (Month 88), n=27 | -3.0 (9.46)
  Hemoglobin, Visit 25 (Month 92), n=25: number analyzed (Participants) | 25
  Hemoglobin, Visit 25 (Month 92), n=25 | -2.3 (8.09)
  Hemoglobin, Visit 26 (Month 96), n=24: number analyzed (Participants) | 24
  Hemoglobin, Visit 26 (Month 96), n=24 | -4.0 (8.26)
  Hemoglobin, Visit 27 (Month 100), n=20: number analyzed (Participants) | 20
  Hemoglobin, Visit 27 (Month 100), n=20 | -2.8 (5.82)
  Hemoglobin, Visit 28 (Month 104), n=16: number analyzed (Participants) | 16
  Hemoglobin, Visit 28 (Month 104), n=16 | -2.9 (9.54)
  Hemoglobin, Visit 29 (Month 108), n=13: number analyzed (Participants) | 13
  Hemoglobin, Visit 29 (Month 108), n=13 | -8.1 (8.56)
  Hemoglobin, Visit 30 (Month 112), n=4: number analyzed (Participants) | 4
  Hemoglobin, Visit 30 (Month 112), n=4 | -12.5 (6.14)
  Hemoglobin, Visit 31 (Month 116), n=3: number analyzed (Participants) | 3
  Hemoglobin, Visit 31 (Month 116), n=3 | 3.0 (22.52)
  Hemoglobin, Visit 32 (Month 120), n=1: number analyzed (Participants) | 1
  Hemoglobin, Visit 32 (Month 120), n=1 | 25.0 (NA) — Standard deviation could not be calculated as only 1 participant was analyzed.
  Hemoglobin, Follow up, n=256: number analyzed (Participants) | 256
  Hemoglobin, Follow up, n=256 | -0.1 (8.89)

16. Primary Outcome: Change From Baseline in Hematology Parameter Red Blood Cells (RBC)
Description: The hematology parameters included RBC. The clinical laboratory evaluation were performed at all study visits during the Open-Label Treatment Phase. Baseline assessment in this OLE study was defined as the last assessment of that endpoint in VRX-RET-E22-302 taken prior to the first active treatment with retigabine. Change from Baseline was calculated by subtracting the Baseline value from the post Baseline values. NA indicates standard deviation could not be calculated as only 1 participant was analyzed. Only those participants with data available at the specified time points were analyzed (represented by n=X in the category titles).
Time Frame: Baseline and up to 122 months
Population: Safety Population
Measure: Mean (Standard Deviation); unit: 10^12 cells per liter
Arm/Group | Retigabine
Number analyzed (Participants) | 376
10^12 cells per liter
  RBC, Visit 1 (Month 1), n=349: number analyzed (Participants) | 349
  RBC, Visit 1 (Month 1), n=349 | -0.07 (0.226)
  RBC, Visit 1a (Month 2), n=65: number analyzed (Participants) | 65
  RBC, Visit 1a (Month 2), n=65 | 0.00 (0.236)
  RBC, Visit 2 (Month 3), n=316: number analyzed (Participants) | 316
  RBC, Visit 2 (Month 3), n=316 | -0.02 (0.237)
  RBC, Visit 2a (Month 4), n=82: number analyzed (Participants) | 82
  RBC, Visit 2a (Month 4), n=82 | -0.06 (0.233)
  RBC, Visit 3 (Month 6), n=279: number analyzed (Participants) | 279
  RBC, Visit 3 (Month 6), n=279 | -0.04 (0.243)
  RBC, Visit 3a (Month 8), n=99: number analyzed (Participants) | 99
  RBC, Visit 3a (Month 8), n=99 | -0.05 (0.269)
  RBC, Visit 4 (Month 9), n=244: number analyzed (Participants) | 244
  RBC, Visit 4 (Month 9), n=244 | -0.03 (0.256)
  RBC, Visit 4a (Month 10), n=113: number analyzed (Participants) | 113
  RBC, Visit 4a (Month 10), n=113 | -0.02 (0.235)
  RBC, Visit 5 (Month 12), n=226: number analyzed (Participants) | 226
  RBC, Visit 5 (Month 12), n=226 | -0.04 (0.255)
  RBC, Visit 6 (Month 16), n=199: number analyzed (Participants) | 199
  RBC, Visit 6 (Month 16), n=199 | -0.01 (0.264)
  RBC, Visit 7 (Month 20), n=174: number analyzed (Participants) | 174
  RBC, Visit 7 (Month 20), n=174 | -0.02 (0.243)
  RBC, Visit 8 (Month 24), n=164: number analyzed (Participants) | 164
  RBC, Visit 8 (Month 24), n=164 | -0.03 (0.281)
  RBC, Visit 9 (Month 28), n=142: number analyzed (Participants) | 142
  RBC, Visit 9 (Month 28), n=142 | 0.00 (0.271)
  RBC, Visit 10 (Month 32), n=126: number analyzed (Participants) | 126
  RBC, Visit 10 (Month 32), n=126 | -0.05 (0.286)
  RBC, Visit 11 (Month 36), n=115: number analyzed (Participants) | 115
  RBC, Visit 11 (Month 36), n=115 | -0.09 (0.283)
  RBC, Visit 12 (Month 40), n=109: number analyzed (Participants) | 109
  RBC, Visit 12 (Month 40), n=109 | -0.02 (0.275)
  RBC, Visit 13 (Month 44), n=98: number analyzed (Participants) | 98
  RBC, Visit 13 (Month 44), n=98 | -0.06 (0.287)
  RBC, Visit 14 (Month 48), n=101: number analyzed (Participants) | 101
  RBC, Visit 14 (Month 48), n=101 | -0.10 (0.280)
  RBC, Visit 15 (Month 52), n=88: number analyzed (Participants) | 88
  RBC, Visit 15 (Month 52), n=88 | -0.08 (0.285)
  RBC, Visit 16 (Month 56), n=76: number analyzed (Participants) | 76
  RBC, Visit 16 (Month 56), n=76 | -0.08 (0.252)
  RBC, Visit 17 (Month 60), n=89: number analyzed (Participants) | 89
  RBC, Visit 17 (Month 60), n=89 | -0.07 (0.323)
  RBC, Visit 18 (Month 64), n=54: number analyzed (Participants) | 54
  RBC, Visit 18 (Month 64), n=54 | -0.01 (0.263)
  RBC, Visit 19 (Month 68), n=50: number analyzed (Participants) | 50
  RBC, Visit 19 (Month 68), n=50 | 0.01 (0.255)
  RBC, Visit 20 (Month 72), n=55: number analyzed (Participants) | 55
  RBC, Visit 20 (Month 72), n=55 | -0.03 (0.239)
  RBC, Visit 21 (Month 76), n=40: number analyzed (Participants) | 40
  RBC, Visit 21 (Month 76), n=40 | 0.02 (0.346)
  RBC, Visit 22 (Month 80), n=35: number analyzed (Participants) | 35
  RBC, Visit 22 (Month 80), n=35 | 0.09 (0.338)
  RBC, Visit 23 (Month 84), n=32: number analyzed (Participants) | 32
  RBC, Visit 23 (Month 84), n=32 | 0.00 (0.290)
  RBC, Visit 24 (Month 88), n=27: number analyzed (Participants) | 27
  RBC, Visit 24 (Month 88), n=27 | 0.00 (0.314)
  RBC, Visit 25 (Month 92), n=25: number analyzed (Participants) | 25
  RBC, Visit 25 (Month 92), n=25 | 0.05 (0.337)
  RBC, Visit 26 (Month 96), n=24: number analyzed (Participants) | 24
  RBC, Visit 26 (Month 96), n=24 | 0.06 (0.317)
  RBC, Visit 27 (Month 100), n=20: number analyzed (Participants) | 20
  RBC, Visit 27 (Month 100), n=20 | 0.13 (0.251)
  RBC, Visit 28 (Month 104), n=16: number analyzed (Participants) | 16
  RBC, Visit 28 (Month 104), n=16 | 0.14 (0.365)
  RBC, Visit 29 (Month 108), n=13: number analyzed (Participants) | 13
  RBC, Visit 29 (Month 108), n=13 | -0.04 (0.328)
  RBC, Visit 30 (Month 112), n=4: number analyzed (Participants) | 4
  RBC, Visit 30 (Month 112), n=4 | 0.08 (0.386)
  RBC, Visit 31 (Month 116), n=3: number analyzed (Participants) | 3
  RBC, Visit 31 (Month 116), n=3 | 0.10 (0.346)
  RBC, Visit 32 (Month 120), n=1: number analyzed (Participants) | 1
  RBC, Visit 32 (Month 120), n=1 | 0.00 (NA) — Standard deviation could not be calculated as only 1 participant was analyzed.
  RBC, Follow up, n=256: number analyzed (Participants) | 256
  RBC, Follow up, n=256 | -0.01 (0.263)

17. Primary Outcome: Change From Baseline in Urine Specific Gravity
Description: Urine specific gravity is a measure of the concentration of solutes in the urine. It measures the ratio of urine density compared with water density and provides information on the kidney's ability to concentrate urine. Urinalysis assessments were performed at all study visits during the Open-Label Treatment Phase. Baseline assessment in this OLE study was defined as the last assessment of that endpoint in VRX-RET-E22-302 taken prior to the first active treatment with retigabine. Change from Baseline was calculated by subtracting the Baseline value from the post Baseline values. NA indicates standard deviation could not be calculated as only 1 participant was analyzed. Only those participants with data available at the specified time points were analyzed (represented by n=X in the category titles).
Time Frame: Baseline and up to 122 months
Population: Safety Population
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | Retigabine
Number analyzed (Participants) | 376
Ratio
  Specific gravity, Visit 1 (Month 1), n=348: number analyzed (Participants) | 348
  Specific gravity, Visit 1 (Month 1), n=348 | -0.0011 (0.00936)
  Specific gravity, Visit 1a (Month 2), n=1: number analyzed (Participants) | 1
  Specific gravity, Visit 1a (Month 2), n=1 | 0.0000 (NA) — Standard deviation could not be calculated as only 1 participant was analyzed.
  Specific gravity, Visit 2 (Month 3), n=312: number analyzed (Participants) | 312
  Specific gravity, Visit 2 (Month 3), n=312 | -0.0011 (0.00918)
  Specific gravity, Visit 3 (Month 6), n=270: number analyzed (Participants) | 270
  Specific gravity, Visit 3 (Month 6), n=270 | 0.0003 (0.00896)
  Specific gravity, Visit 4 (Month 9), n=243: number analyzed (Participants) | 243
  Specific gravity, Visit 4 (Month 9), n=243 | 0.0002 (0.00984)
  Specific gravity, Visit 5 (Month 12), n=221: number analyzed (Participants) | 221
  Specific gravity, Visit 5 (Month 12), n=221 | -0.0010 (0.01014)
  Specific gravity, Visit 6 (Month 16), n=196: number analyzed (Participants) | 196
  Specific gravity, Visit 6 (Month 16), n=196 | 0.0006 (0.01016)
  Specific gravity, Visit 7 (Month 20), n=170: number analyzed (Participants) | 170
  Specific gravity, Visit 7 (Month 20), n=170 | 0.0015 (0.00901)
  Specific gravity, Visit 8 (Month 24), n=157: number analyzed (Participants) | 157
  Specific gravity, Visit 8 (Month 24), n=157 | 0.0002 (0.01015)
  Specific gravity, Visit 9 (Month 28), n=137: number analyzed (Participants) | 137
  Specific gravity, Visit 9 (Month 28), n=137 | 0.0007 (0.00922)
  Specific gravity, Visit 10 (Month 32), n=124: number analyzed (Participants) | 124
  Specific gravity, Visit 10 (Month 32), n=124 | 0.0001 (0.00986)
  Specific gravity, Visit 11 (Month 36), n=111: number analyzed (Participants) | 111
  Specific gravity, Visit 11 (Month 36), n=111 | -0.0016 (0.01058)
  Specific gravity, Visit 12 (Month 40), n=106: number analyzed (Participants) | 106
  Specific gravity, Visit 12 (Month 40), n=106 | 0.0004 (0.01007)
  Specific gravity, Visit 13 (Month 44), n=97: number analyzed (Participants) | 97
  Specific gravity, Visit 13 (Month 44), n=97 | 0.0004 (0.00944)
  Specific gravity, Visit 14 (Month 48), n=99: number analyzed (Participants) | 99
  Specific gravity, Visit 14 (Month 48), n=99 | 0.0000 (0.01019)
  Specific gravity, Visit 15 (Month 52), n=83: number analyzed (Participants) | 83
  Specific gravity, Visit 15 (Month 52), n=83 | -0.0100 (0.10022)
  Specific gravity, Visit 16 (Month 56), n=71: number analyzed (Participants) | 71
  Specific gravity, Visit 16 (Month 56), n=71 | 0.0003 (0.01089)
  Specific gravity, Visit 17 (Month 60), n=84: number analyzed (Participants) | 84
  Specific gravity, Visit 17 (Month 60), n=84 | -0.0008 (0.01022)
  Specific gravity, Visit 18 (Month 64), n=53: number analyzed (Participants) | 53
  Specific gravity, Visit 18 (Month 64), n=53 | 0.0006 (0.00894)
  Specific gravity, Visit 19 (Month 68), n=50: number analyzed (Participants) | 50
  Specific gravity, Visit 19 (Month 68), n=50 | 0.0014 (0.01052)
  Specific gravity, Visit 20 (Month 72), n=55: number analyzed (Participants) | 55
  Specific gravity, Visit 20 (Month 72), n=55 | -0.0021 (0.00882)
  Specific gravity, Visit 21 (Month 76), n=39: number analyzed (Participants) | 39
  Specific gravity, Visit 21 (Month 76), n=39 | 0.0030 (0.00837)
  Specific gravity, Visit 22 (Month 80), n=35: number analyzed (Participants) | 35
  Specific gravity, Visit 22 (Month 80), n=35 | 0.0015 (0.00939)
  Specific gravity, Visit 23 (Month 84), n=31: number analyzed (Participants) | 31
  Specific gravity, Visit 23 (Month 84), n=31 | 0.0024 (0.00917)
  Specific gravity, Visit 24 (Month 88), n=28: number analyzed (Participants) | 28
  Specific gravity, Visit 24 (Month 88), n=28 | 0.0043 (0.00994)
  Specific gravity, Visit 25 (Month 92), n=25: number analyzed (Participants) | 25
  Specific gravity, Visit 25 (Month 92), n=25 | 0.0046 (0.00861)
  Specific gravity, Visit 26 (Month 96), n=26: number analyzed (Participants) | 26
  Specific gravity, Visit 26 (Month 96), n=26 | 0.0035 (0.00857)
  Specific gravity, Visit 27 (Month 100), n=20: number analyzed (Participants) | 20
  Specific gravity, Visit 27 (Month 100), n=20 | 0.0029 (0.00718)
  Specific gravity, Visit 28 (Month 104), n=16: number analyzed (Participants) | 16
  Specific gravity, Visit 28 (Month 104), n=16 | 0.0026 (0.00713)
  Specific gravity, Visit 29 (Month 108), n=13: number analyzed (Participants) | 13
  Specific gravity, Visit 29 (Month 108), n=13 | 0.0020 (0.00709)
  Specific gravity, Visit 30 (Month 112), n=4: number analyzed (Participants) | 4
  Specific gravity, Visit 30 (Month 112), n=4 | 0.0020 (0.00673)
  Specific gravity, Visit 31 (Month 116), n=3: number analyzed (Participants) | 3
  Specific gravity, Visit 31 (Month 116), n=3 | 0.0030 (0.01082)
  Specific gravity, Visit 32 (Month 120), n=1: number analyzed (Participants) | 1
  Specific gravity, Visit 32 (Month 120), n=1 | -0.0010 (NA) — Standard deviation could not be calculated as only 1 participant was analyzed.
  Specific gravity, Follow up, n=247: number analyzed (Participants) | 247
  Specific gravity, Follow up, n=247 | 0.0008 (0.00889)

18. Primary Outcome: Change From Baseline in Urine Potential of Hydrogen (pH)
Description: Urinalysis parameters included urine pH. pH is calculated on a scale of 0 to 14, such that, the lower the number, more acidic the urine and higher the number, more alkaline the urine with 7 being neutral. Urinalysis assessments were performed at all study visits during the Open-Label Treatment Phase. Baseline assessment in this OLE study was defined as the last assessment of that endpoint in VRX-RET-E22-302 taken prior to the first active treatment with retigabine. Change from Baseline was calculated by subtracting the Baseline value from the post Baseline values. NA indicates standard deviation could not be calculated as only 1 participant was analyzed. Only those participants with data available at the specified time points were analyzed (represented by n=X in the category titles).
Time Frame: Baseline and up to 122 months
Population: Safety Population
Measure: Mean (Standard Deviation); unit: Points on a scale
Arm/Group | Retigabine
Number analyzed (Participants) | 376
Points on a scale
  pH, Visit 1 (Month 1), n=349: number analyzed (Participants) | 349
  pH, Visit 1 (Month 1), n=349 | -0.13 (0.685)
  pH, Visit 1a (Month 2), n=1: number analyzed (Participants) | 1
  pH, Visit 1a (Month 2), n=1 | 0.50 (NA) — Standard deviation could not be calculated as only 1 participant was analyzed.
  pH, Visit 2 (Month 3), n=313: number analyzed (Participants) | 313
  pH, Visit 2 (Month 3), n=313 | -0.09 (0.699)
  pH, Visit 3 (Month 6), n=270: number analyzed (Participants) | 270
  pH, Visit 3 (Month 6), n=270 | -0.07 (0.634)
  pH, Visit 4 (Month 9), n=245: number analyzed (Participants) | 245
  pH, Visit 4 (Month 9), n=245 | 0.02 (0.633)
  pH, Visit 5 (Month 12), n=222: number analyzed (Participants) | 222
  pH, Visit 5 (Month 12), n=222 | -0.02 (0.616)
  pH, Visit 6 (Month 16), n=196: number analyzed (Participants) | 196
  pH, Visit 6 (Month 16), n=196 | 0.07 (0.651)
  pH, Visit 7 (Month 20), n=170: number analyzed (Participants) | 170
  pH, Visit 7 (Month 20), n=170 | 0.04 (0.686)
  pH, Visit 8 (Month 24), n=158: number analyzed (Participants) | 158
  pH, Visit 8 (Month 24), n=158 | 0.09 (0.672)
  pH, Visit 9 (Month 28), n=138: number analyzed (Participants) | 138
  pH, Visit 9 (Month 28), n=138 | 0.17 (0.787)
  pH, Visit 10 (Month 32), n=124: number analyzed (Participants) | 124
  pH, Visit 10 (Month 32), n=124 | 0.17 (0.715)
  pH, Visit 11 (Month 36), n=111: number analyzed (Participants) | 111
  pH, Visit 11 (Month 36), n=111 | 0.26 (0.663)
  pH, Visit 12 (Month 40), n=107: number analyzed (Participants) | 107
  pH, Visit 12 (Month 40), n=107 | 0.30 (0.700)
  pH, Visit 13 (Month 44), n=97: number analyzed (Participants) | 97
  pH, Visit 13 (Month 44), n=97 | 0.36 (0.736)
  pH, Visit 14 (Month 48), n=99: number analyzed (Participants) | 99
  pH, Visit 14 (Month 48), n=99 | 0.38 (0.722)
  pH, Visit 15 (Month 52), n=83: number analyzed (Participants) | 83
  pH, Visit 15 (Month 52), n=83 | 0.27 (0.621)
  pH, Visit 16 (Month 56), n=71: number analyzed (Participants) | 71
  pH, Visit 16 (Month 56), n=71 | 0.34 (0.840)
  pH, Visit 17 (Month 60), n=84: number analyzed (Participants) | 84
  pH, Visit 17 (Month 60), n=84 | 0.32 (0.662)
  pH, Visit 18 (Month 64), n=53: number analyzed (Participants) | 53
  pH, Visit 18 (Month 64), n=53 | 0.33 (0.627)
  pH, Visit 19 (Month 68), n=50: number analyzed (Participants) | 50
  pH, Visit 19 (Month 68), n=50 | 0.42 (0.785)
  pH, Visit 20 (Month 72), n=55: number analyzed (Participants) | 55
  pH, Visit 20 (Month 72), n=55 | 0.27 (0.686)
  pH, Visit 21 (Month 76), n=39: number analyzed (Participants) | 39
  pH, Visit 21 (Month 76), n=39 | 0.36 (0.688)
  pH, Visit 22 (Month 80), n=35: number analyzed (Participants) | 35
  pH, Visit 22 (Month 80), n=35 | 0.23 (0.657)
  pH, Visit 23 (Month 84), n=31: number analyzed (Participants) | 31
  pH, Visit 23 (Month 84), n=31 | 0.35 (0.661)
  pH, Visit 24 (Month 88), n=28: number analyzed (Participants) | 28
  pH, Visit 24 (Month 88), n=28 | 0.29 (0.517)
  pH, Visit 25 (Month 92), n=25: number analyzed (Participants) | 25
  pH, Visit 25 (Month 92), n=25 | 0.36 (0.621)
  pH, Visit 26 (Month 96), n=26: number analyzed (Participants) | 26
  pH, Visit 26 (Month 96), n=26 | 0.21 (0.551)
  pH, Visit 27 (Month 100), n=20: number analyzed (Participants) | 20
  pH, Visit 27 (Month 100), n=20 | 0.45 (0.724)
  pH, Visit 28 (Month 104), n=16: number analyzed (Participants) | 16
  pH, Visit 28 (Month 104), n=16 | 0.13 (0.342)
  pH, Visit 29 (Month 108), n=13: number analyzed (Participants) | 13
  pH, Visit 29 (Month 108), n=13 | 0.77 (0.753)
  pH, Visit 30 (Month 112), n=4: number analyzed (Participants) | 4
  pH, Visit 30 (Month 112), n=4 | 0.50 (0.577)
  pH, Visit 31 (Month 116), n=3: number analyzed (Participants) | 3
  pH, Visit 31 (Month 116), n=3 | -0.17 (0.764)
  pH, Visit 32 (Month 120), n=1: number analyzed (Participants) | 1
  pH, Visit 32 (Month 120), n=1 | 0.00 (NA) — Standard deviation could not be calculated as only 1 participant was analyzed.
  pH, Follow up, n=248: number analyzed (Participants) | 248
  pH, Follow up, n=248 | 0.22 (0.746)

19. Primary Outcome: Change From Baseline in Post-Void Residual (PVR) Bladder Ultrasound Volume
Description: The post-void residual urine volume in the bladder was evaluated by transabdominal ultrasound. The urine bladder was sonicated from two directions perpendicular to one another, and the volume calculated automatically. A PVR bladder ultrasound to assess urinary retention was performed during the first year at Months 1, 3 and 12 and at the end of each 12 month study cycle that the participant was enrolled (i.e., second year, third year, fourth year, etc.) in the Open-Label Treatment Phase of the study. Baseline assessment in this OLE study was defined as the last assessment of that endpoint in VRX-RET-E22-302 taken prior to the first active treatment with retigabine. Change from Baseline was calculated by subtracting the Baseline value from the post Baseline values. Only those participants with data available at the specified time points were analyzed (represented by n=X in the category titles).
Time Frame: Baseline and up to 122 months
Population: Safety Population
Measure: Mean (Standard Deviation); unit: Milliliters
Arm/Group | Retigabine
Number analyzed (Participants) | 376
Milliliters
  PVR urine volume, Visit 1 (Month 1), n=337: number analyzed (Participants) | 337
  PVR urine volume, Visit 1 (Month 1), n=337 | 4.6 (52.10)
  PVR urine volume, Visit 2 (Month 3), n=307: number analyzed (Participants) | 307
  PVR urine volume, Visit 2 (Month 3), n=307 | 4.1 (40.88)
  PVR urine volume, Visit 5 (Month 12), n=223: number analyzed (Participants) | 223
  PVR urine volume, Visit 5 (Month 12), n=223 | 4.1 (52.38)
  PVR urine volume, Visit 8 (Month 24), n=111: number analyzed (Participants) | 111
  PVR urine volume, Visit 8 (Month 24), n=111 | 5.5 (67.28)
  PVR urine volume, Visit 11 (Month 36), n=106: number analyzed (Participants) | 106
  PVR urine volume, Visit 11 (Month 36), n=106 | 5.0 (46.29)
  PVR urine volume, Visit 14 (Month 48), n=96: number analyzed (Participants) | 96
  PVR urine volume, Visit 14 (Month 48), n=96 | -2.3 (39.69)
  PVR urine volume, Visit 17 (Month 60), n=77: number analyzed (Participants) | 77
  PVR urine volume, Visit 17 (Month 60), n=77 | 22.2 (87.43)
  PVR urine volume, Visit 20 (Month 72), n=53: number analyzed (Participants) | 53
  PVR urine volume, Visit 20 (Month 72), n=53 | 7.1 (49.87)
  PVR urine volume, Visit 23 (Month 84), n=29: number analyzed (Participants) | 29
  PVR urine volume, Visit 23 (Month 84), n=29 | 15.7 (74.06)
  PVR urine volume, Visit 26 (Month 96), n=24: number analyzed (Participants) | 24
  PVR urine volume, Visit 26 (Month 96), n=24 | 2.0 (38.54)
  PVR urine volume, Visit 29 (Month 108), n=10: number analyzed (Participants) | 10
  PVR urine volume, Visit 29 (Month 108), n=10 | 21.9 (63.58)
  PVR urine volume, Visit 32 (Month 120), n=0: number analyzed (Participants) | 0
  PVR urine volume, Follow up, n=186: number analyzed (Participants) | 186
  PVR urine volume, Follow up, n=186 | -4.0 (47.11)

20. Primary Outcome: Change From Baseline in the Urinary Voiding Function [UVF] (Assessed Using the American Urological Association [AUA] Symptom Index)
Description: AUA Symptom Index was completed during the first year at Months 1, 3, 12 and at the end of each 12 month study cycle that the participant was enrolled in the Open-Label Treatment Phase (second, third, fourth year) to assess the participant UVF. The questions were scored on a scale of 0 to 5, with 0 (not at all) to 5 (almost always). A Symptom Index is determined by adding the scores. The lowest possible score is 0 and the highest possible score is 35, which would represent the highest level of pain and discomfort. Baseline assessment in this OLE study was defined as the last assessment of that endpoint in VRX-RET-E22-302 taken prior to the first active treatment with retigabine. Change from Baseline was calculated by subtracting the Baseline value from the post Baseline values. NA indicates standard deviation could not be calculated as only 1 participant was analyzed. Only those participants with data available at the specified time points were analyzed represented by (n=x).
Time Frame: Baseline and up to 122 months
Population: Safety Population
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Retigabine
Number analyzed (Participants) | 376
Scores on a scale
  AUA Overall Score, Visit 1 (Month 1), n=348: number analyzed (Participants) | 348
  AUA Overall Score, Visit 1 (Month 1), n=348 | -0.4 (3.82)
  AUA Overall Score, Visit 2 (Month 3), n=325: number analyzed (Participants) | 325
  AUA Overall Score, Visit 2 (Month 3), n=325 | -0.5 (3.80)
  AUA Overall Score, Visit 5 (Month 12), n=228: number analyzed (Participants) | 228
  AUA Overall Score, Visit 5 (Month 12), n=228 | -0.5 (3.58)
  AUA Overall Score, Visit 8 (Month 24), n=114: number analyzed (Participants) | 114
  AUA Overall Score, Visit 8 (Month 24), n=114 | -0.5 (3.84)
  AUA Overall Score, Visit 11 (Month 36), n=115: number analyzed (Participants) | 115
  AUA Overall Score, Visit 11 (Month 36), n=115 | -0.3 (5.22)
  AUA Overall Score, Visit 14 (Month 48), n=102: number analyzed (Participants) | 102
  AUA Overall Score, Visit 14 (Month 48), n=102 | -0.6 (4.89)
  AUA Overall Score, Visit 17 (Month 60), n=87: number analyzed (Participants) | 87
  AUA Overall Score, Visit 17 (Month 60), n=87 | -0.4 (5.02)
  AUA Overall Score, Visit 20 (Month 72), n=56: number analyzed (Participants) | 56
  AUA Overall Score, Visit 20 (Month 72), n=56 | -0.1 (5.52)
  AUA Overall Score, Visit 23 (Month 84), n=32: number analyzed (Participants) | 32
  AUA Overall Score, Visit 23 (Month 84), n=32 | 0.8 (6.61)
  AUA Overall Score, Visit 26 (Month 96), n=26: number analyzed (Participants) | 26
  AUA Overall Score, Visit 26 (Month 96), n=26 | 0.5 (5.58)
  AUA Overall Score, Visit 29 (Month 108), n=13: number analyzed (Participants) | 13
  AUA Overall Score, Visit 29 (Month 108), n=13 | 0.0 (1.68)
  AUA Overall Score, Visit 32 (Month 120), n=1: number analyzed (Participants) | 1
  AUA Overall Score, Visit 32 (Month 120), n=1 | 0.0 (NA) — Standard deviation could not be calculated as only 1 participant was analyzed.
  AUA Overall Score, Follow up, n=217: number analyzed (Participants) | 217
  AUA Overall Score, Follow up, n=217 | 0.0 (4.43)

21. Primary Outcome: Change From Baseline in Quality of Life in Epilepsy-31-Problems (QOLIE-31-P) Questionnaire
Description: The QOLIE-31-P questionnaire contained 30 items. The subscale scores (seizure worry, overall QOL, emotional well-being, energy-fatigue, cognitive, medication effects, social functioning), the final QOLIE-31-P score and the weighted total score (overall assessment) were calculated according to the scoring algorithm defined by the author. Scores range from 0 to 100 with higher scores indicating better function. Baseline was defined as the last assessment of that endpoint in VRX-RET-E22-302 taken prior to the first active treatment with retigabine. Change from Baseline was calculated by subtracting the Baseline value from the post Baseline values. NA indicates standard deviation could not be calculated as only 1 participant was analyzed. Only those participants with data available at the specified time points were analyzed (represented by n=X in the category titles).
Time Frame: Baseline and up to 122 months
Population: Safety Population
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Retigabine
Number analyzed (Participants) | 376
Scores on a scale
  Final QOLIE-31-P Score, Visit 2 (Month 3), n=296: number analyzed (Participants) | 296
  Final QOLIE-31-P Score, Visit 2 (Month 3), n=296 | 1.33 (14.409)
  Final QOLIE-31-P Score, Visit 3 (Month 6), n=262: number analyzed (Participants) | 262
  Final QOLIE-31-P Score, Visit 3 (Month 6), n=262 | 0.87 (14.618)
  Final QOLIE-31-P Score, Visit 4 (Month 9), n=229: number analyzed (Participants) | 229
  Final QOLIE-31-P Score, Visit 4 (Month 9), n=229 | 0.27 (14.365)
  Final QOLIE-31-P Score, Visit 5 (Month 12), n=214: number analyzed (Participants) | 214
  Final QOLIE-31-P Score, Visit 5 (Month 12), n=214 | 1.24 (14.498)
  Final QOLIE-31-P Score, Visit 8 (Month 24), n=142: number analyzed (Participants) | 142
  Final QOLIE-31-P Score, Visit 8 (Month 24), n=142 | 3.76 (12.406)
  Final QOLIE-31-P Score, Visit 11 (Month 36), n=97: number analyzed (Participants) | 97
  Final QOLIE-31-P Score, Visit 11 (Month 36), n=97 | 2.77 (13.784)
  Final QOLIE-31-P Score, Visit 14 (Month 48), n=83: number analyzed (Participants) | 83
  Final QOLIE-31-P Score, Visit 14 (Month 48), n=83 | 0.78 (13.976)
  Final QOLIE-31-P Score Visit 17 (Month 60), n=68: number analyzed (Participants) | 68
  Final QOLIE-31-P Score Visit 17 (Month 60), n=68 | 2.37 (15.197)
  Final QOLIE-31-P Score Visit 20 (Month 72), n=47: number analyzed (Participants) | 47
  Final QOLIE-31-P Score Visit 20 (Month 72), n=47 | 3.07 (16.172)
  Final QOLIE-31-P Score Visit 23 (Month 84), n=26: number analyzed (Participants) | 26
  Final QOLIE-31-P Score Visit 23 (Month 84), n=26 | 4.31 (13.849)
  Final QOLIE-31-P Score Visit 26 (Month 96), n=24: number analyzed (Participants) | 24
  Final QOLIE-31-P Score Visit 26 (Month 96), n=24 | 4.07 (11.745)
  Final QOLIE-31-P Score Visit 29 (Month 108), n=12: number analyzed (Participants) | 12
  Final QOLIE-31-P Score Visit 29 (Month 108), n=12 | 6.35 (14.783)
  Final QOLIE-31-P Score Visit 32 (Month 120), n=1: number analyzed (Participants) | 1
  Final QOLIE-31-P Score Visit 32 (Month 120), n=1 | 14.36 (NA) — Standard deviation could not be calculated as only 1 participant was analyzed.
  Final QOLIE-31-P Score, Follow up, n=224: number analyzed (Participants) | 224
  Final QOLIE-31-P Score, Follow up, n=224 | -0.83 (14.256)

22. Primary Outcome: Percentage of Participants With Abnormal Results of Physical Examination
Description: A complete physical examination was performed at the end of each 12 month study cycle (i.e., first year, second year, third year, etc.) during the Open-Label Treatment Phase. The investigator assessed the skin at every clinic visit. If abnormal skin discoloration was confirmed, the participant continued to be followed by the dermatologist. If the abnormal skin discoloration was not confirmed, the investigator resumed assessing the participants skin at all scheduled clinic visits. Only data for abnormal values on physical examination have been presented. Only those participants available at the specified time points were analyzed.
Time Frame: Baseline and up to 122 months
Population: Safety Population
Measure: Number; unit: Percentage of participants
Arm/Group | Retigabine
Number analyzed (Participants) | 376
Percentage of participants
  Visit 5 (Month 12), n=234: number analyzed (Participants) | 234
  Visit 5 (Month 12), n=234 | 18
  Visit 8 (Month 24), n=166: number analyzed (Participants) | 166
  Visit 8 (Month 24), n=166 | 17
  Visit 11 (Month 36), n=121: number analyzed (Participants) | 121
  Visit 11 (Month 36), n=121 | 21
  Visit 14 (Month 48), n=104: number analyzed (Participants) | 104
  Visit 14 (Month 48), n=104 | 19
  Visit 17 (Month 60), n=88: number analyzed (Participants) | 88
  Visit 17 (Month 60), n=88 | 19
  Visit 20 (Month 72), n=58: number analyzed (Participants) | 58
  Visit 20 (Month 72), n=58 | 24
  Visit 23 (Month 84), n=32: number analyzed (Participants) | 32
  Visit 23 (Month 84), n=32 | 34
  Visit 26 (Month 96), n=26: number analyzed (Participants) | 26
  Visit 26 (Month 96), n=26 | 35
  Visit 29 (Month 108), n=13: number analyzed (Participants) | 13
  Visit 29 (Month 108), n=13 | 38
  Follow up visit, n=260: number analyzed (Participants) | 260
  Follow up visit, n=260 | 27

23. Primary Outcome: Percentage of Participants With Abnormal Results of Neurological Examination
Description: A complete neurological examination was performed at the end of each 12 month study cycle (i.e., first year, second year, third year, etc.) during the Open-Label Treatment Phase. Abnormal results were categorized as Abnormal-Not Clinically Significant (A-NCS) and Abnormal and Clinically Significant (A-CS). Only data for abnormal values on neurological examination have been presented. Only those participants available at the specified time points were analyzed.
Time Frame: Baseline and up to 122 months
Population: Safety Population
Measure: Number; unit: Percentage of participants
Arm/Group | Retigabine
Number analyzed (Participants) | 376
Percentage of participants
  Visit 1 (Month 1), A-NCS, n=356: number analyzed (Participants) | 356
  Visit 1 (Month 1), A-NCS, n=356 | 23
  Visit 1 (Month 1), A-CS, n=356: number analyzed (Participants) | 356
  Visit 1 (Month 1), A-CS, n=356 | 10
  Visit 2 (Month 3), A-NCS, n=328: number analyzed (Participants) | 328
  Visit 2 (Month 3), A-NCS, n=328 | 23
  Visit 2 (Month 3), A-CS, n=328: number analyzed (Participants) | 328
  Visit 2 (Month 3), A-CS, n=328 | 9
  Visit 3 (Month 6), A-NCS, n=287: number analyzed (Participants) | 287
  Visit 3 (Month 6), A-NCS, n=287 | 22
  Visit 3 (Month 6), A-CS, n=287: number analyzed (Participants) | 287
  Visit 3 (Month 6), A-CS, n=287 | 10
  Visit 4 (Month 9), A-NCS, n=252: number analyzed (Participants) | 252
  Visit 4 (Month 9), A-NCS, n=252 | 23
  Visit 4 (Month 9), A-CS, n=252: number analyzed (Participants) | 252
  Visit 4 (Month 9), A-CS, n=252 | 11
  Visit 5 (Month 12), A-NCS, n=234: number analyzed (Participants) | 234
  Visit 5 (Month 12), A-NCS, n=234 | 27
  Visit 5 (Month 12), A-CS, n=234: number analyzed (Participants) | 234
  Visit 5 (Month 12), A-CS, n=234 | 12
  Visit 6 (Month 16), A-NCS, n=202: number analyzed (Participants) | 202
  Visit 6 (Month 16), A-NCS, n=202 | 24
  Visit 6 (Month 16), A-CS, n=202: number analyzed (Participants) | 202
  Visit 6 (Month 16), A-CS, n=202 | 9
  Visit 7 (Month 20), A-NCS, n=179: number analyzed (Participants) | 179
  Visit 7 (Month 20), A-NCS, n=179 | 25
  Visit 7 (Month 20), A-CS, n=179: number analyzed (Participants) | 179
  Visit 7 (Month 20), A-CS, n=179 | 9
  Visit 8 (Month 24), A-NCS, n=166: number analyzed (Participants) | 166
  Visit 8 (Month 24), A-NCS, n=166 | 34
  Visit 8 (Month 24), A-CS, n=166: number analyzed (Participants) | 166
  Visit 8 (Month 24), A-CS, n=166 | 10
  Visit 9 (Month 28), A-NCS, n=146: number analyzed (Participants) | 146
  Visit 9 (Month 28), A-NCS, n=146 | 32
  Visit 9 (Month 28), A-CS, n=146: number analyzed (Participants) | 146
  Visit 9 (Month 28), A-CS, n=146 | 8
  Visit 10 (Month 32), A-NCS, n=127: number analyzed (Participants) | 127
  Visit 10 (Month 32), A-NCS, n=127 | 32
  Visit 10 (Month 32), A-CS, n=127: number analyzed (Participants) | 127
  Visit 10 (Month 32), A-CS, n=127 | 8
  Visit 11 (Month 36), A-NCS, n=121: number analyzed (Participants) | 121
  Visit 11 (Month 36), A-NCS, n=121 | 35
  Visit 11 (Month 36), A-CS, n=121: number analyzed (Participants) | 121
  Visit 11 (Month 36), A-CS, n=121 | 8
  Visit 12 (Month 40), A-NCS, n=112: number analyzed (Participants) | 112
  Visit 12 (Month 40), A-NCS, n=112 | 28
  Visit 12 (Month 40), A-CS, n=112: number analyzed (Participants) | 112
  Visit 12 (Month 40), A-CS, n=112 | 10
  Visit 13 (Month 44), A-NCS, n=105: number analyzed (Participants) | 105
  Visit 13 (Month 44), A-NCS, n=105 | 31
  Visit 13 (Month 44), A-CS, n=105: number analyzed (Participants) | 105
  Visit 13 (Month 44), A-CS, n=105 | 9
  Visit 14 (Month 48), A-NCS, n=104: number analyzed (Participants) | 104
  Visit 14 (Month 48), A-NCS, n=104 | 28
  Visit 14 (Month 48), A-CS, n=104: number analyzed (Participants) | 104
  Visit 14 (Month 48), A-CS, n=104 | 11
  Visit 15 (Month 52), A-NCS, n=91: number analyzed (Participants) | 91
  Visit 15 (Month 52), A-NCS, n=91 | 31
  Visit 15 (Month 52), A-CS, n=91: number analyzed (Participants) | 91
  Visit 15 (Month 52), A-CS, n=91 | 9
  Visit 16 (Month 56), A-NCS, n=77: number analyzed (Participants) | 77
  Visit 16 (Month 56), A-NCS, n=77 | 32
  Visit 16 (Month 56), A-CS, n=77: number analyzed (Participants) | 77
  Visit 16 (Month 56), A-CS, n=77 | 9
  Visit 17 (Month 60), A-NCS, n=89: number analyzed (Participants) | 89
  Visit 17 (Month 60), A-NCS, n=89 | 29
  Visit 17 (Month 60), A-CS, n=89: number analyzed (Participants) | 89
  Visit 17 (Month 60), A-CS, n=89 | 9
  Visit 18 (Month 64), A-NCS, n=58: number analyzed (Participants) | 58
  Visit 18 (Month 64), A-NCS, n=58 | 29
  Visit 18 (Month 64), A-CS, n=58: number analyzed (Participants) | 58
  Visit 18 (Month 64), A-CS, n=58 | 10
  Visit 19 (Month 68), A-NCS, n=53: number analyzed (Participants) | 53
  Visit 19 (Month 68), A-NCS, n=53 | 36
  Visit 19 (Month 68), A-CS, n=53: number analyzed (Participants) | 53
  Visit 19 (Month 68), A-CS, n=53 | 9
  Visit 20 (Month 72), A-NCS, n=59: number analyzed (Participants) | 59
  Visit 20 (Month 72), A-NCS, n=59 | 41
  Visit 20 (Month 72), A-CS, n=59: number analyzed (Participants) | 59
  Visit 20 (Month 72), A-CS, n=59 | 7
  Visit 21 (Month 76), A-NCS, n=43: number analyzed (Participants) | 43
  Visit 21 (Month 76), A-NCS, n=43 | 40
  Visit 21 (Month 76), A-CS, n=43: number analyzed (Participants) | 43
  Visit 21 (Month 76), A-CS, n=43 | 7
  Visit 22 (Month 80), A-NCS, n=37: number analyzed (Participants) | 37
  Visit 22 (Month 80), A-NCS, n=37 | 41
  Visit 22 (Month 80), A-CS, n=37: number analyzed (Participants) | 37
  Visit 22 (Month 80), A-CS, n=37 | 5
  Visit 23 (Month 84), A-NCS, n=32: number analyzed (Participants) | 32
  Visit 23 (Month 84), A-NCS, n=32 | 47
  Visit 23 (Month 84), A-CS, n=32: number analyzed (Participants) | 32
  Visit 23 (Month 84), A-CS, n=32 | 3
  Visit 24 (Month 88), A-NCS, n=29: number analyzed (Participants) | 29
  Visit 24 (Month 88), A-NCS, n=29 | 45
  Visit 24 (Month 88), A-CS, n=29: number analyzed (Participants) | 29
  Visit 24 (Month 88), A-CS, n=29 | 7
  Visit 25 (Month 92), A-NCS, n=25: number analyzed (Participants) | 25
  Visit 25 (Month 92), A-NCS, n=25 | 40
  Visit 25 (Month 92), A-CS, n=25: number analyzed (Participants) | 25
  Visit 25 (Month 92), A-CS, n=25 | 8
  Visit 26 (Month 96), A-NCS, n=26: number analyzed (Participants) | 26
  Visit 26 (Month 96), A-NCS, n=26 | 42
  Visit 26 (Month 96), A-CS, n=26: number analyzed (Participants) | 26
  Visit 26 (Month 96), A-CS, n=26 | 15
  Visit 27 (Month 100), A-NCS, n=19: number analyzed (Participants) | 19
  Visit 27 (Month 100), A-NCS, n=19 | 21
  Visit 27 (Month 100), A-CS, n=19: number analyzed (Participants) | 19
  Visit 27 (Month 100), A-CS, n=19 | 16
  Visit 28 (Month 104), A-NCS, n=17: number analyzed (Participants) | 17
  Visit 28 (Month 104), A-NCS, n=17 | 24
  Visit 28 (Month 104), A-CS, n=17: number analyzed (Participants) | 17
  Visit 28 (Month 104), A-CS, n=17 | 24
  Visit 29 (Month 108), A-NCS, n=13: number analyzed (Participants) | 13
  Visit 29 (Month 108), A-NCS, n=13 | 31
  Visit 29 (Month 108), A-CS, n=13: number analyzed (Participants) | 13
  Visit 29 (Month 108), A-CS, n=13 | 8
  Follow up visit, A-NCS, n=263: number analyzed (Participants) | 263
  Follow up visit, A-NCS, n=263 | 22
  Follow up visit, A-CS, n=263: number analyzed (Participants) | 263
  Follow up visit, A-CS, n=263 | 8

24. Secondary Outcome: Percentage of Participants With Retinal Pigmentary Abnormalities (RPA)
Description: RPA was determined by either an ophthalmologist or retina specialist. RPA is the composite endpoint assessed by its components: pigmentary abnormalities (PA) in the macula, PA in the peripheral retina (PR), PA in both macula and PR and PA at location unspecified. Only those participants with >=1 ophthalmology exam on or before last dose of retigabine are presented..
Time Frame: Up to 121 months
Population: Safety Population
Measure: Number; unit: Percentage of participants
Arm/Group | Retigabine
Number analyzed (Participants) | 54
Percentage of participants
  RPA | 31
  PA in the macula | 22
  PA of the PR | 22
  PA in both the macula and PR | 13
  PA: location unspecified | 2

25. Secondary Outcome: Percentage of Participants With Pigmentation of Non-retinal Ocular Tissue (Non-ret. Pig. Abn)
Description: Non-retinal ocular tissue abnormalities were determined by either an ophthalmologist or retina specialist. Non-ret. Pig. Abn is a composite endpoint assessed by its components: abnormal pigmentation (ABP) of the sclera and/or conjunctiva, ABP of the cornea, ABP of the iris and ABP of the lens. Only those participants with >=1 ophthalmology exam on or before last dose of retigabine are presented.
Time Frame: Up to 121 months
Population: Safety Population
Measure: Number; unit: Percentage of participants
Arm/Group | Retigabine
Number analyzed (Participants) | 54
Percentage of participants
  Non-ret. Pig. Abn | 28
  ABP of sclera and/or conjunctiva | 13
  ABP of the cornea | 4
  ABP of the iris | 17
  ABP of the lens | 0

26. Secondary Outcome: Percentage of Participants With Abnormal Pigmentation of Skin, Including the Skin Around the Eyes and the Eyelids, Lips, Nails, or Mucosa
Description: Abnormal discoloration of the skin was determined by a dermatologist. The parameters assessed were abnormal discoloration of the skin, abnormal discoloration of the lips, abnormal discoloration of the nails, abnormal discoloration of the mucosa, abnormal discoloration of sun-exposed tissue, abnormal discoloration of non sun-exposed tissue. Only those participants with at least one skin exam by the investigator or dermatologist on or before the last dose of retigabine or dermatologist-confirmed discoloration with start date on or before the date of last dose of retigabine are presented.
Time Frame: Up to 121 months
Population: Safety Population
Measure: Number; unit: Percentage of participants
Arm/Group | Retigabine
Number analyzed (Participants) | 46
Percentage of participants
  Any abnormal dermatologic discoloration | 50
  Abnormal discoloration of skin | 37
  Abnormal discoloration of lips | 26
  Abnormal discoloration of nails | 41
  Abnormal discoloration of mucosa | 30
  Abnormal discoloration of sun-exposed tissue | 48
  Abnormal discoloration of non sun-exposed tissue | 37

27. Secondary Outcome: Percentage of Participants With a Clinically Significant Decrease (CSD) in Visual Acuity (VA) From Initial Examination
Description: VA refers to the clarity of vision. The parameters assessed were CSD in VA from initial examination which can be explained and CSD in VA from initial examination which cannot be explained. Only those participants with both initial and at least 1 follow-up exam while on retigabine are presented.
Time Frame: Up to 121 months
Population: Safety Population
Measure: Number; unit: Percentage of participants
Arm/Group | Retigabine
Number analyzed (Participants) | 38
Percentage of participants
  CSD in VA from initial examination, n=38 | 13
  CSD which can be explained (Form 2), n=34: number analyzed (Participants) | 34
  CSD which can be explained (Form 2), n=34 | 12
  CSD which can not be explained (Form 2), n=34: number analyzed (Participants) | 34
  CSD which can not be explained (Form 2), n=34 | 0

28. Secondary Outcome: Percentage of Participants With Decrease in Confrontation Visual Field From Initial Examination
Description: The parameter assessed was decrease in confrontation visual field from initial examination. Only those participants with data available at the indicated time point were analyzed. Only those participants with both initial and at least 1 follow-up exam while on retigabine are presented.
Time Frame: Up to 121 months
Population: Safety Population
Measure: Number; unit: Percentage of participants
Arm/Group | Retigabine
Number analyzed (Participants) | 38
Percentage of participants | 13

29. Secondary Outcome: Number of Participants With Resolution of Abnormal Eye Pigmentation After Discontinuation of Retigabine
Description: The ophthalmologist/retina specialist determined the presence or absence of retinal and non-retinal ocular abnormalities. Retinal abnormalities included abnormalities in the macula and/or the peripheral retina. Only those participants available at the specified time points were analyzed.
Time Frame: 3 years and 10 months
Population: All SFUCP Subjects Population included participants with one or more finding(s) of abnormal pigmentation of the retina or unexplained vision loss, pigmentation of non-retinal ocular tissue or discoloration of skin, lips, nails or mucosa at the treatment phase withdrawal/follow-up visit and who enter the SFUCP phase.
Measure: Count of Participants; unit: Participants
Groups:
- SFUCP: Participants who withdraw from retigabine and who were found to have abnormal pigmentation of the retina or unexplained vision loss, pigmentation of non-retinal ocular tissue or discoloration of skin, lips, nails or mucosa entered the SFUCP. During the SFUCP, participants underwent 6-monthly comprehensive eye examinations and/or skin assessments by the investigator, ophthalmologist, retinal specialist or dermatologist as appropriate. Participants were followed up in the SFUCP until the dermatology/ophthalmology finding(s) either resolved or stabilized. Stabilization was defined in the protocol as no changes on two consecutive 6-monthly assessments over at least over 12 months after discontinuation of retigabine.
Arm/Group | SFUCP
Number analyzed (Participants) | 26
Participants
  Retinal pigmentary abnormality | 0
  Pigmentary abnormality of macula | 1
  Pigmentary abnormality of peripheral retina | 2
  Non-retinal ocular pigmentary abnormality | 8

30. Secondary Outcome: Number of Participants With Resolution of Dermatologist Confirmed Abnormal Discoloration After Discontinuation of Retigabine
Description: An assessment of the participant's nails, lips, skin and mucosa was completed by the investigator at the 6 monthly SFUCP study visits. The assessment of the participant's skin included assessment of the skin around the eyes and the eyelids, lips, nails, and mucosa.
Time Frame: 3 years and 10 months
Population: All SFUCP Subjects Population
Measure: Count of Participants; unit: Participants
Arm/Group | SFUCP
Number analyzed (Participants) | 26
Participants | 7

31. Secondary Outcome: Time From Discontinuation of Retigabine to Resolution of Abnormal Eye Pigmentation
Description: Retinal pigmentary abnormality was determined by either an ophthalmologist or retina specialist. Retinal pigmentary abnormality included pigmentary abnormality of macula, pigmentary abnormality of the peripheral retina and non-retinal ocular pigmentary abnormality. If a participant had pigmentary abnormality of macula and pigmentary abnormality of the peripheral retina both should be resolved in order for retinal pigmentary abnormality to be considered resolved. If a participant had non-retinal ocular pigmentary abnormality in more than location (conjunctiva, sclera, cornea, iris or lens), all should be resolved for non-retinal pigmentary abnormality to be considered resolved. Only participants with resolution of the specified pigmentation are included in this analysis.
Time Frame: 3 years and 10 months
Population: All SFUCP Subjects Population
Measure: Median (Full Range); unit: Days
Arm/Group | SFUCP
Number analyzed (Participants) | 26
Days
  Retinal Pigmentary Abnormality, n=0: number analyzed (Participants) | 0
  Pigmentary Abnormality of Macula, n=1: number analyzed (Participants) | 1
  Pigmentary Abnormality of Macula, n=1 | 233.0 [233 to 233]
  Pigmentary Abnormality of Peripheral Retina, n=2: number analyzed (Participants) | 2
  Pigmentary Abnormality of Peripheral Retina, n=2 | 307.0 [245 to 369]
  Non-Retinal Ocular Pigmentary Abnormality, n=8: number analyzed (Participants) | 8
  Non-Retinal Ocular Pigmentary Abnormality, n=8 | 312.0 [9 to 538]

32. Secondary Outcome: Time From Discontinuation of Retigabine to Resolution of All Dermatologist-Confirmed Abnormal Discoloration
Description: Assessments were at approximately 6-monthly intervals (timed relative to the participants previous dermatology assessment) until the abnormal discoloration either resolved or stabilized (as defined by no changes over 2 consecutive 6-monthly assessments performed by the dermatologist over at least 12 months after discontinuation of retigabine). The assessment of the participant's skin included assessment of the skin around the eyes and the eyelids, lips, nails, and mucosa. Only participants with resolution of the specified tissue are included in this analysis.
Time Frame: 3 years and 10 months
Population: All SFUCP Subjects Population
Measure: Median (Full Range); unit: Days
Arm/Group | SFUCP
Number analyzed (Participants) | 26
Days
  All, n=7: number analyzed (Participants) | 7
  All, n=7 | 380.0 [197 to 672]
  Skin, n=6: number analyzed (Participants) | 6
  Skin, n=6 | 382.5 [162 to 425]
  Lips, n=5: number analyzed (Participants) | 5
  Lips, n=5 | 379.0 [197 to 672]
  Nails,n=7: number analyzed (Participants) | 7
  Nails,n=7 | 379.0 [197 to 462]
  Mucosa, n=8: number analyzed (Participants) | 8
  Mucosa, n=8 | 201.0 [175 to 425]

33. Secondary Outcome: Percentage Change in the 28-day Partial Seizure Rate From the Baseline Phase (Obtained During the 8-week Baseline Period of Study VRX-RET-E22-302) to Open-label Treatment.
Description: 28-day partial seizure rate observed during the OLE period was compared to the 28-day partial seizure rate observed during the Baseline phase of the double-blind parent study VRX-R ET-E22-302. Percent change from Baseline in 28-day total partial seizure rate was calculated as ([28-day partial seizure frequency for the period of interest - Baseline 28-day partial seizure frequency] / Baseline 28-day partial seizure frequency) × 100 percent. A negative percent change indicated a reduction (improvement) from Baseline, so the best possible outcome was -100 percent. Only those participants with data available at the indicated time point were analyzed.
Time Frame: Baseline and up to 121 months
Population: Safety Population
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | Retigabine
Number analyzed (Participants) | 371
Percent change | -36.1 (95.77)

34. Secondary Outcome: Percentage of Participants With 50% Reduction in Seizure Frequency From Baseline Phase of the Parent Study (VRX-RET-E22-302) to Open Label Treatment
Description: A Responder was defined as a participant with >=50 percent decrease from Baseline in the 28-day partial seizure frequency, i.e., a percent change from Baseline less than or equal to -50 percent. The percentage of responders from Baseline phase of the parent study (VRX-RET-E22-302) to open label treatment have been presented.
Time Frame: Baseline and up to 121 months
Population: Safety Population
Measure: Number; unit: Percentage of participants
Arm/Group | Retigabine
Number analyzed (Participants) | 371
Percentage of participants | 52

35. Secondary Outcome: Number of Participants Who Were Seizure Free for Any 6 Continuous Months
Description: Seizure free for any continuous 6 months is defined as no seizures occuring during any consecutive 180 days between the first date (Baseline) and the last date (before tapering of dose). The number of participants who were seizure free for 6 continuous months within the 121 month OLE period have been presented.
Time Frame: Up to 6 continuous months within the 121 months period
Population: Safety Population
Measure: Number; unit: Participants
Arm/Group | Retigabine
Number analyzed (Participants) | 279
Participants | 36

36. Secondary Outcome: Number of Participants Who Were Seizure Free for Any 12 Continuous Months
Description: Seizure free for any continuous 12 months is defined as no seizures occurring during any consecutive 360 days. Number of participants who were seizure free for 12 continuous months within the 121 month OLE period have been presented.
Time Frame: Up to 12 continuous months within the 121 months period
Population: Safety Population
Measure: Number; unit: Participants
Arm/Group | Retigabine
Number analyzed (Participants) | 222
Participants | 22

37. Secondary Outcome: Percentage of Seizure Free Days
Description: A seizure free day is defined as the number of applicable days without any seizures (partial, generalized or unclassified). Only the days in which a subject had non-missing seizure data were considered as applicable days. Percentage of seizure free days is calculated as Number of seizure free days / number of applicable days × 100 percent. Only those participants with data available at the indicated time point were analyzed.
Time Frame: Up to 121 months
Population: Safety Population
Measure: Mean (Standard Deviation); unit: Percentage of days
Arm/Group | Retigabine
Number analyzed (Participants) | 371
Percentage of days | 76.8 (26.11)

ADVERSE EVENTS:
Time Frame: Serious adverse events (SAEs) and non-serious adverse events (AEs) were collected from the start of the study treatment up to 122 months.
Description: Safety population was used to assess AEs and SAEs.
Arm/Group | Retigabine
All-Cause Mortality (participants affected / at risk) | 7/376
Serious Adverse Events (participants affected / at risk) | 78/376
Other Adverse Events (participants affected / at risk) | 239/376
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Retigabine (N=376)
Seizure (Nervous system disorders) | 16
Epilepsy (Nervous system disorders) | 6
Generalised tonic-clonic seizure (Nervous system disorders) | 5
Status epilepticus (Nervous system disorders) | 5
Dizziness (Nervous system disorders) | 3
Focal dyscognitive seizures (Nervous system disorders) | 3
Coma (Nervous system disorders) | 2
Arachnoid cyst (Nervous system disorders) | 1
Ataxia (Nervous system disorders) | 1
Cerebrovascular accident (Nervous system disorders) | 1
Depressed level of consciousness (Nervous system disorders) | 1
Dysarthria (Nervous system disorders) | 1
Facial paralysis (Nervous system disorders) | 1
Incoherent (Nervous system disorders) | 1
Partial seizures (Nervous system disorders) | 1
Partial seizures with secondary generalisation (Nervous system disorders) | 1
Seizure cluster (Nervous system disorders) | 1
Psychotic disorder (Psychiatric disorders) | 4
Confusional state (Psychiatric disorders) | 3
Psychogenic seizure (Psychiatric disorders) | 2
Aggression (Psychiatric disorders) | 1
Agitation (Psychiatric disorders) | 1
Anxiety (Psychiatric disorders) | 1
Disorientation (Psychiatric disorders) | 1
Epileptic psychosis (Psychiatric disorders) | 1
Hallucination (Psychiatric disorders) | 1
Hallucination, auditory (Psychiatric disorders) | 1
Hallucinations, mixed (Psychiatric disorders) | 1
Obsessive-compulsive personality disorder (Psychiatric disorders) | 1
Postictal psychosis (Psychiatric disorders) | 1
Suicidal ideation (Psychiatric disorders) | 1
Suicide attempt (Psychiatric disorders) | 1
Accidental overdose (Injury, poisoning and procedural complications) | 1
Burns second degree (Injury, poisoning and procedural complications) | 1
Burns third degree (Injury, poisoning and procedural complications) | 1
Fall (Injury, poisoning and procedural complications) | 1
Femoral neck fracture (Injury, poisoning and procedural complications) | 1
Foot fracture (Injury, poisoning and procedural complications) | 1
Head injury (Injury, poisoning and procedural complications) | 1
Hip fracture (Injury, poisoning and procedural complications) | 1
Humerus fracture (Injury, poisoning and procedural complications) | 1
Intentional overdose (Injury, poisoning and procedural complications) | 1
Jaw fracture (Injury, poisoning and procedural complications) | 1
Near drowning (Injury, poisoning and procedural complications) | 1
Radius fracture (Injury, poisoning and procedural complications) | 1
Rib fracture (Injury, poisoning and procedural complications) | 1
Road traffic accident (Injury, poisoning and procedural complications) | 1
Skull fractured base (Injury, poisoning and procedural complications) | 1
Appendicitis (Infections and infestations) | 1
Bronchitis (Infections and infestations) | 1
Cellulitis (Infections and infestations) | 1
Gastroenteritis (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 1
Pneumonia mycoplasmal (Infections and infestations) | 1
Pneumonia streptococcal (Infections and infestations) | 1
Septic shock (Infections and infestations) | 1
Typhoid fever (Infections and infestations) | 1
Retinal pigmentation (Eye disorders) | 3
Diplopia (Eye disorders) | 1
Vision blurred (Eye disorders) | 1
Sudden unexplained death in epilepsy (General disorders) | 3
Chest pain (General disorders) | 1
Non-cardiac chest pain (General disorders) | 1
Adenocarcinoma of colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Non-Hodgkin's lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Plasma cell myeloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Deep vein thrombosis (Vascular disorders) | 1
Hypertensive crisis (Vascular disorders) | 1
Peripheral arterial occlusive disease (Vascular disorders) | 1
Peripheral ischaemia (Vascular disorders) | 1
Angina pectoris (Cardiac disorders) | 1
Atrial fibrillation (Cardiac disorders) | 1
Cardiac arrest (Cardiac disorders) | 1
Acute abdomen (Gastrointestinal disorders) | 1
Intestinal obstruction (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 1
Cholecystitis (Hepatobiliary disorders) | 1
Cholelithiasis (Hepatobiliary disorders) | 1
Drug-induced liver injury (Hepatobiliary disorders) | 1
Hyponatraemia (Metabolism and nutrition disorders) | 2
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1
Hydronephrosis (Renal and urinary disorders) | 1
Nephropathy toxic (Renal and urinary disorders) | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 2
Vertigo (Ear and labyrinth disorders) | 1
Adrenal insufficiency (Endocrine disorders) | 1
Pigmentation disorder (Skin and subcutaneous tissue disorders) | 1
Treatment noncompliance (Social circumstances) | 1
Tracheostomy (Surgical and medical procedures) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Retigabine (N=376)
Dizziness (Nervous system disorders) | 83
Somnolence (Nervous system disorders) | 78
Headache (Nervous system disorders) | 61
Tremor (Nervous system disorders) | 34
Memory impairment (Nervous system disorders) | 26
Seizure (Nervous system disorders) | 22
Aphasia (Nervous system disorders) | 20
Amnesia (Nervous system disorders) | 19
Viral upper respirator tract infection (Infections and infestations) | 30
Influenza (Infections and infestations) | 24
Urinary tract infection (Infections and infestations) | 21
Fatigue (General disorders) | 43
Back pain (Musculoskeletal and connective tissue disorders) | 22
Oral mucosal discolouration (Gastrointestinal disorders) | 20
Vertigo (Ear and labyrinth disorders) | 19

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.

DOCUMENTS (2):
  • Study Protocol (2008-08-14): https://cdn.clinicaltrials.gov/large-docs/88/NCT00310388/Prot_000.pdf
  • Statistical Analysis Plan (2007-02-26): https://cdn.clinicaltrials.gov/large-docs/88/NCT00310388/SAP_001.pdf